

# **Galáp**agos

Document title AMENDED CLINICAL STUDY PROTOCOL

Study official title Efficacy and safety of 3 doses of S201086/GLPG1972

> administered orally once daily in patients with knee osteoarthritis. A 52-week international, multi-regional, double-blind, multi-center, randomized, placebo-

controlled, dose-ranging study

ROCCELLA Study

Efficacy of S201086/GLPG1972 in patients with knee Study brief title

osteoarthritis

Test drug code S201086/GLPG1972

Indication Osteoarthritis

Development phase Phase 2

Protocol code CL2-201086-002/GLPG1972-CL-201

EudraCT Number 2017-004581-10

Universal Trial Number U1111-1205-0321

Investigational New Drug

Application Number

133039

Sponsor GALAPAGOS NV (US)

Institut de Recherches Internationales Servier (I.R.I.S.)

(ex-US)

Date of the document

09 December 2019

Version of the document Final version

# Amendment integrated

| No | Final version date | Countries concerned |
|----|--------------------|---------------------|
| 1 | 11/JUL/2018 | ALL |
| 1 | 12/JUL/2018 | US |
| 2 | 12/MAR/2019 | ALL |
| 3 | 09/DEC/2019 | US |

# CONFIDENTIAL

# **CONFIDENTIALITY STATEMENT**

This document is the confidential property of: INSTITUT DE RECHERCHES INTERNATIONALES SERVIER (I.R.I.S.) and Galapagos NV (Galapagos). It is intended for your personal information. You hereby covenant that, for a period of twenty (20) years from the date of receipt of this document, this document shall:

(a) be protected and kept in strict confidence by you;

- (b) neither be disclosed nor caused to be disclosed whether directly or indirectly to any third party or persons without I.R.I.S.' or Galapagos' prior written agreement;
- (c) not be used in whole or in part for any purpose other than as prior agreed in writing by I.R.I.S. or Galapagos;
- (d) neither be copied, nor otherwise reproduced nor duplicated in whole or in part where such copying, reproduction or duplication have not been specifically authorized in writing by I.R.I.S. or Galapagos.

# FOLLOW-UP OF VERSIONS

| | Amendment<br>No | Final<br>version<br>date | Countries concerned | Nature of modifications |
|---|---|---|---|---|
| Initial protocol | NA | 27/FEB/<br>2018 | ALL | Not Applicable |
| Initial<br>protocol,<br>US<br>specific | NA | 27/FEB/<br>2018 | US | The initial protocol has been adapted related to the following: - Addition of Galapagos logo and address on front page. - Addition of confidentiality statement on page 2. - Change of signature page, addition of Galapagos representative on signature page. - Addition of emergency contact information, specific for the US. - Minor textual changes. |
| Amended<br>protocol | 1 | 11/JUL/2<br>018 | ALL | <ul> <li>Increase the age of female patients of non-childbearing potential to 50 years old instead of 40 years old (inclusion criterion n°1) (except for female patients surgically sterile).</li> <li>Management of an overdose of S201086/GLPG1972 has been added on section 5.5.1 withdrawal criteria and section 8.9.2.4 special situations.</li> <li>Additional withdrawal criterion "delta &gt; 60 ms over baseline value (inclusion)" on ECG parameters (section 5.5.1 withdrawal criteria).</li> <li>Statistical analysis between Japanese patients and non-Japanese patients (section 10).</li> <li>Clarifications have been made.</li> <li>For a complete list of modifications, see Appendix 5.</li> </ul> |
| Amended<br>protocol,<br>US<br>specific | 1 | 12/JUL/2<br>018 | US | Changes as described in substantial Amendment No 1 (see Appendix 5) have been made as well as updated description of informed consent procedure (i.e. collection of one original informed consent form; see section 13.3 and 13.4). For an overview of US-specific modifications, see Appendix 6. |

| Amended<br>protocol | 2 | 12 MAR<br>2019 | ALL | <ul> <li>Update of inclusion criteria n°7, <ul> <li>9 in section 5.1 and exclusion criteria n° 24, 25, 27, 28, 29, 31, 32, 33, 38, 40, 44 in section 5.2</li> </ul> </li> <li>Update of section 6.6 forbidden/authorised concomitant treatments</li> <li>For a complete list of modifications, see Appendix 7.</li> </ul> |
|---|---|---|---|---|
| Amended | 3 | 09<br>DEC<br>2019 | US | <ul> <li>Update in emergency contact information, specific for the US.</li> <li>Addition of an exploratory endpoint regarding</li> <li>Changes in organisation and measures to minimize bias because of (see Section 4.3).</li> <li>Additional minor corrections have been made.</li> <li>For a complete list of modifications, see Appendix 9.</li> </ul> |



#### STUDY SUMMARY SHEET



| Name of the sponsor:<br>I.R.I.S. (ex-US)/Galapagos NV (US) | Individual<br>Referring to Pa | Study<br>art of the | | (For National Authority Use only) |
|---|---|---|---|---|
| Name of Finished Product: Not applicable | Volume: | | | |
| Name of Active Ingredient:<br>S201086-1/G504572 | Page: | | | |
| Title of study: Efficacy and safety of 3 doses of S201086 osteoarthritis. A 52-week international controlled, dose-ranging study. ROCCELLA study. Protocol No.: CL2-201086-002/GLPG197 National Coordinators and Investigator National coordinators and investigators: list Study centers: | multi-regiona | al, multic | center, r | |
| Planned total number of centers = 90-110<br>Planned total number of countries = 12 | -15 | | | |
| Study period: | | | Stu | idy development phase: 2 |
| - Study duration for the patient: max. 61 | weeks | | | |
| - Study initiation date (FVFP): Q2 2018 | | | | |
| - Study completion date (LVLP): Q4 20 | 20 | | | |

## **Objectives:**

The objectives of this study are to evaluate the efficacy and safety of 3 doses of S201086/GLPG1972 compared to placebo in patients with knee osteoarthritis (OA).

**The primary objective** of the study is to demonstrate the efficacy of at least one dose (among 3 doses) of S201086/GLPG1972 compared to placebo after 52 weeks of treatment in reducing cartilage loss measured by cartilage thickness using quantitative magnetic resonance imaging (qMRI) of the central medial tibiofemoral compartment (cMTFC) of the target knee.

#### The secondary objectives are:

To assess the safety and tolerability of 3 doses of S201086/GLPG1972.

To assess efficacy of 3 doses of S201086/GLPG1972 versus placebo after 52 weeks of treatment on:

- √ the proportion of "structural progressors\*" based on cartilage thickness using qMRI of the cMTFC of
  the target knee
- ✓ pain, function, and stiffness measured with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
- ✓ pain measured with a 100-mm visual analog scale (VAS)
- ✓ patient global assessment (PGA) of disease activity measured with 100-mm VAS
- ✓ reduction of cartilage loss measured by cartilage thickness using qMRI of the total tibiofemoral compartment (tTFC) of the target knee
- ✓ Joint Space Width (JSW) measured by x-ray

To assess efficacy of 3 doses of S201086/GLPG1972 versus placebo after 28 and 52 weeks of treatment on bone area using qMRI of the medial femoral condyle surface of the target knee.

To assess the pharmacokinetics of S201086/GLPG1972 (and metabolite[s] if applicable).

To assess efficacy of 3 doses of S201086/GLPG1972 versus placebo after 52 weeks of treatment on analgesic consumption.

Exploratory objectives are:

<sup>\*</sup>defined as patient who had at least 8% cartilage loss in the cMTFC between baseline and week 52 (W052).

| Name of the sponsor: | Individual | Study | Table | (For National Authority Use only) |
|---|---|---|---|---|
| I.R.I.S. (ex-US)/Galapagos NV (US) | Referring to | Part of the | Dossier | |
| Name of Finished Product: | Volume: | | | |
| Not applicable | | | | |
| Name of Active Ingredient: | Page: | | | |
| S201086-1/G504572 | _ | | | |

#### Methodology:

Study design: international, multi-regional, multicenter, randomized, double-blind, parallel groups, placebo-controlled dose-ranging phase 2 study.

The randomization will be stratified by zone (Japan, South Korea/Taiwan and Rest of the World).

The study will consist of:

- Screening period without study treatment: up to 5 weeks to assess the eligibility of patients
- Randomization and double-blind treatment period: 52 weeks with 4-parallel groups (doses: 75, 150 and 300 mg/day of S201086/GLPG1972 and matching placebo)
- Follow-up period without study treatment: 2 weeks

A Data and Safety Monitoring Board (**DSMB**) will be put in place in order to independently review the available safety data at regular pre-specified time points. The functioning of this DSMB is specified in a separate DSMB charter.

#### **Number of patients:**

Planned: approximately 852 patients

Per treatment group (arm): approximately 213 patients

#### Diagnosis and main criteria for inclusion:

The target population is male or female of non-childbearing potential patients suffering from mild to moderate clinical and radiologic knee OA.

Main screening criteria are:

Male patients or female patients of non-childbearing potential, age 40-75 years for male patients and female surgically sterile patients, and 50-75 years for postmenopausal female patients, body weight > 40 kg, body mass index (BMI) < 40 kg/m², diagnosed for knee osteoarthritis based on **clinical and radiological criteria** of the American College of Rheumatology, with a history of knee pain for at least 6 months and on the majority of days (> 50%) during the preceding month and with a severity  $\geq$  40 mm and  $\leq$  90 mm on VAS (100 mm). Patients will be selected based on symptom severity defined by a pain  $\geq$  40 mm and  $\leq$  90 mm on a 100 mm VAS at screening and inclusion visits, with knee OA classified as radiographic grade 2 or 3 of the Kellgren and Lawrence (KL) scale and OARSI grade 1 or 2 medial tibiofemoral joint space narrowing (JSN) and will have a documented need for symptomatic as needed-treatment for OA in the target knee with systemic non-steroidal anti-inflammatory drugs (NSAIDs) and/or other analgesics.

# Investigational Medicinal Product (IMP): test drug and comparator:

Test drug:

**Name:** S201086/GLPG1972 **Doses:** 75 mg – 150 mg – 300 mg

**Dosage form:** film-coated tablet containing 75 mg S201086-1/G504572 (S201086-1/G504572 is the compound

code for S201086/GLPG1972)

Comparator: Name: placebo

Dosage form: film-coated matching tablet

**Mode of administration:** take 4 tablets once a day, from the blister, with a glass of water, preferably in the morning

#### **Duration of treatment:**

Run-in period: no treatment up to 5 weeks of screening period

| Name of the sponsor: | Individual Study Table (For National Authority Use only) |
|---|---|
| I.R.I.S. (ex-US)/Galapagos NV (US) | Referring to Part of the Dossier |
| Name of Finished Product: | Volume: |
| Not applicable | |
| Name of Active Ingredient: | Page: |
| S201086-1/G504572 | |

Active treatment period: fifty-two (52) weeks of treatment period Follow-up period: no treatment during 2 weeks follow-up period

#### Criteria for evaluation:

Efficacy measurements:

Primary efficacy endpoint:

The change from baseline to W052 in cartilage thickness of the cMTFC of the target knee: qMRI.

Secondary efficacy endpoints:

- Proportion of structural progressors\* at W052 based on cartilage thickness of the cMTFC of the target knee: qMRI
- The change from baseline to W052 in WOMAC total score and subscales scores of the target knee for pain, function and stiffness
- The change from baseline to W052 in pain of the target knee: 100-mm VAS
- The change from baseline to W052 in PGA of disease activity of the target knee: 100-mm VAS
- The proportion of Outcome Measures in Rheumatology (OMERACT)-OARSI responders\*\* at W052: defined according to WOMAC and PGA
- The change from baseline to W052 in cartilage thickness of the tTFC of the target knee: qMRI
- The change from baseline to W028 and to W052 in bone area of the medial femoral condyle surface of the target knee: qMRI
- The change from baseline to W052 in JSW of the target knee: X-Ray
- Pain: Analgesic consumption at every visit up to W052
- \*\* based on OMERACT-OARSI Initiative: Osteoarthritis Research Society International set of responder criteria for osteoarthritis clinical trials revisited Pham et al. 2004. Defined according to WOMAC and patient's global assessment as a patient who had:
  - high improvement in pain or in function ≥ 50% and absolute change ≥ 20 or
  - moderate improvement in at least 2 of the 3 following:
    - Pain ≥ 20% and absolute change ≥ 10
    - Function ≥ 20% and absolute change ≥ 10
    - Patient's global assessment  $\geq$  20% and absolute change  $\geq$  10.

Other secondary endpoints:

#### Safety

The safety and tolerability assessed by the incidence of adverse events (AEs), changes over time in safety parameters and incidence of abnormal safety parameters throughout the study.

#### Pharmacokinetics:

Pharmacokinetics of S201086/GLPG1972 (and metabolite[s] if applicable)

Explorator<u>y</u> endpoints:



| Name of the sponsor:<br>I.R.I.S. (ex-US)/Galapagos NV (US) | Individual<br>Referring to I | Study<br>Part of the | (For National Authority Use only) |
|---|---|---|---|
| Name of Finished Product:<br>Not applicable | Volume: | | |
| Name of Active Ingredient:<br>S201086-1/G504572 | Page: | | |
| • | | | |

#### Statistical methods:

#### Analysis sets:

## - Modified Randomized Set (mRS):

The modified Randomised Set (mRS) will be constituted of all included patients to whom a therapeutic unit was randomly assigned using interactive web response system IWRS. The RS will be used for efficacy analyses. Patients will be analysed according to the randomised treatment.

#### - Safety Set (SS):

The Safety Set (SS) will be constituted of all patients having taken at least one dose of IMP. The SS will be used for safety analyses. Patients will be analysed according to treatment actually received at inclusion.

#### Sample size calculation:

The determination of the sample size was performed considering the change from baseline to W052 in cartilage thickness in the cMTFC, expressed in mm and measured by qMRI.

The primary objective is to demonstrate that at least one S201086/GLPG1972 dose is superior to placebo in the mRS, based on a two-sided Dunnett test for multiple comparisons. The Dunnett test is used in order to maintain the experiment wise type I error at 5% (two-sided setting).

Two hundred and thirteen (213) patients per treatment group will provide a minimal power of approximately 70% to conclude for at least one dose that S201086/GLPG1972 is superior to placebo if the true difference is 0.0825mm for at least one dose, assuming a standard deviation of 0.30 mm (Lohmander et al., 2014).

#### Efficacy analysis:

In order to take into account the multiplicity of comparisons induced by the assessment of three S201086/GLPG1972 doses versus placebo, a Dunnett procedure will be used.

#### Primary endpoint:

In order to meet the primary objective of the study, the efficacy of at least one dose of S201086/GLPG1972 as compared to placebo after 52 weeks of treatment in reducing cartilage loss in patients with knee OA will be assessed from the change from baseline to W052 in cartilage thickness as measured in the medial central tibiofemoral compartment on the target knee, in patients of the mRS. A restricted maximum likelihood (REML)-based, mixed-effects model for repeated measures approach (so called Mixed-effects Model for Repeated Measures – MMRM) using all longitudinal observations at each post-baseline visit will be used (main analysis). The MMRM as a primary analysis will assume that patients would keep the benefit of the randomized treatment after study discontinuation. A missing data Handling will be used for this analysis. The treatment comparisons associated with the primary analysis will be the contrasts between each dose of S201086/GLPG1972 and placebo at the change from baseline to W052. Analysis will include the fixed, categorical effects of treatment, regions, time and treatment-by-time interaction, as well as the continuous, fixed covariates of baseline, time-by-baseline interaction.

The analysis will fit an unstructured covariance matrix, and the assumptions underlying the model will be checked.

| Name of the sponsor: | Individual | Study | Table | (For National Authority Use only) |
|---|---|---|---|---|
| I.R.I.S. (ex-US)/Galapagos NV (US) | Referring to | Part of the | Dossier | |
| Name of Finished Product: | Volume: | | | |
| Not applicable | | | | |
| Name of Active Ingredient: | Page: | | | |
| S201086-1/G504572 | _ | | | |

The consistency of the results between the Asian population and the non-Asian population (respectively between Japanese population and non-Japanese population) will be evaluated on primary endpoint, according to the Method 2 defined in Ministry of Health Labor and Welfare Notification (MHLW) Notification "Basic principles on Global Clinical Trials". Treatment effect estimates and confidence intervals will be provided, for each dose, in Asian population and non-Asian population (respectively between Japanese population and non-Japanese population). In case of a statistically significant overall treatment effect (in favor of S201086/GLPG1972) at a considered dose, the results will be considered consistent if the observed treatment effects in Asian and non-Asian patients are (respectively between Japanese population and non-Japanese population) in favor of S201086/GLPG1972.

Sensitivity analyses will be performed to assess the robustness of the primary analysis results to the method of handling missing data.

# Secondary endpoints:

For the proportion of "structural progressors" and proportion of OMERACT-OARSI responders at W052, the difference between each S201086/GLPG1972 dose and placebo will be studied in patients of the mRS, considering a multiple imputation for handling all missing data and using a logistic model, including the fixed, categorical effects of treatment, regions (Asia and Rest of the World), as well as the continuous, fixed covariates of baseline.

The difference between each S201086/GLPG1972 dose and placebo will be studied in patients of the mRS, on continuous secondary efficacy endpoints at W052, with the same strategy as the main analysis of the primary endpoint: multiple imputation for patients without any post-baseline value followed by a MMRM using all the longitudinal observations at each post-baseline visit. Analysis will include the fixed, categorical effects of treatment, regions (Asia and Rest of the World), visit and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline, visit-by-baseline interaction.

For the change from baseline to W052 in JSW and the change from baseline to W028 in bone area, the difference between each S201086/GLPG1972 dose and placebo will be studied in patients of the mRS at W052 (respectively W028), considering a multiple imputation method for handling all missing data at W052 (respectively W028), and using an ANCOVA. Analysis will include the fixed, categorical effects of treatment, regions (Asia and Rest of the World), as well as the continuous, fixed covariate of baseline.

For analgesic consumption, number and percentage of patients by treatment reported will be provided, overall and by treatment group.

For each treatment group, descriptive statistics will be provided for all secondary endpoints, overall and by regions.

Study patients (disposition, baseline characteristics and follow-up) and safety analysis: Descriptive statistics will be provided.

#### Pharmacokinetic analysis:

Plasma concentrations of S201086/GLPG1972 (and those of metabolite[s] if applicable) will be documented with descriptive statistics (mean, median, standard deviation, minimum and maximum) at each time-point and each dose for trough plasma concentration (Ctrough) values.

S201086/GLPG1972 (and metabolite[s] if applicable) plasma concentration measurement will be used in order to build a population pharmacokinetics model. This analysis will provide pharmacokinetic parameters and their associated variability. The influence of covariates will be investigated. The pharmacokinetic analysis will be described in separate Data Analysis Plan (DAP) and report.

| Name of the sponsor: | | (For Nationa | l Authority Use only) |
|---|---|---|---|
| I.R.I.S. (ex-US)/Galapagos NV (US) Name of Finished Product: | Referring to Part of the Dossier Volume: | | |
| Not applicable | volume: | | |
| Name of Active Ingredient: | Page: | | |
| S201086-1/G504572 | - 1.5.1 | | |
| Contractual signatories | | | |
| I, the undersigned, have read the foregoin<br>attached to the protocol and agree to con<br>Practice (GCP) and the applicable regulate | nduct the study in compliance w | | |
| | NAME | DATE | SIGNATURE |
| INVESTIGATOR : | | | |
| CENTER | | | |
| NUMBER | | | |
| GALAPAGOS NV REPRESENTATIV | Æ | | |
| CITATIONI DESCRIT OBMERE LE LA DE | | | |
| CLINICAL DEVELOPMENT LEADE | R: | | |

# **EMERGENCY CONTACT INFORMATION – US ONLY**

In case of medical **questions** during the course of the study, the investigator must contact the CRO Medical Monitor or, if unavailable, his/her back up.





# **Table of contents**

| CONFIDENTIALITY STATEMENT | 2 |
|-----------------------------------------------------------------------|----|
| FOLLOW-UP OF VERSIONS | 3 |
| STUDY SUMMARY SHEET | 5 |
| Emergency Contact Information – US ONLY | 11 |
| Table of contents | 12 |
| List of tables | 16 |
| List of figures | 17 |
| List of appendices | 18 |
| List of abbreviations | 19 |
| EMERGENCY CONTACT INFORMATION – US ONLY | 11 |
| 1. ADMINISTRATIVE STRUCTURE OF THE STUDY | 22 |
| 2. BACKGROUND INFORMATION | 23 |
| 3. STUDY OBJECTIVES AND PURPOSE | 30 |
| 4. STUDY DESIGN | 31 |
| 4.1. Endpoints | 31 |
| 4.2. Experimental design | |
| 4.2.1. Study plan | 32 |
| 4.2.2. Investigation schedule | |
| 4.3. Measures to minimize bias | |
| 4.4. Data and safety monitoring board | 36 |
| 5. INCLUSION OF PATIENTS | 37 |
| 5.1. Inclusion criteria | 37 |
| 5.2. Exclusion criteria | 37 |
| 5.3. Contraception | 39 |
| 5.4. Discontinuation of the study | |
| 5.4.1. Premature discontinuation of the study or temporary halt | |
| 5.4.2. Discontinuation of the study in the event of objective reached | |
| 5.5. Patient withdrawal | |
| 5.5.1. Withdrawal criteria | 40 |
| 5.5.2. Procedure | 41 |
| 5.5.3. Lost to follow-up | 42 |
| 6. TREATMENT OF PATIENTS | 43 |
| 6.1. Study products and blinding systems | |
| 6.1.1. Products administered | |
| 6.1.2. IMP management | |
| 6.1.3. Management of blinding systems | |
| 6.2. IMPs administered | |
| 6.3. IMPs dispensing | |
| 6.4. IMP compliance | 46 |

| 6.5. | Discontinuation of the IMP. | 46 |
|---|---|---|
| 6.6. | Previous and concomitant treatments | 46 |
| 7 A | SSESSMENT OF EFFICACY | 49 |
| 7. 21 | | 1> |
| 7.1. | | |
| | Methods and measurement times. | |
| | Medical imaging | |
| | . WOMAC for measurement of pain, function and stiffness (Appendix 2) | |
| | . VAS for pain intensity (Appendix 3) | |
| 7.2.4 | . VAS for Patient Global Assessment of disease activity (PGA) (Appendix 4) | 50 |
| 7.2.5 | . Analgesic consumption | 51 |
| 8. SA | AFETY MEASUREMENTS | 52 |
| 8.1. | Specification of safety parameters | 52 |
| 8.2. | Methods and measurement times. | |
| 8.3. | Definition of Adverse events | |
| 8.4. | Definition of Serious adverse events | |
| 8.5. | Definition of special situations | |
| 8.6. | Definition of Adverse event of special interest | |
| 8.7. | Definition of Events requiring an immediate notification (ERIN) | |
| 8.8. | Classification of an adverse event (seriousness, severity, causality) | |
| 8.9. | Reporting procedures | |
| | . Time frame for adverse event reporting | |
| | Responsibilities of the investigator | |
| 8.9.2 | • | |
| 8.9.2 | | |
| 8.9.2 | ± | |
| 8.9.2 | | |
| 8.9.2 | | |
| 8.9.2 | | |
| 8.9.2 | • | |
| | Responsibilities of the sponsor | |
| 0.9.3<br>Q 10 | Responsibilities of data safety monitoring board | 61 |
| 8.10. | Responsibilities of data safety monitoring board | 01 |
| | THER ASSESSMENTS NOT SPECIFICALLY RELATED TO EFFICACY | |
| O | R SAFETY | 62 |
| 9.1. | Pharmacokinetics | 62 |
| 9.2. | | 62 |
| 9.2.1 | | |
| 9.2.2 | | 62 |
| 9.2.3 | | |
| 9.2.4 | | 63 |
| 9.2.5 | | 63 |
| 9.2.6 | | 64 |
| | Assessment related to exclusion criteria | |
| 10. | STATISTICS | 65 |
| 10. | ~ | 05 |

| | Statistical analysis | |
|---|---|---|
| 10.1. | 1. Endpoints | 65 |
| | 1.1. Efficacy endpoints | |
| 10.1. | 1.1.1. Primary efficacy endpoint | 65 |
| | 1.1.2. Secondary efficacy endpoints | |
| 10.1. | 1.2. Safety endpoints | 65 |
| 10.1. | 1.3. | 66 |
| 10.1. | 1.4. Other endpoints | 67 |
| | 1.5. Pharmacokinetics endpoints | |
| | 2. Analysis sets and subgroups / Treatment groups | |
| | 2.1. Analysis sets and subgroups | |
| | 2.2. Treatment groups | |
| | 3. Statistical methods | |
| | 3.1. General considerations | |
| | 3.1.1. Multiplicity issues | |
| | 3.1.2. Handling of missing data | |
| | 3.1.3. Statistical elements | |
| | 3.1.3.1. Descriptive statistics | |
| | 3.1.3.2. Estimations and statistical tests. | |
| | 3.2. Study patients: Disposition, baseline characteristics and follow-up | |
| | 3.3. Efficacy analysis | |
| | 3.3.1. Primary efficacy endpoint | |
| | 3.3.1.1. Primary analysis | |
| | 3.3.1.2. Secondary analyses | |
| | 3.3.2. Secondary efficacy endpoints | |
| | 3.4. Safety analysis | |
| | 3.4.1. Adverse events | |
| | 3.4.2. Clinical laboratory evaluation | |
| | 3.4.3. Vital signs, clinical examination and other observations related to safety | |
| | 3.4.3.1. Vital signs and clinical examination | |
| | 3.4.3.2. Electrocardiogram | |
| | 3.4.3.3. Special situations not associated with an AE | |
| | 3.5. Exploratory analysis | |
| | 4. Interim analysis | |
| 10.2. | Determination of sample size | 73 |
| | 1 | |
| 11. | DIRECT ACCESS TO SOURCE DATA / DOCUMENTS | 74 |
| <b>12.</b> | QUALITY CONTROL AND QUALITY ASSURANCE | 75 |
| 12.1 | Study monitoring | 75 |
| | Study monitoring | |
| | · | |
| | 2. During the study | |
| | Computerized medical file | |
| | Audit - Inspection | |
| 12.4. | Supervisory committees | / / |
| 13. | ETHICS | 78 |
| 12 1 | Institutional Paviary Poord(s)/Indopendent Ethics Committee(s) | 70 |
| | Institutional Review Board(s)/Independent Ethics Committee(s) | |
| 13.2. | Study conduct | / 8 |

| 13.3. | . Patient information and informed consent | 78 |
|------------|---------------------------------------------------------|----|
| 13.4. | . Modification of the information and consent form | 79 |
| 14. | DATA HANDLING AND RECORD KEEPING | 80 |
| | . Source data | |
| | . Study data | |
| | . Data management | |
| 14.4. | . Archiving | 82 |
| 15. | INSURANCE | 83 |
| 15.1. | For non US countries: | 83 |
| | For US country only: | |
| | .1. Indemnification | |
| | .2. Insurance | |
| 16. | | |
| P | UBLICATION POLICY | 84 |
| <b>17.</b> | ADMINISTRATIVE CLAUSES | 85 |
| 17.1. | . Concerning the sponsor and the investigator | 85 |
| | .1. Persons to inform. | |
| 17.1. | .2. Substantial protocol amendment and amended protocol | 85 |
| | .3. Final study report | |
| | . Concerning the sponsor | |
| | . Concerning the investigator | |
| | .1. Confidentiality - Use of information | |
| | .2. Organization of the center | |
| | .3. Documentation supplied to the sponsor | |
| 18. | REFERENCES | 88 |
| 19. | APPENDICES | 01 |

# List of tables

| Table (4.2.2) 1 - Investigation schedule | 34 |
|---|---|
| Table (6.1.1) 1 – Description of the IMPs. | |
| Table (6.1.1) 2 – Description of packaging | |
| Table (6.6) 1 - Treatment prohibited during the study (non-exhaustive list) | |
| Table (6.6) 2 – Treatment authorized during the study with particular conditions for use | 48 |
| Table (6.6) 3 – Treatment authorized during the study | 48 |

# List of figures

# List of appendices

| Appendix 1: World Medical Association Declaration of Helsinki | 91 |
|---|---|
| Appendix 2: Western Ontario and McMaster Universities Osteoarthritis Index | |
| (WOMAC) | 97 |
| Appendix 3: Knee Pain Visual Analog Scale | 103 |
| Appendix 4: Patient Global Assessment of disease activity Visual Analog Scale | 104 |
| Appendix 5: Substantial Amendment No 1 to the clinical study protocol | 105 |
| Appendix 6: Local Amendment US No 1 to the clinical study protocol | 122 |
| Appendix 7: Substantial Amendment No 2 to the clinical study protocol | 125 |
| Appendix 8: Paper version of the VAS (pain & PGA) | 142 |
| Appendix 9: Non-substantial Amendment No 3 to the clinical study protocol | 145 |

#### List of abbreviations

AE : adverse event

ACR : American College of Rheumatology

ADAMTS : a disintegrin and metalloproteinase with thrombospondin motif

ADL : activities of daily living
ALT : ALanine aminoTransferase
ALP : alkaline phosphatase

Alu : aluminum

ANCOVA : analysis of covariance

ARGS : alanine-arginine-glycine-serine AST : ASpartate aminoTransferase

AUC<sub>0-24h</sub> : area under the plasma concentration-time curve from time 0 to

24 hours postdose

 $AUC_{0-\infty}$  : area under the concentration-time curve from time 0 extrapolated

to infinity

AUC<sub>T</sub> : area under the concentration-time curve for the dosing interval

BAP : blood arterial pressure

BINAP : (+/-)-2,2'-Bis(diphenylphosphino)-1,1'-binaphthyl

BMI : Body Mass Index

bpm : beats per minute (heart rate unit)

C<sub>max</sub>: maximum observed plasma concentration

CMP : clinical monitoring plan

cMTFC : central medial tibiofemoral compartment

CPK : creatinine phosphokinase

CRO : Contract Research Organisation

<u>CRP</u> : C-reactive protein

CSP : Clinical Study Protocol

CTCAE : Common Terminology Criteria for Adverse Events

C<sub>trough</sub>: trough plasma concentration

CV : curriculum vitae
CYP : cytochrome P450
DAP : data analysis plan
DBP : diastolic blood pressure
DC : direct compression

DMM : destabilization of the medial meniscus DMOAD : disease modifying osteoarthritis drug

DSMB : data safety monitoring board EAE : emergent adverse event

Eavg<sub>(0-24h)</sub> : average % reduction from time 0 to 24 h postdose

ECG : electrocardiogram

eCRF : electronic case report form
e.g. : exempli gratia (for example)
EMA : European Medicines Agency

ePRO : electronic patient reported outcome ERIN : Event Requiring Immediate Notification

g : gram

GAG : glycosaminoglycan GCP : Good Clinical Practice GFR : glomerular filtration rate

GGT : gamma glutamyl transferase (Gamma-Glutamyl Transpeptidase)

GLP : Good Laboratory Practice

h : hour

HBs : Surface antigen of Hepatitis B virus

HCV : hepatitis C virus

HDL : high density lipoprotein

hERG : human ether-a-go-go related gene

HIPAA : Health Insurance Portability and Accountability Act

HIV : human immunodeficiency virus

HR : heart rate

IC<sub>50</sub> : half maximal inhibitory concentration

ICF : informed consent form

ICH : International Conference on Harmonisation

i.e. : *id est* (that is)

IEC : independent ethics committee

IL1α : interleukin-1 alpha IL1β : interleukin-1 beta

IMP : Investigational Medicinal Product: a pharmaceutical form of an

active ingredient or placebo being tested or used as a reference

in a clinical trial (test drug / placebo)

IND : Investigational New Drug
INR : international normalized ratio
IRB : institutional review board

I.R.I.S. : Institut de Recherches Internationales Servier

IU : International Unit

IWRS : interactive web response system

JSN : joint space narrowing JSW : joint space width

kg : kilogram

KL : Kellgren and Lawrence system for classification of knee

osteoarthritis (X-ray)

L : liter

LDH : lactate dehydrogenase LDL : low density lipoprotein

MCH : mean corpuscular hemoglobin

MCHC : mean corpuscular hemoglobin concentration

MCV : mean corpuscular volume

MDRD : Modification of the Diet in Renal Disease MedDRA : Medical Dictionary for Regulatory Activities

mg : milligram min : minute

MHLW : Ministry of Health Labor and Welfare Notification

mL : Milliliter mm : Millimeter

mmHG : Millimetre of mercury

mmol : millimole

MMP : matrix metalloproteinase

MMRM : mixed-effects model for repeated measures

MNX : meniscectomy

MRI : magnetic resonance imaging mRS : modified Randomized Set

MTFC : Medial Tibiofemoral Compartment

msec : millisecond µmol : micromole

NDA : New Drug Application

ng : nanogram

NOAEL : no observed adverse effect level NSAIDS : non-steroidal anti-inflammatory drugs

NYHA : New York Heart Association

OA : osteoarthritis

OARSI : Osteoarthritis Research Society International

OMERACT : Outcome Measures in Rheumatology

PCSA : Potentially Clinically Significant Abnormalities

PGA : patient global assessment

PVC : polyvinylchloride QC : quality control

q.d. : quaque die, once daily

qMRI : quantitative magnetic resonance imaging

QTcF : QT interval corrected for heart rate by Fridericia formula

REML : restricted maximum likelihood

ROW : Rest of World

SAE : serious adverse event
SAP : statistical analysis plan
SAR : Serious Adverse Reactions
SBP : Systolic Blood Pressure
SCW : streptococcal cell wall

sec : second SS : Safety Set

TEAE : treatment-emergent adverse event t<sub>1/2</sub> : terminal elimination half-life tTFC : total tibiofemoral compartment t.i.d. : ter in die (three times a day)

T/L : Tera (10<sup>12</sup>) per litre

test drug : Drug substance in a given dosage form, tested in a clinical trial.

It corresponds to S201086/GLPG1972 product

t<sub>max</sub> : time to maximum observed plasma concentration

TSH : thyroid-stimulating hormone

TU : therapeutic unit

TUTF : Therapeutic Unit Tracking Form

ULN : upper limit of normal

V : Visit

VAS : visual analog scale

vs.WweekWDwithdrawalWGwet granulation

WHO-DRUG : World Health Organization, Drug Dictionary

WMA : World Medical Association

WOCBP : women of child-bearing potential

WOMAC : Western Ontario and McMaster Universities Osteoarthritis Index

## 1. ADMINISTRATIVE STRUCTURE OF THE STUDY

Galapagos will act as sponsor of the Study in the United States of America (including its territories and possessions) (the "US Territory") and Servier will act as sponsor of the Study in all countries except the US Territory (the "ROW Territories"). Each of Galapagos and Servier shall be solely responsible for the activities conducted in their respective territories, *i.e.*, Galapagos for the US Territory and Servier for the ROW Territories.

Non-sponsor parties, sponsors parties, and contract research organization (CRO) parties responsible for local management of the study are described in a separate document.

The list of investigators for each country is given in separate documents attached to the protocol.

The composition and role of the supervisory committees are described in Sections 8.3 and 12.4.

## 2. BACKGROUND INFORMATION

S201086 is also developed by Galapagos N.V. under the code GLPG1972.

# **Definition and epidemiology of osteoarthritis**

Osteoarthritis (OA) is a degenerative joint disease involving the structure of all joint tissues including articular cartilage, subchondral bone, ligaments, capsule, and synovial membrane. It may develop in any joint but most commonly affects the knees, hips, and hands.

The global prevalence of radiographically confirmed symptomatic OA has been estimated to be 3.8% for knee and 0.8% for hip (Cross, 2014), but this prevalence increases up to 10-40% in the elderly ((WHO, 2013), Framingham OA study). The prevalence of OA is expected to increase in the upcoming years, mainly due to the increasing prevalence of obesity and the ageing population (Elders, 2000; Zhang W et al., 2010).

# Standard of care treatment

Standard of care is a combination of non-pharmacological and symptomatic pharmacological treatments which should be personalized to the need of the individual patient. Despite a number of investigations of potential therapies, there are currently no approved disease-modifying drugs. Effective and safe long-term treatment for most OA patients is thus not available, creating a clear unmet medical need for structural protection (Karsdal, 2016).

# Aggrecanase in OA

Degradation of the cartilage extracellular matrix is a central feature of OA and is widely thought to be mediated by proteinases that degrade structural components of the matrix, primarily aggrecan and collagen. Among the different attempts to develop new agents for OA, inhibition of aggrecanase activity in diseased cartilage is thus considered a valid therapeutic approach (Karsdal, 2016). Aggrecan plays a central role on cartilage compressibility and elasticity during exercises or movements.

In OA, aggrecan is proteolyzed mainly by matrix metalloproteases (MMPs) and aggrecanases (a disintegrin and metalloproteinase with thrombospondin motifs [ADAMTS] 4 and -5). The cleavage of aggrecan by ADAMTS-5 is a crucial event in OA pathogenesis, both in rodents and in humans ((Fosang, 2008); (Verma and Dalal, 2011)). By breaking down the interaction between aggrecan and important structural components of the extracellular matrix (Heinegard and Saxne, 2011), an early event in OA, it favors the degradation of the matricial network of cartilage and alters the pericellular environment, ultimately leading to chondrocyte death.

The important contribution of ADAMTS-5 to OA pathogenesis was first demonstrated in preclinical models of OA. In a model of OA induced by destabilization of the medial meniscus, ADAMTS-5 knockout mice were protected from cartilage degradation (Glasson et al., 2005). Additionally, early preclinical candidates (small chemical entities/antibodies) demonstrated chondroprotective activity linked to ADAMTS-5 inhibition in animal models of OA ((Chockalingam, 2011); (Chiusaroli, 2013); (Chen P et al., 2014), (Caselli et al., 2015)). Importantly, ADAMTS-5 deficient mice did not develop mechanical allodynia associated with osteoarthritis, demonstrating that in addition to disease modifying OA drug (DMOAD) activity, ADAMTS-5 inhibition was also effective in pain relief in this model (Malfait et al., 2010); (Miller et al., 2016).

Degradation of aggrecan by ADAMTS-5 was identified as being involved in patients with OA. The expression of ADAMTS-5 was increased in articular cartilage samples obtained from OA patients (Chen S et al., 2014), and several studies reported that aggrecan fragments (ARGS,

NITEGE) generated after cleavage at the aggrecanase site were found at higher levels in cartilage, synovial fluid and sera from OA patients (Lohmander et al., 1993); (Sandy and Verscharen, 2001); (Struglics et al., 2011); (Zhang E et al., 2013); (Germaschewski, 2014). It was also demonstrated that compared to MMPs, ADAMTS-5 was the major contributor to aggrecan catabolism during OA (Lohmander et al., 1993); (Sandy, 2006); (Durigova, 2011).

Aggrecan cleavage by ADAMST-5 results in the release of the N-terminal neo-epitope ARGS fragments and these fragments were found to be increased in human knee synovial fluid and blood after joint injuries in OA patients waiting for a total knee replacement (Larsson et al., 2014).

In conclusion, ADAMTS-5 activity is exacerbated during OA, and its inhibition protects from cartilage degradation and is effective in reducing allodynia in preclinical models of OA, suggesting that it is a highly relevant target for DMOAD treatment.

# Overview of S201086/GLPG1972

S201086 also named GLPG1972, is a potent and selective inhibitor of ADAMTS-5 currently being developed as an oral treatment for OA.

ADAMTS-5 (aggrecanase-2, ADAMTS-11) is a member of the ADAMTS protein family. ADAMTS-5 is expressed in many tissues, with highest expression in uterus, placenta, and cartilage. ADAMTS-5 is the major aggrecanase in experimentally induced OA mouse models. Aggrecan cleavage by ADAMTS-5 results in the release of the N-terminal ARGS neoepitope fragments and these fragments were found to be increased in human knee synovial fluid after joint injuries and in OA. The discovery that ADAMTS-5 plays a major role in OA suggests that this enzyme may be a suitable target for the development of new drugs designed to inhibit cartilage destruction in arthritis.







#### Clinical studies

# Safety data

In Study GLPG1972-CL-101, administration of single (up to 2100 mg) and multiple (up to 1050 mg *q.d.* for 14 days) ascending oral doses of S201086/GLPG1972 in healthy subjects was well tolerated. No deaths, other serious adverse events (SAEs), or treatment-emergent adverse events (TEAE) leading to study drug discontinuation were reported during the study. All reported TEAEs were rated mild in intensity, were not dose-related, and were resolved by the end of the study.

In Study GLPG1972-CL-103, administration of single doses (600 mg) of S201086/GLPG1972 as oral solution in fasted state and as oral direct compression (DC) tablet in fasted and fed state in healthy male subjects was well tolerated. No deaths, other SAEs, or TEAEs leading to study drug discontinuation were reported during the study. All but 1 TEAE (moderate presyncope) were mild in intensity and all TEAEs were resolved by the end of the study.

In Study GLPG1972-CL-105, administration of a single dose (300 mg) of S201086/GLPG1972 as oral solution or wet granulation (WG) tablet in fasted state and as WG or DC tablet in fed state in healthy male subjects was well tolerated. No deaths or other SAEs were reported during the study. One subject experienced a TEAE of moderate migraine which led to study drug discontinuation. All other TEAEs were mild in intensity and all TEAEs were resolved/resolving by the end of the study.

In Study GLPG1972-CL-106, administration of 300 mg 201086/ GLPG1972 once daily (*q.d.*) for 10 days with or without a single 2-mg dose of midazolam in healthy male subjects was well tolerated. No deaths, other SAEs, or TEAEs leading to study drug discontinuation were reported during the study. All TEAEs were mild in intensity and all TEAEs were resolved by follow-up.

In Study GLPG1972-CL-104, administration of multiple oral doses of S201086/GLPG1972 (100, 200 or 300 mg q.d.) for 29 days in patients with OA was generally well tolerated. One patient dosed with GLPG1972 300 mg q.d. prematurely discontinued the study due to an increase in alanine aminotransferase (ALT) on Day  $15 \ge 3$  x the upper limit of normal (ULN), which was considered probably related to the study drug.

There were no overall trends in lab abnormalities over time or significant changes in vital signs, physical examinations, 12-lead ECG, and Holter parameters.

Overall, at the time of writing this protocol, the number of subjects/patients randomized in the clinical program was 113, of whom 101 to have been exposed to S201086/GLPG1972. The

studies conducted enrolled 83 healthy adult male subjects aged 18-50 years and 30 (male and female) adult OA patients aged 50-75 years.

In general, the treatment was well tolerated. Up to now, no Serious Adverse Reactions (SARs), overdose, interaction, medication errors, abuse/misuse, pregnancy and/or lactation cases were reported and no life-threatening events or deaths occurred. No SAEs related to special patient groups were reported.

No specific important risks have been identified for S201086/GLPG1972 at present. As with any new compound in early clinical development, cardiovascular safety, hepatic safety, biochemistry, hematology, coagulation and other laboratory safety parameters will be closely monitored throughout the clinical studies.

As there is limited clinical experience with S201086/GLPG1972 so far, the study drug should not be administered to subjects with renal or hepatic impairment.

#### **Pharmacokinetics**

S201086/GLPG1972 given as a single dose oral solution, from 60 to 2100 mg, in the fasted state was rapidly absorbed with a median time to maximum concentration range of 1-4 h and eliminated with an overall mean apparent half-life of 10 h in healthy subjects.

After q.d. dosing for 14 days in healthy subjects, S201086/GLPG1972 exposure (both Cmax and area under the concentration-time curve for the dosing interval [AUCT]) increased dose-proportionally over the entire dose range (300 to 1050 mg q.d.). Steady-state in S201086/GLPG1972 plasma concentrations was reached after 2 dosing days with a minimal accumulation. The excretion of unchanged S201086/GLPG1972 in urine over a 24 h period was less than 11% of the administered dose.

The PK parameters of S201086/GLPG1972 in patients with OA were not different from those observed in healthy subjects at the same dose level.

No food effect with the WG tablets of S201086/GLPG1972 (1.3- and 1.1-fold increase in  $C_{max}$  and area under the concentration-time curve from time 0 extrapolated to infinity  $[AUC_{0-\infty}]$ , respectively) was observed.

After 10 daily doses of S201086/GLPG1972 in healthy subjects, co-administration with midazolam, a sensitive cytochrome P450 type 3A4 (CYP3A4) substrate, led to a slight decrease in midazolam exposure when compared to midazolam alone. The apparent midazolam terminal half-life was slightly reduced. As a result, S201086/GLPG1972 is classified as a weak inducer of CYP3A4 (decrease in substrate exposure between 20 and 50%).

# Clinical pharmacodynamics

After a single administration of 300, 600, or 1050 mg of S201086/GLPG1972 in healthy subjects, no significant reduction of neoepitope ARGS levels *vs.* baseline was observed compared to placebo.

After dosing of 300, 600, or 1050 mg for 14 days, a significant reduction of ARGS levels vs. baseline was observed at Day 14 when compared to placebo. The mean average % reduction from time 0 to 24 h postdose (Eavg<sub>(0-24h)</sub>) increased with the dose, but there were no statistically significant differences between the 3 tested doses. More subjects achieved a % reduction vs.

baseline of at least 60% when receiving a higher dose of S201086/GLPG1972. However there was no statistically significant dose-effect. Neoepitope ARGS were also determined in predose samples at Days 1, 3, 4, 5, 6, 8, 10, and 14. A progressive reduction over time was observed reaching a maximum inhibition of 50-60% at Day 14.

After dosing of 100, 200 or 300 mg for 29 days in patients with OA, a statistically significantly higher reduction compared with placebo in neoepitope ARGS levels vs. baseline was observed. The values of mean % reduction vs. baseline were dose-dependent. Neoepitope ARGS levels went back to baseline 14 and 21 days post-last dose (Day 43 and 50), indicating that the target engagement is reversible.

# Rationale for study design

Recent literature provides strong evidence for a central role of ADAMTS-5 in OA and positions this enzyme as a key target for the discovery of DMOADs. GLPG1972 is a potent inhibitor of ADAMTS-5 which is capable to reach the joint cartilage upon oral administration and shows significant disease modification in 2 rodent surgery-induced OA models.

By virtue of these properties, it is expected that S201086/GLPG1972 would exert a particular benefit in patients with OA.

# Study Design

The study is a prospective, international, multiregional, multicenter, randomized ratio: 1:1:1:1, double-blind, placebo-controlled, dose-ranging study. The objectives of this study are to evaluate the efficacy and safety of 3 doses of S201086/GLPG1972 compared to placebo in patients with knee OA and the primary objective is to demonstrate the efficacy of at least one dose (among 3 doses) compared to placebo in reducing cartilage loss of the target knee in these patients.

The 52-week treatment duration was chosen in order to observe minimum natural cartilage degradation in the placebo arm and ensure a sufficiently long exposure to treatment allowing the demonstration of the activity of the drug, and to collect relevant safety data on S201086/GLPG1972.

# Study population

It is planned to randomize 852 patients (213 in each treatment arm). The target population will consist of patients diagnosed with knee OA based on the clinical and radiological criteria of the American College of Rheumatology (ACR) and classified as radiographic grade 2 or 3 of the Kellgren and Lawrence (KL) scale and grade 1 or 2 OARSI medial tibiofemoral joint space narrowing (JSN) (Altman et al., 2007). This population is likely to progress sufficiently to permit detection of cartilage loss as measured by cartilage thickness by quantitative magnetic resonance imaging (qMRI) (Lohmander et al., 2014); (Maschek, 2014)). This population is consistent with the recommendation of the current European Medicines Agency (EMA) guideline on clinical investigation of medicinal products used in the treatment of OA (CPMP/EWP/784/97 Rev.1, 2010) as well as OARSI recommendations for potential structure modifying drugs.

# Study primary outcome

X-ray provides an indirect measure of the cartilage thickness, however only calcified bone can be visualized. Measurement of joint space width (JSW) has some evidence for construct and predictive validity, with good reliability and responsiveness; however studies of at least 1 and probably 2 years duration will be required. The choice to use qMRI for the primary outcome was based on the fact that this technique provides objective quantitative assessment of morphology (thickness, volume, and area) and integrity (quality) of the articular cartilage (Conaghan, 2011). (Eckstein et al., 2015) showed an association between loss in medial tibiofemoral cartilage thickness on qMRI and radiographic and pain progression in OA. It is expected that qMRI of cartilage thickness of the central medial tibiofemoral compartment (cMTFC) will have the highest responsiveness, allowing for observing significant changes after one year of treatment.

# Choice of doses

The choice of doses (75, 150, and 300 mg daily) was based on pharmacokinetics and pharmacodynamics results in humans as well as data obtained in toxicological studies and pharmacological studies.

Moreover, the dose of 300 mg

was well tolerated in healthy subjects and up to 1 months of treatment in patients with OA (GLPG1972-CL-104). The lower dose of 75 mg/day is proposed in regard to estimations showing that exposures at this dose are sufficient to decrease ARGS level and are similar to those at which an effect on cartilage is observed in animal models.

The study will be conducted in compliance with the protocol, Good Clinical Practice (GCP), the ethical principles that have their origin in the Declaration of Helsinki and the applicable regulatory requirements.

The safety for use during pregnancy has not been established. No data have been generated in nursing women and no data are available on teratogenicity and excretion in milk. Therefore as precaution, women of child-bearing potential (WOCBP) must be excluded from clinical studies with S201086/GLPG1972.

## 3. STUDY OBJECTIVES AND PURPOSE

# **Objectives:**

The objectives of this study are to evaluate the efficacy and safety of 3 doses of S201086/GLPG1972 compared to placebo in patients with knee OA.

The primary objective of the study is to demonstrate the efficacy of at least one dose (among 3 doses) of S201086/GLPG1972 compared to placebo after 52 weeks of treatment in reducing cartilage loss measured by cartilage thickness using qMRI of the cMTFC of the target knee.

# The secondary objectives are:

To assess the safety and tolerability of 3 doses of S201086/GLPG1972.

To assess efficacy of 3 doses of S201086/GLPG1972 versus placebo after 52 weeks of treatment on:

- the proportion of "structural progressors\*" based on cartilage thickness using qMRI of the cMTFC of the target knee
- pain, function, and stiffness measured with WOMAC
- pain measured with a 100-mm visual analog scale (VAS)
- patient global assessment (PGA) of disease activity measured with 100-mm VAS
- reduction of cartilage loss measured by cartilage thickness using qMRI of the total tibiofemoral compartment (tTFC) of the target knee
- JSW measured by x-ray

\*defined as patient who had at least 8% cartilage loss in the cMTFC between baseline and W052.

To assess efficacy of 3 doses of S201086/GLPG1972 versus placebo after 28 and 52 weeks of treatment on bone area using qMRI of the medial femoral condyle surface of the target knee.

To assess the pharmacokinetics of S201086/GLPG1972 (and metabolite[s] if applicable).

To assess efficacy of 3 doses of S201086/GLPG1972 versus placebo after 52 weeks of treatment on analgesic consumption.

# Exploratory objectives are:



#### 4. STUDY DESIGN

This study is a phase 2, international, multi-regional, multicenter, randomized, double-blind, parallel-group, placebo-controlled, dose-ranging study of 52 weeks.

# 4.1. Endpoints

# The primary efficacy endpoint:

The change from baseline to W052 in cartilage thickness of the cMTFC of the target knee: qMRI.

# **Secondary efficacy endpoints:**

- Proportion of structural progressors\* at W052 based on cartilage thickness of the cMTFC of the target knee: qMRI
- The change from baseline to W052 in WOMAC total score and subscales scores of the target knee for pain, function, and stiffness
- The change from baseline to W052 in pain of the target knee: 100-mm VAS
- The change from baseline to W052 in PGA of disease activity of the target knee: 100-mm VAS
- The proportion of Outcome Measures in Rheumatology (OMERACT)-OARSI responders\*\* at W052: defined according to WOMAC and PGA
- The change from baseline to W052 in cartilage thickness of the tTFC of the target knee: qMRI
- The change from baseline to W028 and to W052 in bone area of the medial femoral condyle surface of the target knee: qMRI
- The change from baseline to W052 in JSW of the target knee: X-Ray
- Pain: analgesic consumption at every visit up to W052

- high improvement in pain or in function  $\geq 50\%$  and absolute change  $\geq 20$  or
- moderate improvement in at least 2 of the 3 following:
  - Pain  $\geq$  20% and absolute change  $\geq$  10
  - Function  $\geq 20\%$  and absolute change  $\geq 10$
  - Patient's global assessment  $\geq 20\%$  and absolute change  $\geq 10$ .

# Other secondary endpoints:

## Safety

The safety and tolerability assessed by the incidence of adverse events (AEs), changes over time in safety parameters, and incidence of abnormal safety parameters throughout the study.

#### Pharmacokinetics:

- Pharmacokinetics of S201086/GLPG1972 (and metabolite[s] if applicable)

<sup>\*</sup> defined as patient who had at least 8% cartilage loss in the cM- TFC between baseline and W052.

<sup>\*\*</sup> based on OMERACT-OARSI Initiative: Osteoarthritis Research Society International set of responder criteria for OA clinical trials revisited Pham et al. 2004. Defined according to WOMAC and patient's global assessment as a patient who had:

# Exploratory endpoints:



# 4.2. Experimental design

# 4.2.1. Study plan

The expected duration of patient participation will be 61 weeks maximum.

The study is divided into the following periods:

- An up to 5-week **screening period** without study treatment from screening visit (ASSE) to inclusion visit (W000). The screening period (up to 5 weeks) will allow enough time to obtain results from X-ray examination, ECG, laboratory examination, and to perform the baseline qMRI (before IMP intake).
- A double-blind treatment period of 52 weeks (from W000 to W052 visit). Eligible
  patients will be included and randomly assigned to receive 75 mg/day, 150 mg/day or
  300 mg/day S201086/GLPG1972, or matching placebo on a 1:1:1:1 ratio.
- A 2-week follow-up period (WEND) (from W052 or prematurely withdrawn to WEND): each patient must have a study end visit 2 weeks after completed or discontinued the study (definitely stopping study treatment), unless the patient withdraws consent.

The study plan is shown in Figure (4.2.1) 1.



The study initiation is defined as the date of the first visit of the first patient.

End of Trial is defined as the date of the last follow-up visit of the last patient (including a contact phone), or the date of the last contact attempt if the last patient is declared lost to follow-up.

# 4.2.2. Investigation schedule

Table (4.2.2) 1 describes the measurement of efficacy and safety assessed during the study.

Table (4.2.2) 1 - Investigation schedule

| | Screening<br>ASSE<br>(up to<br>5w) | Inclusion<br>W000 | W004<br>(+/-5d) | W008<br>(+/-5d) | W012<br>(+/-5d) | W020<br>(+/-7d) | W028<br>(+/-7d) | W040<br>(+/-7d)<br>(end of<br>morning or<br>afternoon<br>visit) | W052<br>(+/-7d) | Premature<br>withdrawal<br>(WD) | End of<br>study<br>WEND<br>(2w+/-<br>7d) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed consent | X | | | | | | | | | | |
| Inclusion /exclusion criteria | X | X | | | | | | | | | |
| Demographics and Height | X | | | | | | | | | | |
| Relevant medical / surgical history | X | | | | | | | | | | |
| Previous and concomitant treatments <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | X |
| IWRS <sup>2</sup> | X | X | X | X | X | X | X | X | | X | |
| Allocation of IMP | | X | X | X | X | X | X | X | | | |
| Compliance | | | X | X | X | X | X | X | X | X | |
| Efficacy measurements | | | | | | | | | | | |
| Primary | | | | | | | | | | | |
| qMRI (centralised) | | $X^3$ | | | | | X | | X | $X^4$ | |
| Secondary | | | | | | | | | | | |
| WOMAC [ePRO or paper (only if ePRO is unvailable)] | | X | | | X | | X | X | X | X | |
| VAS (pain) [ePRO or paper (only if ePRO is unavailable)] | X <sup>5</sup> | X | X | X | X | X | X | X | X | X | X |
| VAS (PGA) [ePRO or paper (only if ePRO is unavailable)] | | X | | | X | | X | X | X | X | |
| X-ray (centralized) | $X^6$ | | | | | | | | X | $X^7$ | |
| Analgesic consumption | | X | X | X | X | X | X | X | X | X | X |
| Safety measurements | | | | | | | | | | | |
| Adverse events <sup>8</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Physical examination including knees | X | X | X | X | X | X | X | X | X | X | X |
| Body weight | X | X | | | X | | X | | X | X | X |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X |
| Laboratory examinations: ✓ Hematology/biochemistry (central) ✓ Urinalysis (local) | X <sup>9</sup> | X | X | X | X | X | X | X | X | X | X |
| 12-lead ECG (centralized) | $X^{10}$ | $X^{10}$ | X | | | | X | | X | X | X |

| | Screening<br>ASSE<br>(up to<br>5w) | Inclusion<br>W000 | W004<br>(+/-5d) | W008<br>(+/-5d) | W012<br>(+/-5d) | W020<br>(+/-7d) | W028<br>(+/-7d) | W040<br>(+/-7d)<br>(end of<br>morning or<br>afternoon<br>visit) | W052<br>(+/-7d) | Premature<br>withdrawal<br>(WD) | End of<br>study<br>WEND<br>(2w+/-<br>7d) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Pharmacokinetics<br>Blood samples | | | X <sup>11</sup> | | X <sup>11</sup> | | X <sup>12</sup> | X <sup>13</sup> | X <sup>11</sup> | X <sup>11</sup> | |
| Diood samples | | | 21 | | 21 | | - 1 | - 21 | 21 | 21 | |
| | | Х | х | | X | | X | | X | X | x |
| | | X<br>X | X<br>X | | X<br>X | | X<br>X | | X<br>X | X<br>X | X<br>X |
| Optional measurements | | X<br>X | | | | | | | Х | | |

- 1. Previous treatments are all treatments stopped within 6 months before screening visit; concomitant treatments are treatments on-going at screening visit as well as new treatments initiated during the study
- IWRS connection to obtain patient's number (ASSE), randomization of patient following confirmation of inclusion eligibility, treatment allocation at W000, W004, W008, W012, W020, W028 and W040 and in case of premature withdrawal
- 3. The qMRI at baseline should be performed after getting results of screening criteria (lab, ECG, X-Ray) and before the first IMP intake
- 4. To be performed only if the previous qMRI (W000 or W028) is done  $\geq$  2 months before the premature withdrawal (time window between 2 qMRI)
- 5. Assessment of pain on both knees at screening visit only. Further assessments of pain will be performed on the target knee only
- 6. X-Ray on both knees at the screening visit only. Further assessment will be performed on the target knee only
- 7. To be performed only if the previous X-Ray (W000) is done more than 9 months before the premature withdrawal (time window between 2 X-Ray)
- 8. See section 8.9 for reporting methods
- 9. Including Hepatitis B, C and HIV. If a sample could not be analysed, or in case of unexpected abnormal lab results, resampling of the patient for a re-test is allowed once.
- 10. ECGs should be triplicate at ASSE and W000
- 11. Pre dose PK samples means that patients have to take their IMP at the site (after the PK-sample was drawn). At W052 or WD, no IMP should be taken.
- 12. Pre dose PK sample + one post dose PK sample (interval 2-4h post dose). Patients have to take their IMP at the site.
- 13. One post dose PK sample (interval 4-8h post dose). Patients have to take their IMP at least 4 hrs. before sampling and report the time of dosing to the study staff

For further practical details, methods of measurement are provided in sections 7, 8 and 9.

#### 4.3. Measures to minimize bias

- This is a double-blind, placebo-controlled study.
- The appearance and taste of the tablets will be the same for all study drugs, in order to protect the blinding with regard to the patients and the investigators.
- The treatment, S201086/GLPG1972 75 mg/day, 150 mg/day, 300 mg/day or matching placebo, will be assigned at randomized visit (W000) by a balanced (1:1:1:1), non-adaptive randomization, with stratification by zone (Japan, South Korea/Taiwan and Rest of the World).
- Treatment randomizations and allocations will be centralized by Interactive Web Response System (IWRS). The structure responsible for designing and constructing the randomization lists in blind will be the biostatistics department of I.R.I.S.



- The following measures (centralized) will be taken to optimize the homogeneity and the reliability of the study data:
  - MRI and X-Ray reading will be centralized. The CRO in charge of medical imaging management will organize the training and validation of sites participating in the study and will perform imaging quality controls and X-ray reading, and manage the MRI transfer to the central reading service provider.
  - o ECG reading and interpretation will be centralized throughout the study by a CRO. All study centers will be supplied with an ECG device by the CRO central reading,
  - Laboratory parameters will be assessed centrally by a CRO.
- Pain VAS, WOMAC if applicable and PGA VAS will be recorded using electronic patient reported outcome (ePRO).
- Samples for pharmacokinetic analysis will be sent to the central laboratory and transferred to the assay center. The assay center in charge of S201086/GLPG1972 measurement in biological matrices will be provided with the treatment codes so that only samples from patients being treated with S201086/GLPG1972 will be assayed (patients under active treatment).



# 4.4. Data and safety monitoring board

A Data and Safety Monitoring Board (DSMB) will be put in place in order to independently review the available safety data at regular pre-specified time points. The functioning of this DSMB is specified in a separate DSMB charter.
#### 5. INCLUSION OF PATIENTS

#### 5.1. Inclusion criteria

All patients included should present the following characteristics:

- 1a. Male patients or female patients of non-childbearing potential and not breastfeeding.

  Note: Female patients will be considered of non-childbearing potential if they are either surgically sterile (e.g. tubal ligation, hysterectomy) or postmenopausal (at least 12 consecutive months of amenorrhea in the absence of other biological or physiological causes AND 50 years of age or older).
- 2. Age between 40 to 75 years (both inclusive).
- 3. Body weight > 40 kg.
- 4. Body mass index (BMI)  $\leq 40 \text{ kg/m}^2$ .
- 5. Diagnosed for knee OA based on the clinical and radiological criteria of the ACR (documented diagnosis), *i.e.*:
  - a- Knee pain

b- and, at least one of the following:

- age more than 50 years
- morning stiffness < 30 minutes duration
- crepitus on active motion

*c- and,* presence of osteophytes

- 6. History of knee pain for at least 6 months and on the majority of days (> 50%) during the preceding month.
- 7a. Symptom severity defined by a pain  $\geq 40$  mm and  $\leq 90$  mm on a 100 mm VAS at screening and inclusion visits (at screening <u>both</u> knees should be assessed for pain and at least one knee should fulfill pain severity defined on this criterion). A knee not meeting the pain criteria at screening must not be eligible as target knee at inclusion.
- 8. Documented need for symptomatic as needed-treatment for OA in the target knee with systemic non-steroidal anti-inflammatory drugs (NSAIDs) and/or other analgesics
- 9b. Disease stage based on a fixed flexion weight-bearing X-ray of the target knee\* and central read out of:
  - a. Predominant medial compartment radiographic disease
  - b. KL grade 2 or 3
  - c. And OARSI grade 1 or 2 medial tibiofemoral joint space narrowing (JSN)

\*The target knee (right or left) to be followed-up throughout the study:

- If both knees fulfill the clinical screening criteria (as described in Section 5.1) and radiological inclusion criteria, the knee to be chosen should be the most severely affected knee on X-ray (higher KL score); in case of similar KL scores, the higher JSN score will be selected.
- If both knees display the same radiological scores, the knee to be chosen should be the most clinically painful one (Higher VAS score at screening).
- If both knees display the same radiological scores and are equally painful, the choice should be left to the investigator's discretion.
- 10. Informed consent obtained as described in section 13.3 of the protocol.

#### 5.2. Exclusion criteria

11. Unlikely to cooperate in the study.

- 12. Participation in another interventional study within 3 months before screening; participation in non-interventional registries or epidemiological studies is allowed.
- 13. Re-screened patient.
- 14. Patient unable to understand the study.
- 15. Poor compliance anticipated by the investigator.
- 16. Investigator or other study staff or related thereof who is directly involved in the conduct of the study.
- 17. Severe clinical knee malalignment according to the investigator.
- 18. Knee prosthesis already implanted (< 1 year) or not well-tolerated (contralateral side).
- 19. Knee prosthesis already foreseen within the study period (whichever side).
- 20. Hip prosthesis recently implanted (< 1 year) or foreseen within the study period (whichever side).
- 21a. Previous osteotomy on the inferior limbs (whichever side) other than intervention for hallux valgus with full clinical recovery after surgery.
- 22a. Any surgical operations on the target knee (arthroscopic and non-arthroscopic), other than diagnostic arthroscopy, within the 12 months prior to the screening visit or planned during the study period.
- 23a. Diagnostic arthroscopy of the target knee within the 6 months prior to the screening visit or planned during the study period.
- 24b. Other current or medical history of pathologies affecting the target knee such as: septic arthritis, inflammatory joint disease, gout, major chondrocalcinosis (pseudogout), Paget's disease of the bone, ochronosis, acromegaly, haemochromatosis, Wilson's disease, rheumatic symptoms due to malignancies, primary osteochondromatosis, osteonecrosis, osteochondritis dissecans, documented severe intra-articular knee injury (e.g. intra-articular fracture), hemophilia, etc.
  - Note: Patients with common risk factors for knee OA e.g. obesity, meniscectomy are <u>not</u> excluded.
- 25a. Patients with widespread chronic musculoskeletal pain of unclear etiology (*i.e.* functional somatic syndromes such as fibromyalgia, with or without previously documented diagnosis).
- 26. Chronic oral corticosteroid therapy within one month prior to enrolment into the study other than stable doses of  $\leq 7.5$  mg daily prednisolone or equivalent.
- 27a. Corticosteroid or hyaluronic acid intra-articular injections in the target knee in the previous 3 months.
- 28a. Chronic use of medications with and for MMP-inhibitory properties (*i.e.* Tetracycline or structurally related compounds) during the 3 months prior to the screening visit.
- 29a. Bisphosphonates, denosumab, teriparatide, strontium ranelate, romosozumab use (in oral or injectable form) in the previous 12 months.
- 30. Use of other unapproved drugs for osteoarthritis treatment during the 3 months prior to the screening visit.
- 31b. Chronic use of strong opioids and use of possible drug/drug interaction treatment during 7 days prior to the screening visit (section 6.6).
- 32a. Any contraindication to MRI according to local MRI guidelines, or the inability to undergo a knee MRI exam because of inability to fit in the scanner or knee coil. The presence of pacemaker or any other implanted electronic devices is considered a contraindication to MRI in this study (accommodations will not be made).
- 33a. Non-pharmacological standard of care for the target knee (physiotherapy, electrotherapy, *etc...*) <u>if initiated less than</u> 4 weeks before screening visit.
- 34. Severe or unstable disease of any type that could interfere with safety and efficacy assessments (e.g., uncontrolled cardiovascular, pulmonary, infectious, severe immune-

- deficiency, autoimmune, renal, hepatic, gastro-intestinal, endocrine, blood disorders) according to investigator's judgment
- 35. History of malignancy in the past 5 years, with the exception of: basal cell carcinoma, resected cutaneous squamous cell carcinoma in situ, prostate cancer in situ with a normal prostate-specific antigen post treatment, cervical carcinoma in situ, gastric cancer in situ, colon cancer in situ adequately treated with no significant progression over the past 2 years.
- 36. Class III or class IV Heart failure according to the New York Heart Association (NYHA) classification.
- 37a. Moderate to severe renal impairment; *i.e.*, estimated Glomerular Filtration Rate (GFR) < 45 mL/min/1.73 m<sup>2</sup> (Modification of the Diet in Renal Disease [MDRD] formula).
- 38b. The following abnormalities detected on a 12-lead ECG performed at screening visit of either rhythm or conduction (QT interval corrected for HR according to Fridericia's formula [QTcF] interval > 450 ms for males and > 470 ms for females, bradycardia with HR < 50 bpm, measured and stable PR-interval > 280 ms, or second (except Mobitz Type 1) or third degree Atrio-Ventricular Block and complete left branch block) as assessed by central reading.
  - Any other abnormalies are left to the investigator's judgment for final decision.
- 39. Known severe hepatic impairment (*i.e.*, cirrhosis, active liver disease) or known liver enzymes abnormalities such as:
  - a. Aspartate aminotransferase (AST) and/or ALT values > 2 x upper limit of normal (ULN)
  - b. Alkaline phosphatase (ALP)  $> 3 \times ULN$ ,
  - c. Total bilirubin > 1.5 x ULN (except in case of Gilbert syndrome)
- 40a. Positive for anti-human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBs), or anti-hepatitis C virus (HCV) antibodies with a positive test for HCV viral RNA or completion of antiviral HCV treatment ≤ 12 weeks before screening.
- 41. Severe malabsorption according to investigator's judgment.
- 42. Unexplained significant weight loss (> 10% of body weight within the last year).
- 43. Alcohol abuse or drug abuse or addiction according to investigator's judgment.
- 44b. Documented hypersensitivity to the active substance or to any of the excipients (e.g.: lactose).

## 5.3. Contraception

Within the frame of this study, as the effect of S201086/GLPG1972 on sperm in man is unknown, male clinical study patients and their female partners of child-bearing potential must use highly effective contraception (as described in the informed consent form) in combination with a barrier contraceptive to prevent pregnancy and to avoid the risk of exposure of the embryo or fetus during the study and up to 12 weeks after the last dose received.

Male patients agree to not donate sperm from the time of first study drug intake during the study and until 12 weeks after the last study drug intake.

## **5.4.** Discontinuation of the study

## 5.4.1. Premature discontinuation of the study or temporary halt

This study may be temporarily halted or prematurely discontinued at any time for any sufficient reasonable cause.

After having informed the national coordinators, the sponsor or the institutional review board (IRB)/independent ethics committee (IEC) or the Regulatory Agencies may terminate the study before its scheduled term. Two copies of the written confirmation will be dated and signed by the coordinators. The IRB/IECs and Regulatory Agencies will be informed according to local regulations.

If the study is prematurely discontinued, the patients still included in the study should be seen as soon as possible and the same assessments as described in Section 5.5 should be performed.

The premature withdrawal visit should be notified via IWRS (refer to investigation schedule Table (4.2.2) 1).

Under some circumstances, the investigator may be informed of additional procedures to be followed in order to ensure that adequate consideration is given to the protection of the patient's interests.

In case of study suspension (temporary halt), the study may resume once concerns about safety, protocol compliance, data quality are addressed and satisfy the Sponsor, the DSMB, the IRB/IEC and Regulatory Agencies.

## 5.4.2. Discontinuation of the study in the event of objective reached

Not applicable

#### 5.5. Patient withdrawal

#### 5.5.1. Withdrawal criteria

A patient may be discontinued from the clinical study at any time without the patient's consent if the investigator or sponsor determines that it is not in the best interest of the patient to continue participation. In such case, the reason for withdrawal will be documented in the source documents, and the patient will complete the premature withdrawal (WD) visit and follow-up visit (WEND) for safety assessments.

Treatment with IMP must be discontinued by the investigator and the patient must be withdrawn from the clinical study (preferably after discussion with the monitor, who may consult and must inform the sponsor's study physician if applicable) for any of the following conditions:

- Life-threatening adverse event (AE) or a SAE that places the patient at immediate risk.
- Confirmed pregnancy
- The following ECG and/or laboratory parameter abnormalities:
  - QTcF > 500 ms or a delta > 60 ms over baseline value (inclusion) on at least two separate ECGs
  - Increase in liver function tests:
    - 1. ALT or AST > 8x ULN (discontinue the treatment immediately),
    - 2. ALT or AST > 5x ULN for more than 2 weeks (a decision to stop the study drug should be taken after a confirmed retest),
    - 3. ALT or AST > 3x ULN and (total bilirubin > 2x ULN or international normalized ratio [INR] > 1.5),
    - 4. ALT or AST > 3x ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%),

5. Presence of evocative clinical symptoms such as jaundice.

In general, an increase of serum aminotransferase (AT) to > 3xULN should be followed by repeat testing preferably within 48h after laboratory results are received by the investigator of all four of the usual serum measures (ALT, AST, ALP, and TBL) to confirm or not the abnormalities.

Based on the re-test results, it should be determine together with monitor if the discontinuation criteria are confirmed. If confirmed, the patient must be withdrawn from the clinical study.

In any case of liver toxicity, additional investigations are needed (such as: assessment of alcohol or recreational drugs intake, hepatitis infection, etc...)

- Any AE or any condition incompatible with continuation of the investigational medicinal product (IMP) according to the judgment of the investigator

The investigator may also decide to stop the treatment with IMP (preferably after consultation with the sponsor's study physician if applicable) for any of the following reasons:

- Use of concurrent therapy that was not permitted
- Noncompliance with the IMP treatment including overdose
- Noncompliance with the clinical study procedures
- Serious or severe AEs
- Worsening of disease condition, which in the investigator's opinion needs an alternative treatment approach not being covered in the clinical study

Patients will be informed prior to clinical study entry that they are allowed to withdraw from the clinical study. At any time and for any reason, a patient's participation in the clinical study may terminate at his/her request without prejudice to his/her future medical care. The patient will be encouraged to share the reason(s) for withdrawal so this can be documented in the source documents, and to complete the WD visit and follow-up visit (WEND) for safety assessments, but will not be obliged to do so.

The sponsor has the right to terminate the clinical study at any time in case of safety concerns or if special circumstances concerning the IMP or the company itself occur, making further treatment of patients impossible. In this event, the investigators and relevant authorities will be informed of the reason for clinical study termination.

Information to be collected during the last visit of these patients is listed in Section 5.5.2. These follow-up assessments are included to ensure the efficacy and safety evaluation of all patients who received the IMP.

#### 5.5.2. Procedure

- In the case of premature withdrawal from the study due to an AE, the investigator must make every effort to collect the information relating to the outcome of the event. If necessary, the information will be collected afterwards (see Section 8.9). This information is recorded in that part of the eCRF which concerns adverse events. If the investigator cannot collect the information from a visit, every effort must be made ensuring the follow-up of the patient.
- If the study is stopped / IMP is discontinued as a result of an event requiring immediate notification, the procedure described in Section 8.9.2.4 has to be implemented.

The actions to be taken after the IMP discontinuation are described in Section 6.5.

# 5.5.3. Lost to follow-up

When the investigator has no news of the patient, he/she must make every effort to contact him/her or a person around him/her (phone calls, letters including registered ones, etc....), to establish the reason for the discontinuation of IMP and to suggest the patient comes to an end-of-study visit. If all these attempts to contact the patient fail, the investigator can then declare the patient "lost to follow-up". The investigator should document all these attempts in the corresponding medical file.

#### 6. TREATMENT OF PATIENTS

## 6.1. Study products and blinding systems

#### 6.1.1. Products administered

IMPs (also mentioned as study drug in this protocol) in this study are the study drug S201086/GLPG1972 (at dose of 75 mg, 150 mg or 300 mg) and matching placebo.

The study drug S201086/GLPG1972 will be provided as film-coated tablets for oral use, containing 75 mg S201086-1/G504572 each (S201086-1/G504572 is the compound code for S201086/GLPG1972). The placebo will be provided as matching film-coated tablets for oral use.

The oral tablets will be packaged in polyvinylchloride (PVC)/aluminum (Alu) blisters, which are grouped in a carton box.

Table (6.1.1) 1 provides a description of the IMP(s).

S201086/GLPG1972
75 mg

Pharmaceutical form
Film-coated tablet
Film-coated matching tablet
Unit dosage
Appearance, color
Composition\*

S201086/GLPG1972
Film-coated matching tablet
orange
orange

**Table (6.1.1) 1 – Description of the IMPs** 

Table (6.1.1) 2 provides a description of the packaging of the IMP

#### Table (6.1.1) 2 – Description of packaging

Number of units of the pharmaceutical form per primary 28 tablets of S201086/GLPG1972 75 mg and/or packaging placebo per blister

Number of primary packaging per secondary packaging 5 blisters per small box

The number of TU boxes which will be dispensed to patient at each visit will be different depends on visit: W000, W004, W008 (1 box), W0012, W020 (2 boxes), W028, W040 (3 boxes).

The labeling of packages complies with the regulatory requirements of each country involved in the study.

#### 6.1.2. IMP management

Treatment units will be supplied from the « Unité d'Appui Clinique », Les Laboratoires Servier Industrie, 905 route de Saran, 45520 Gidy, France.

IMP receipt, dispensing according to the experimental design of the study (for the description of dispensing methods, refer to section 6.3), accountability and collection are the responsibility of the investigator, delegated person of the study team and/or pharmacist of the medical institution.

<sup>\*</sup>excipient with known effect

Destruction of the IMP is the responsibility of the sponsor and the person responsible for the IMP management.

Remaining treatments (used and unused IMPs) will subsequently be collected and stored according to the local procedures and requirements, by the person responsible for the IMP management.

A certificated destruction will be performed according to standard modalities for that class of product and the attestation must be sent to the sponsor. The practical procedures for destruction of unused IMP will be defined by the sponsor and adapted to the center. An IMP collection and destruction form will be completed before the shipment of IMP to destruction. Destruction of IMP may be possible (after drug accountability and sponsor authorization) when the product has been used, has expired or after at least the last visit of the last treated patient. The IMP should be stored in a secure area with restricted access.

IMP management will be verified on a regular basis by the study monitor.

The investigator and/or the pharmacist of the medical institution and/or a designated person from their study team must complete all the documents provided by the sponsor concerning IMP management in real time (therapeutic unit tracking form or an equivalent document, therapeutic unit (TU) label collection form). Therapeutic unit tracking form, or an equivalent document, is the source document to be completed.

The investigator and/or the pharmacist of the medical institution should only use the IMP provided for the patients involved in the study.

All defects or deterioration of IMPs or their packaging are to be reported to section 8.9.2.4.2 (special situations), and to the IWRS. The investigator will notify of all complaints set out by a patient (appearance...).

In the event of advanced return of IMPs to the sponsor (batch recall), the sponsor will prepare an information letter intended for the investigator and/or pharmacist of the medical institution. This letter will be sent by the person locally responsible for the study to each study centre. On receipt of the letter, the investigator and/or the pharmacist will identify the patients in possession of the IMP at the moment the incident becomes known, by using, among other tools, the therapeutic unit tracking form, or an equivalent document, and will contact them immediately.

#### 6.1.3. Management of blinding systems

The patient treatment code should only be broken in case of emergency where the further treatment of the patient is dependent on the treatment he or she is receiving.

In the cases where the blind needs to be broken by the investigators for imperative justified medical reason, a centralized decoding system integrated with the IWRS is adopted for the study. No sealed envelopes will be used.

The centralized decoding procedure will be performed by the investigators by contacting the IWRS. The system is available 24 hours a day, 7 days a week. The procedure to be followed by the investigator or authorized person is detailed in the IWRS manual.

If IWRS is not available, the helpdesk of the IWRS will be contacted by phone.

For all countries except US:

Additionally, decoding will be possible by calling the Emergency Phone Number of I.R.I.S. (+33 1 55 72 60 00) 7/7d and 24/24h) to reach the Emergency Permanency that will have a sealed decoding list not available to other I.R.I.S. personnel during the study. A code list will be kept in a safe place by the I.R.I.S. Clinical Supplies Coordinating Department and will be accessible to any person authorized to unblind.

#### 6.2. IMPs administered

No IMPs will be administered during screening and follow up periods.

From the day of inclusion until the W052 Visit, the patient will take four (4) tablets orally once a day with a glass of water preferably in the morning (at the same time), corresponding to:

- S201086/GLPG1972 75 mg/day: 1 tablet of 75 mg + 3 matching tablets of placebo,
- S201086/GLPG1972 150 mg/day: 2 tablets of 75 mg + 2 matching tablets of placebo,
- S201086/GLPG1972 300 mg/day: 4 tablets of 75 mg,
- 4 matching tablets of placebo.

During visits, the IMP will be taken at the site (during the visit with the newly dispensed TU box) except for W040 (for PK sampling) where IMP will be taken <u>at home</u> prior to the visit and the exact intake time will be reported, and W052 (the end of treatment visit), where no new TU box is dispensed.

# 6.3. IMPs dispensing

Investigator and/or the pharmacist of the medical institution and / or a designated person from their study team will use the IWRS, as described in the IWRS manual, to perform the following actions:

- To create the patient number at ASSE visit,
- To randomize the patient and allocate the treatment at W000 visit,
- To allocate treatment at W004, W008, W012, W020, W028, and W040 visits,
- To register "Premature withdrawal" if applicable.

The IWRS manual will detail all instructions for randomization and allocation of the treatment. The IMP is dispensed at W000, W004, W008, W012, W020, W028 and W040 visits.

The detachable portion of the label on the IMP box must be stuck by the investigator or a delegated person on an IMP label collection form or on the prescription/IRS form where the IMPs are dispensed by a pharmacist or designee.

#### **6.4.** IMP compliance

The number of tablets dispensed and the number of tablets returned by the patient are to be counted by the investigator or a designated person from his/her team and recorded in the electronic case report form and therapeutic unit tracking form, or an equivalent document.

If the patient did not bring back all blisters dispensed at the previous visit, the investigator must estimate the number of IMP units taken by the patient since the previous visit, by questioning him/her and must document the reason in the medical file.

Compliance will be assessed at each visit or in case of premature withdrawal.

The compliance will be assessed from the method described above and from the questioning of the patient.

#### 6.5. Discontinuation of the IMP

After the discontinuation of the IMP, the patients' treatment is left to the physician's discretion. As the study drug is not on the market, it will not be available.

Specific rules may be followed in some countries according to local regulation.

#### 6.6. Previous and concomitant treatments

Previous treatments are all treatments stopped within 6 months before screening visit; concomitant treatments are treatments ongoing at screening visit as well as new treatments initiated during the study.

Previous and concomitant treatment (prescriptions or over-the-counter medications) must be reported in the eCRF. Reported information will include a description of the type of the drug, treatment period, dosing regimen, route of administration and its indication. Any change in dosage must also be reported in the Concomitant Treatments eCRF section. Data on concomitant medication will be collected up to the last follow-up visit, even after withdrawal of a patient.

Table (6.6) 1 - Treatment prohibited during the study (non-exhaustive list)

# Type of treatment

| Symptomatic drugs | Oral | Chronic corticosteroids > 7.5 mg/d Prednisolone or equivalent |
|---|---|---|
| | Intra-articular injection in the target knee | Corticosteroids Hyaluronic acid |
| Experimental or unapproved treatments | Intra-articular injection in the target knee | e.g. amniotic cytokines, platelet-rich plasma |
| Drugs with a potential effect on cartilage | | e.g. Chronic use of tetracycline or structurally related compounds |
| Drugs with an effect on subchondral bone | Oral or injection | Bisphosphonates Denosumab Teriparatide Strontium ranelate Romosozumab |



Table (6.6) 2 – Treatment authorized during the study with particular conditions for use

# Type of treatment

| Symptomatic oral drugs | Glucosamine (sulphate or others) Chondroitin sulfate | Under condition of stable dosing for at least 3 months prior to W000 (inclusion) visit and stable dosing for at least 3 months prior W052 visit |
|---|---|---|
| | Diacerein | |
| | Avocado/soybean unsaponifiables | |
| Intra-articular injection of drugs (except target knee) | Corticosteroids | Allowed if ≥ 1 month prior to W000 (inclusion) visit and ≥ 1 month prior to W052 visit |
| Strong opioids | Short-acting, Morphine sulfate Codeine sulfate Oxycodone Hydrocodone (with or without aspirin, acetaminophen, ibuprofen) Hydromorphone Meperidine hydrochloride Fentanyl citrate transmucosal Oxymorphone Long-acting Buprenorphine Morphine sulfate sustained release Fentanyl transdermal Levorphanol tartrate Oxycodone HCL controlled release Methadone | |
| Non-pharmacological standard of care in the target knee | Physiotherapy, electrotherapy, etc | Allowed if initiated $\geq \frac{4}{\text{weeks}}$ prior to W000 (inclusion) visit and if initiated $\geq 4$ weeks prior to W052 visit |

Table (6.6) 3 – Treatment authorized during the study

| | Type of treatment |
|-------------------------|-------------------------------------------------|
| NSAIDs/other analgesics | As needed in the context of OA standard of care |

#### 7. ASSESSMENT OF EFFICACY

#### 7.1. Efficacy measurements

Efficacy measurements performed during the study are indicated in Table (4.2.2) 1.

#### 7.2. Methods and measurement times

#### 7.2.1. Medical imaging

Before their participation in the study CL2-201086-002/GLPG1972-CL-201, all centers will receive a specific training/qualification coordinated by the CRO in charge of medical imaging management (MRI qualification protocol). In addition, this CRO will be in charge of:

- o Imaging (MRI and X-ray) reception and quality control (QC),
- o X-ray reading
- o MRI transmission to the MRI reader, and
- o Imaging (MRI and X-ray) data transfer to the Sponsor.

The aim is to ensure standardized and appropriate acquisition and assessments of medical imaging.

#### o qMRI:

MRI of the target knee will be performed after the participant's eligibility (Lab, ECG, X-Ray) has been confirmed and before W000 (inclusion), W028 and W052 visits, and at the withdrawal visit (WD) if the time window between WD and the previous qMRI (W000 or W028) is  $\geq 2$  months.

If a patient withdraws from the study after at least 2 months after W000 or after W028, every effort should be made to schedule for a final qMRI acquisition in order to have a final measurement available.

All MRI images will be transmitted to the medical imaging management CRO. If a scheduled MRI fails QC, one repeat MRI is allowed (for additional MRI repeat the approval of the sponsor is needed). After passing QC, MRI images will be sent to the medical image analysis service provider for central reading and analysis (coded data). The MRI acquisition technique, image tracking and management and reading methods will be described in specific documents that will be available before the center initiation visit.

In addition, ONE of the first 3 patients (preferably 3<sup>rd</sup>) per site will be scanned twice with repositioning at both baseline (W000 visit) and at W052 visit (or if applicable WD visit in case of the patient discontinues the study) for quantitative measurement to calculate the within study variability.

# o Radiography (X-ray):

A weight-bearing X-ray of the knee (both knees at ASSE and the target knee at W052) will be performed in all patients. If a patient withdraws from the study > 9 months after initial X-ray, every effort should be made to schedule for a final X-ray of the target knee in order to have a final measurement available.

All X-rays will be transmitted to the medical imaging management CRO. If a scheduled X-ray fails QC, one repeat X-ray is allowed (for each knee at the screening visit and for the target knee at every visit when X-ray is scheduled) (for additional X-ray repeat the approval of the

sponsor is needed). After passing QC, images will be analyzed by central readers (coded data). A scoring according to the KL grading and OARSI JSN grading will be performed on both knees at screening visit (ASSE) only and transmitted within a specific short timeframe to the investigational site in order to include or exclude the patients. The minimal JSW will be measured using a semi-automated computerized method according to a standardized method detailed by a separate technical protocol.

The X-ray acquisition technique, images tracking and management and reading methods will be described in specific technical documents that will be available in time before the center initiation visit.

# 7.2.2. WOMAC for measurement of pain, function and stiffness (Appendix 2)

The WOMAC index score will be assessed on site at W000, W012, W028, W040, W052 and if applicable at the withdrawal visit (WD).

WOMAC (version LK3.1, copyright holder Nicholas Bellamy) is a questionnaire designed to assess health status and health outcomes in patients with osteoarthritis of the knee. The questionnaire contains 24 questions targeting areas of pain (5 questions), stiffness (2 questions) and physical function (17 questions). The questionnaire is self-administered by the patient and can be completed in less than 5 minutes. It refers to the 48h period prior to assessment and will be completed before the clinical examination, preferably in the waiting room.

The WOMAC will be recorded by:

- ePRO. The questionnaire will be explained to the patient by the investigator (or a delegate person) and will be filled in by patients during the visits on an electronic device (e-PRO). Data entered by the patient will be sent to a central database via a secured transfer,
- paper, in case of unavailability of ePRO, and a copy will be sent to ePRO provider for data entry and the original kept by investigator.

# 7.2.3. VAS for pain intensity (Appendix 3)

After the choice of the target knee to be followed throughout the study has been made by the investigator and explained to the patient, the pain intensity will be assessed during each visit (ASSE on both knees and W000, W004, W008, W012, W020, W028, W040, W052 and WEND on the target knee and if applicable at the withdrawal visit (WD)) by the patient him/herself by marking the level of pain on a 100-mm VAS. The scale should be completed before the clinical examination, with the patient being asked on the level he would rate the pain felt in the selected knee within the last 48 hours on a VAS.

The pain VAS will be recorded by:

- ePRO. The questionnaire will be explained to the patient by the investigator (or a delegate person) and will be filled in by patients during the visits on an electronic device (e-PRO). Before starting, the patient will need to complete training first. Data entered by the patient will be sent to a central database via a secured transfer.
- Paper, in case of unavailability of ePRO, and a copy will be sent to ePRO provider for data entry and the original kept by investigator (paper version on Appendix 8).

## 7.2.4. VAS for Patient Global Assessment of disease activity (PGA) (Appendix 4)

The PGA VAS will be assessed during the following visits: W000 (inclusion), W012, W028, W040, W052 and if at the withdrawal visit (WD) by the patient him/herself by marking the level of "Considering all the ways in which your knee osteoarthritis affects you, please rate on this 100 mm scale how well you are doing today" on a 100 mm VAS.

The PGA VAS will be recorded by:

- ePRO solution. The questionnaire will be explained to the patient by the investigator (or a delegate person) and will be filled in by patients during the visits on an electronic device (e-PRO). Before starting, the patient will need to complete training first. Data entered by the patient will be sent to a central database via a secured transfer.
- paper, in case of unavailability of ePRO, and a copy will be sent to ePRO provider for data entry and the original kept by investigator (paper version on Appendix 8).

# 7.2.5. Analgesic consumption

Drug analgesic consumption of the patient will be recorded on the eCRF at W000 (inclusion), W004, W008, W012, W020, W028, W040, W052, WEND and if applicable at the withdrawal visit (WD).

#### 8. SAFETY MEASUREMENTS

All AEs and other situations relevant to the safety of the patients must be followed up and fully and precisely documented in order to ensure that the sponsor has the necessary information to continuously assess the benefit-risk balance of the clinical study.

#### **8.1.** Specification of safety parameters

Safety measurements performed during the study are indicated in Table (4.2.2) 1.

The safety will be assessed based on of the following information:

- AEs
- Physical assessment including knees
- Vital signs
  - Assessment with automatic blood pressure monitoring of:
    - Systolic blood pressure (SBP) (mmHg)
    - o Diastolic blood pressure (DBP) (mmHg)
    - o Pulse Rate (bpm)
  - Body weight (kg)
- 12-lead-ECG: qualitative and quantitative ECG findings (HR, PR, QRS, QT, QTcF and [RR] intervals) (equipment supplied by the CRO in charge of ECG central reading). At ASSE and W000, ECG will be in triplicate.
- Biological laboratory examinations
  - O Blood biochemistry includes ALT, AST, gamma glutamyltransferase (GGT), ALP, lactate dehydrogenase (LDH), creatinine phosphokinase (CPK), total and conjugated bilirubin, total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL), triglycerides, total protein, albumin, creatinine (with calculation of the GFR), urea, glucose, uric acid, sodium, potassium, chlorides, calcium, bicarbonate, C-reactive protein (CRP)
  - Hematology includes hemoglobin, hematocrit, erythrocytes, differential white cell count (leucocytes, basophils, eosinophils, neutrophils, monocytes, lymphocytes in absolute values), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular volume (MCV), platelets
  - Urinary dipstick (PH, red blood cells, white blood cells, glucose, proteins, ketones, bilirubin).

#### 8.2. Methods and measurement times

**Vital signs** will be evaluated at ASSE, W000, W004, W008, W012, W020, W028, W040, W052, WEND and if applicable at the premature withdrawal visit (WD). Blood pressure will

be measured with automatic blood pressure monitor and will preferably be measured on the same arm (in case of equipment is supplied by the sponsor, equipment has to be used).

**Body Weight** will be evaluated at ASSE, W000, W012, W028, W052, WEND and if applicable at the premature withdrawal visit (WD).

**Physical assessment including knees** performed at ASSE, W000, W004, W008, W012, W020, W028, W040, W052, WEND and if applicable at the premature withdrawal visit (WD).

**ECG** will be performed at ASSE, W000, W004, W028, W052, WEND and if applicable at the premature withdrawal visit (WD). ECG device will be the same for all centers and will be supplied by the CRO in charge of ECG central reading. The ECG device should be used only for the study. All ECGs will be sent anonymized to the CRO for central reading.

Even if the 12-lead **ECG** reading and interpretation will be centralized, a local assessment of ECG is necessary for detection of medical urgencies and must be enclosed in the source data. For Per Protocol inclusion/exclusion/withdrawal criteria, central reading reports overrule local reading.

**Laboratory examinations** will be performed at: ASSE, W000, W004, W008, W012, W020, W028, W040, W052, WEND and if applicable at the premature withdrawal visit (WD).

Urinary dipstick will be performed locally. In case of clinically significant abnormal urinary dipstick result, the investigator or his/her delegate will perform a quantitative urinalysis that will be done locally.

Laboratory results will be assessed by the investigator for clinical significance. In case of clinical significance, AEs/SAEs should be reported.

Laboratory tests analysis will be subcontracted to a central laboratory. The details for sampling, handling, storage and shipping of the samples will be described in a separate manual.

For the laboratory tests, it is recommended for patients to be fasted (if possible) and that patients should avoid very vigorous physical exercise or strenuous physical exertion during the 72 hours immediately prior to each blood-draw.

Additional safety investigations can be performed if deemed necessary should the investigator have a suspicion of any pathology requiring urgent medical intervention.

#### 8.3. Definition of Adverse events

An AE is defined as any untoward medical occurrence in a patient participating in a clinical study, whether or not there is a causal relationship with the IMP and/or experimental procedures, occurring or detected from the date the patient signs the information and consent form, irrespective of the period of the study (periods without administration of the IMP (e.g. run-in period) are also concerned).

An AE can therefore be:

- any unfavorable and unintended sign (including an abnormal finding from an additional examination such as lab tests, X-rays, ECG, ...) which is deemed clinically relevant by the investigator,
- any symptom or disease,

- any worsening during the study of a symptom or a disease already present when the patient entered the study (increase in frequency and/or intensity), including the studied pathology,

and detected during a study visit or at an additional examination or occurred since the previous study visit.

# Of note:

- Any **hospitalization for social reasons**, **educational purpose** (*e.g.* learning of diabetes management by the patient) or routine check-up should not be considered as an adverse event and should not be reported in the eCRF.
- The following procedures, whether planned before the study or not, whether leading to a hospitalization or not, should be reported in the specific page "Procedures not subsequent to an adverse event" of the eCRF:
  - therapeutic procedures related to a non-aggravated medical history (e.g. cataract extraction not due to an aggravation of the cataract during the study, hemodialysis sessions related to a renal insufficiency not aggravated during the study),
  - prophylactic procedures (e.g. sterilization, wisdom teeth removal),
  - comfort procedures (e.g. cosmetic surgery),
  - control procedures of a pre-existing condition without aggravation (e.g. colonoscopy to control the remission of colon cancer).

#### 8.4. Definition of Serious adverse events

Any AE that at, any dose:

- results in death,
- is life-threatening<sup>(1)</sup>,
- requires inpatient hospitalization or prolongation of existing hospitalization,
- results in persistent or significant disability/incapacity<sup>(2)</sup>,
- is a congenital anomaly/birth defect<sup>(3)</sup>,
- is medically significant<sup>(4)</sup>.
- (1) Life-threatening in this context refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.
- (2) Disability/incapacity in this context refers to any event that seriously disrupts the ability of the patient to lead a normal life, in other words leads to a persistent or permanent significant change, deterioration, injury or perturbation of the patient's body functions or structure, physical activity and/or quality of life.
- (3) Congenital anomaly or birth defect refers to the exposure to the IMP before conception (in men) or during pregnancy that resulted in an adverse outcome in the child.
- (4) Any event that might not be immediately life-threatening or result in death or hospitalization, but might jeopardize the patient or might require intervention to prevent one of these outcomes (for example: edema or allergic bronchospasm that required intensive treatment at home, blood dyspraxia, convulsions that do not result in hospitalization, or development of drug dependence or drug abuse). The investigator should exercise his/her scientific and medical judgment to decide whether or not such an event requires expedited reporting to sponsor.

#### **8.5.** Definition of special situations

- Pregnancy of participant or partner of male participant in the study
- Other special situations:

## • Abuse of study drug

The persistent or sporadic, intentional excessive use of the study drug, which is accompanied by harmful physical or psychological effects.

## • Misuse of study drug

Situations where the study drug is intentionally and inappropriately used not in accordance with the authorized product information.

# • Drug interaction with study drug

A situation in which the study drug interacts with another drug when both are administered together.

# • Food interaction with study drug

A situation in which food interacts with the study drug.

#### • Medication error

An unintended failure in the drug treatment process that leads to, or has the potential to lead to, harm to the patient.

# • Occupational exposure

An exposure to the study drug as a result of one's professional or non-professional occupation.

#### Overdose

The administration of a quantity of the study drug given per administration or cumulatively, which is above a certain dose as defined in the protocol (>4 tablets/day).

# • Product complaint or quality defect of study drug

Complaints arising from potential deviations in the manufacture, packaging, or distribution of the study drug.

## 8.6. Definition of Adverse event of special interest

At the time of writing this study protocol, no AE of special interest have been defined.

# 8.7. Definition of Events requiring an immediate notification (ERIN)

An event must be **notified immediately** (*i.e.* without delay and within 24 hours at the latest) to the sponsor if it is:

- a serious adverse event,
- a pregnancy and other special situations.

# 8.8. Classification of an adverse event (seriousness, severity, causality)

It is important that the investigator gives his/her own opinion regarding the **seriousness**, the **severity** of the event as well as the **causal relationship** between an adverse event and the test drug. This evaluation must be assessed by the investigator and reported in the AE page of the eCRF. In addition, the sponsor will be responsible for the evaluation the **expectedness** of the event (See Section 8.9.3).

<u>The Seriousness</u> should be evaluated according to international guidance (see definition Section 8.4, in accordance with ICH Topic E2A and DIRECTIVE 2001/20/EC OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of 4 April).

<u>The Severity</u> of AEs should be graded using the Common Terminology Criteria for Adverse Events (CTCAE) version (v.5). If a CTCAE criterion does not exist, the investigator should use the grade or adjectives: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (lifethreatening) or Grade 5 (fatal) to describe the maximum intensity of the AE. For purposes of consistency with the CTCAE, these intensity grades are defined in the table below.

#### **Grading of Adverse Event Severity**

| Grade | Adjective | Description |
|---|---|---|
| Grade 1 | Mild | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| Grade 2 | Moderate | Local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL* |
| Grade 3 | Severe | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL** |
| Grade 4 | Life-<br>threatening | Urgent intervention indicated |
| Grade 5 | Fatal | Death-related AE |

<sup>\*</sup> Activities of Daily Living (ADL) Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

For AEs associated with laboratory abnormalities, the event should be graded also on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality. This is upon the investigator's assessment.

<u>The causal relationship</u> to the study drug or to the experimental procedure must be assessed when reporting the AE in the AE page of the eCRF. Only cases ticked "related" by the investigator, or judged by the sponsor as having a reasonable suspected causal relationship to the study drug, will be considered as suspected Adverse Drug Reaction.

The following decision table will be used by the investigator to report the causality assessment between the reported event and the investigational medicinal product.

<sup>\*\*</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

| Definitions | Relationship to report<br>in eCRF |
|---|---|
| <b>Unrelated:</b> No relationship between the AE and the administration of study drug; related to other etiologies such as concomitant medications or patient's clinical state. | NOT-RELATED |
| <b>Unlikely:</b> Event or laboratory test abnormality, with a time to drug intake that makes a relationship improbable (but not impossible). Disease or other drugs provide plausible explanations. | |
| <b>Possible:</b> Event or laboratory test abnormality, with reasonable time relationship to drug intake which could also be explained by disease or other drugs. Information on drug withdrawal may be lacking or unclear. | |
| <b>Probable:</b> Event or laboratory test abnormality, with reasonable time relationship to drug intake. Event unlikely to be attributed to disease or other drugs. Response to withdrawal is clinically reasonable and rechallenge not required. | RELATED |
| <b>Certain:</b> Event or laboratory test abnormality, with plausible time relationship to drug intake which cannot be explained by disease or other drugs. Response to withdrawal is plausible (pharmacologically, pathologically). Event definitive pharmacologically or phenomenologically ( <i>i.e.</i> , an objective and specific medical disorder or a recognized pharmacological phenomenon). Rechallenge satisfactory, if necessary. | |

#### 8.9. Reporting procedures

## 8.9.1. Time frame for adverse event reporting

Any event meeting the above mentioned definitions (see sections 8.3 to 8.7) must be reported to the sponsor on an <u>AE form</u> if it occurred:

- before the first intake of the study drug, for event associated with any procedure/condition required by the study protocol: procedure (Imaging, etc.), change or withdrawal of previous/concomitant treatment relating to the conditions of the protocol.
- at any time after the first intake of the **study drug** up to the patient's last study visit for all events.
- after the patient's last study visit:
  - up to 30 calendar days after the last study drug intake for all ERIN, regardless of the supposed role of the research (IMP or experimental procedure).
  - irrespective of the time of onset after the end of the study in case of serious adverse event <u>related</u> to the research (IMP or experimental procedure).

Of note, events occurring between the signature of the informed consent and the first administration of the study drug for which the investigator does not consider an association with any procedure/condition required by the study protocol must be reported as <u>medical</u> history in the dedicated form of the e-CRF.



## 8.9.2. Responsibilities of the investigator

For any adverse event and special situation mentioned above the investigator must:

- Note in the patient's medical file the date on which he/she learned of the event (at a follow-up visit or a telephone contact with the patient or a third person, ...) and any other relevant information which he/she has learned of the event,
- Assess the event in terms of seriousness, severity and causality,
- **Report the event to the sponsor** using the AE form (in case of ERIN, the reporting should be done immediately),
- **Document** the event with additional useful information,
- Ensure the **follow-up** of the event,
- **Fulfill his/her regulatory obligations** to the Regulatory Agencies and/or to the IRB/IEC, in accordance with local regulations.

Moreover, the investigator must report to the sponsor and/or to the IRB/IEC and/or to the Regulatory Agencies in accordance with the local regulation, any new information that might materially influence the benefit-risk assessment of the study drug or that would be sufficient to consider changes in the study drug administration or in the overall conduct of the clinical investigation.

#### 8.9.2.1. Documentation of the event

The investigator must ensure that all events are well documented. In particular for ERIN, he/she should provide the sponsor, as they become available, with anonymized copies of the documents which provide additional useful information, such as hospital admission reports, reports of further consultations, laboratory test reports, reports of other examinations aiding diagnosis, or the autopsy report, if autopsy is performed.

#### 8.9.2.2. Follow-up of adverse events

The investigator must ensure that follow-up of the patient is appropriate to the nature of the event, and that it continues until resolution if deemed necessary.

Any change in terms of diagnosis, severity, seriousness, measures taken, causality or outcome regarding an adverse event already reported must documented in the "Adverse event" page previously created for the event (e-CRF).

If the adverse event has not resolved at the patient's final visit in the study (WEND), the patient will be followed up suitably until satisfactory resolution (*i.e.*, value back to baseline value or stabilization). Additional information on a patient's AE after resolution can be added at the investigators' discretion to the AE page of the eCRF and to the source documents, until closing of the eCRF for that patient. Thereafter, the investigator can continue to follow-up the patient if deemed necessary, however no further information will be reported into the eCRF.

If the follow-up of the patient is not done by the investigator him/herself (hospitalization, followed by a specialist or the patient's general practitioner, ...), the investigator will do everything to establish/maintain contact with the person/department in charge of follow-up of the patient.

# **8.9.2.3.** Recording Methods in the e-CRF

Adverse events must be documented on the AE page of the e-CRF.

In case of chronic disease:

- if the disease is known when the patient enters in the study, only worsening (increased frequency and/or intensity of the episodes/attacks) will be documented as an adverse event,
- if the disease is detected during the study and if repeated episodes enable diagnosis of a chronic disease, the episodes will be grouped on the «Adverse Event» page previously created for the event (e-CRF) which will clearly describe the diagnosis.

## 8.9.2.4. Procedure for an event requiring an immediate notification (ERIN)

Any ERIN (SAE, pregnancy and other special situation) must be reported within 24h of knowledge.

#### 8.9.2.4.1. Serious Adverse Event

In case of Serious Adverse Event (SAE), the investigator must:

- Immediately after being informed of this event, fill in the patient's medical file as well as the «Adverse Event» page of the e-CRF according to the general instructions available in the e-CRF, without waiting for the results of the clinical outcome or of additional investigations. When data will be submitted into Inform, an e-mail will be immediately and automatically sent to the sponsor.
- Provide the sponsor (person designated in the contact details provided in the investigator's study file), as they become available, with anonymized copies of the documents which provide additional useful information,
- Fulfil his/her regulatory obligations to the Regulatory Agencies and/or to the IRB/IEC, in accordance with local regulations.

If an adverse event initially non-serious worsens and becomes serious (ERIN), this must be reported **immediately** on an "Adverse event" page of the e-CRF.

In case the e-CRF is unavailable when the investigator was informed of the ERIN, he/she should:

- **Immediately** fill in a paper "Adverse event" page:
  - For serious event on a paper "Adverse event Initial information" page,
  - For event initially non-serious on a paper "Adverse event Initial information" page, and the worsening leading to seriousness on a paper "Adverse event Additional information" page,
- Immediately send them by fax (or e-mail) to the person(s) designated in the contact details provided in the investigator's study file or outside working hours, the 24-hour phone line is +33.1.55.72.60.00.
- As soon as the e-CRF becomes available, the investigator should enter these data in the «Adverse Event» page of the e-CRF.

## 8.9.2.4.2. Special situations

- In case of a special situation not associated with an AE (except pregnancy), the investigator should report it on a "special situation not associated with an adverse event" page of the e-CRF.
- In case of a special situation associated with an AE, the investigator should report it on an «Adverse Event» page of the eCRF.
  - In case the e-CRF is unavailable when the investigator was informed of a special situation, he/she should, within 24 h of knowledge, complete a paper "Special situation not associated with an adverse event" or "Adverse event" form, send it by fax (or e-mail) to the person(s) designated in the contact details provided in the investigator's study file or outside working hours, the 24-hour phone line is +33.1.55.72.60.00.
  - As soon as the e-CRF becomes available, the investigator should enter these data in the «Special situation not associated with an adverse event » or «Adverse event » page of the e-CRF.
- In case of deliberate or accidental IMP overdose, general measures to maintain or support the basic vital functions should be taken, if deemed necessary. No experiments have been performed to determine a specific antidote to IMP.
- If a special situation concerns a person around the study participant, the investigator should not report this on eCRF but must fill in the paper-based "Special Situations Report form" and send it within 24 h of knowledge by fax (or e-mail) to the person(s) designated in the contact details provided in the investigator's study file.

## **8.9.2.4.3. Pregnancy**

If pregnancy concerns a patient or a partner of a patient, the investigator immediately after being informed of this event **must fill in the paper-based "Pregnancy Report form"** and send it within 24 h of knowledge by fax (or e-mail) to the person(s) designated in the contact details provided in the investigator's study file.

The outcome of pregnancies must be reported. A follow-up contact should be scheduled at the expected time of delivery.

Summary of special situations including pregnancy:

| Type of situation | Where to report it? |
|---|---|
| Special situation with AE concerning | "Adverse event" form of eCRF |
| a participant | |
| Special situation without AE | "Special situation not associated with an adverse |
| concerning a participant | event" form of eCRF |
| Special situation concerning a person | Paper form called "Special situations report form" |
| who is not a participant | |
| Pregnancy concerning the participant | Paper form called "Pregnancy Report form" |
| or his partner | |

## 8.9.3. Responsibilities of the sponsor

In accordance with international guidelines, the assessment of the seriousness and the causality of AE are usually made by the investigator but falls also under sponsor's duties. The causality and the seriousness may be upgraded (but never downgraded) by the sponsor. If the assessments of the investigator and the sponsor are different, both will be reported in the clinical study report.

The sponsor is responsible for ensuring that all suspected unexpected serious adverse reactions are reported to Regulatory Agencies and Ethics Committees.

In addition, the sponsor is responsible for determining whether an AE is **expected or unexpected**. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the Safety Information section of Investigator's Brochure.

Independently of the regulatory obligations of the investigator, the sponsor must report the pharmacovigilance data to the appropriate Authorities and to all the investigators involved, according to the requirements stated in ICH Good Clinical Practice guidelines and local regulations.

The concerned Authorities will be notified as soon as possible by the sponsor of the DSMB recommendations if any, where relevant for the safety of patients (*i.e.* modification or termination of the study).

# 8.10. Responsibilities of data safety monitoring board

In accordance with the DSMB charter and the rules for DSMB functioning (refer to section 12.4 of the clinical study protocol), the DSMB is responsible for reviewing the safety data on a regular basis, and providing written recommendations to the Sponsor regarding the conduct of the study (modification or termination).

# 9. OTHER ASSESSMENTS NOT SPECIFICALLY RELATED TO EFFICACY OR SAFETY

#### 9.1. Pharmacokinetics

S201086/GLPG1972 concentration (and metabolite[s] if applicable) will be analyzed. Plasma analyses for S201086/GLPG1972 will be performed by the assay centre using a validated analytical method.

For all patients, blood samples (5 mL/time-point) will be collected in W004, W012, W028, W040, W052 and if applicable at the withdrawal visit (WD) to determine S201086/GLPG1972 (and metabolite[s] if applicable) plasma concentrations:

- At W004, W012, W052 visits and if applicable at the withdrawal visit (WD), one (1) time-point will be collected (pre-dose PK sample). At these visits, the patient takes the IMP at the site (at W052 or WD, no IMP should be taken).
- At W028 visit, a pre dose and a post dose sample will be collected. The pre dose sample
  is taken at the site. Thereafter the patient takes the IMP at the site. The post dose sample
  is taken 2-4 hours after IMP intake.
- At W040 visit, a post dose sample will be collected. The post dose sample is taken 4-8
  hours after IMP intake. This visit is likely to be scheduled in the afternoon. Patients take
  their IMP at least 4 h before sampling and report the time of dosing to the study staff.

It is also important that for days at which a PK-sample is taken, patients document/report the time of dosing on the previous day (or estimation).

The sampling conditions and handling details will be described in a specific technical document that will be available in time before the center initiation visit.







# 9.3. Assessment related to exclusion criteria

The following assessments will be performed on screening samples: biological laboratory examinations with Hepatitis B and C, and HIV.

#### 10. STATISTICS

#### 10.1. Statistical analysis

The Statistical Analysis Plan and associated templates for Tables, Listings and Graphs, will be written just after finalizing the protocol and definitively completed before breaking the blind of the study These specifications will detail the implementation of all the planned statistical analyses in accordance with the main characteristics stated in the protocol.

## 10.1.1. Endpoints

## 10.1.1.1. Efficacy endpoints

# 10.1.1.1.1. Primary efficacy endpoint

The primary efficacy endpoint is the change from baseline to W052 in cartilage thickness in the cMTFC assessed by qMRI on the target knee (centralized reading).

# 10.1.1.1.2. Secondary efficacy endpoints

The secondary efficacy endpoints are:

- The proportion of "Structural progressors" at W052. A "structural progressors" is defined as a patient who had an 8% cartilage loss in cMTFC between baseline and W052.
- The change from baseline to W052 in WOMAC total score and subscales scores for pain, function and stiffness.
- The change from baseline to W052 in pain in the target knee measured with a 100-mm VAS.
- The change from baseline to W052 in patient global assessment of disease activity measured with 100-mm VAS.
- The proportion of OMERACT-OARSI responders at W052. A responder is defined according to WOMAC and PGA as a patient who had a high improvement in pain or in function  $\geq 50\%$  and absolute change  $\geq 20$  or, improvement in at least 2 of the 3 following:
  - Pain  $\geq 20\%$  and absolute change  $\geq 10$
  - Function  $\geq 20\%$  and absolute change  $\geq 10$
  - Patient's global assessment  $\geq 20\%$  and absolute change  $\geq 10$ .
- The change from baseline to W052 in cartilage thickness of the total tibiofemoral compartment of the target knee using qMRI (centralized reading).
- The change from baseline to W028 and to W052 in bone area of the medial femoral condyle surface of the target knee using qMRI (centralized reading).
- The change from baseline to W052 in JSW of the target knee measured by x-ray (centralized reading).
- Pain: Analgesic consumption: at every visit up to W052

#### 10.1.1.2. Safety endpoints

The safety endpoints are:

- For AEs:
- The number of AEs, the number and percentage of patients reporting at least one AE. The AE are:

- Serious adverse events (SAE) during the study, according to the investigator or sponsor opinion.
- Emergent adverse event (EAE) under treatment. The definition of EAE will be provided in the Statistical Analysis Plan.
- For clinical laboratory evaluation:
  - The value at baseline, value at each post-baseline visit under treatment and last post-baseline value under treatment; as well as the change from baseline to each post baseline visit under treatment and to last post-baseline value under treatment.
  - The number and percentage of patients with at least one high/low emergent abnormal value under treatment, according to the laboratory reference ranges and to the cut-offs for PCSA values for discrete parameters, except for urinary parameters.

The clinical laboratory evaluations are biochemistry, haematology and urinary parameters.

- For vital signs and clinical examination:
  - The value at baseline, value at each post-baseline visit under treatment and last post-baseline value under treatment; as well as the change from baseline to each post baseline visit under treatment and to last post-baseline value under treatment.
  - The number of emergent relevant decreases/increases, number and percentage of patients with at least one emergent relevant decrease/increase.

The vital signs and clinical examination parameters are the body weight (kg), BMI (kg/m²), SBP (mmHg), DBP (mmHg) and pulse rate (bpm).

- For ECG parameters:
  - The value at baseline, value at each post-baseline visit under treatment and last post-baseline value under treatment; as well as, for continuous parameters the change from baseline to each post baseline visit under treatment and to last post-baseline value under treatment.

The electrocardiogram parameters are, the presence of clinically significant ECG abnormalities (yes/no), the heart rate (bpm), the QRS duration (msec), the PR interval (msec), the QT interval (msec), the QTcF – Fridericia's correction formula interval and the RR interval (msec).

Moreover, other endpoints will be derived from the QTcF – Fridericia's correction formula interval's electrocardiogram parameter: the values and changes from baseline in classes, considering threshold defined in ICH E14 (i.e.,  $\leq$  450, ]450; 480]; ]480; 500] and > 500 ms for values, and  $\leq$  30, ]30; 60] and > 60 ms for changes).

- Other safety endpoints:

Special situations (defined in section 8.5) not associated with an AE.





# 10.1.1.4. Other endpoints

Not applicable.

## 10.1.1.5. Pharmacokinetics endpoints

Plasma concentrations of S201086/GLPG1972 (and those of metabolite[s] if applicable) will be documented with descriptive statistics (mean, median, standard deviation, minimum and maximum) at each time-point and each dose for trough plasma concentration (C<sub>trough</sub>) values.

S201086/GLPG1972 (and metabolite[s] if applicable) plasma concentration measurement will be used in order to build a population pharmacokinetics model. This analysis will provide pharmacokinetic parameters and their associated variability. The influence of covariates will be investigated. The pharmacokinetic analysis will be the object of separate data analysis plan (DAP) and report.



## 10.1.2. Analysis sets and subgroups / Treatment groups

## 10.1.2.1. Analysis sets and subgroups

## - Modified Randomised Set (mRS):

The modified Randomised Set (mRS) will be constituted of all included patients to whom a therapeutic unit was randomly assigned using IWRS. The mRS will be used for efficacy analyses. Patients will be analysed according to the randomised treatment.

#### - Safety Set (SS):

The Safety Set (SS) will be constituted of all patients having taken at least one dose of IMP. The SS will be used for safety analyses. Patients will be analysed according to treatment actually received at inclusion.

No formal subgroup analysis is planned for this study.

# 10.1.2.2. Treatment groups

Treatment groups considered will be S201086/GLPG1972 75 mg, S201086/GLPG1972 150 mg, S201086/GLPG1972 300 mg and placebo.

#### 10.1.3. Statistical methods

#### 10.1.3.1. General considerations

## 10.1.3.1.1. Multiplicity issues

In order to take into account the multiplicity of comparisons associated with the primary objective of the study (demonstration of superiority of at least one S201086/GLPG1972 dose as compared to placebo on the primary efficacy endpoint); a Dunnett's procedure will be used for the primary analysis. More details on the strategy defined for handling multiplicity issues are provided in Section 10.1.3.3.

For secondary endpoints, the same strategy as the one use for primary analysis will be used for handling multiplicity issues for doses comparison and no adjustment to control the type I error for multiple endpoints will be used.

## 10.1.3.1.2. Handling of missing data

For the primary analysis, a mixed-effects model for repeated measures approach will be used. In this model, two post-baseline time-points will be considered: W028 and W052. From one patient to another, possible distinct situations of remaining missing data have been identified, justifying different statistical treatments.

For patients with only one missing post-baseline measurement, missing data will not be imputed and handled through MMRM. As a reminder, MMRM analysis use all available data, including subjects with partial data (i.e., with missing data) in order to derive an estimate of the treatment effect without filling in the missing items (Mallinckrodt & al., 2013).

For patients for which no post-baseline measurement will be collected for the primary endpoint (regardless the timing of discontinuation), as they cannot be considered through the MMRM, a MI procedure will be used to impute the missing evaluations as a prior step. This approach allows considering that patients will keep the benefit of the randomized treatment after study discontinuation.

Sensitivity analyses will be performed in order to assess the robustness of the primary analysis results to the handling of missing data method by considering MI, Pattern Mixture Model (PMM) placebo-based imputation, tipping point method and observed cases (Mallinckrodt & al., 2013) detailed in Section 10.1.3.3.1.

More details on the strategy defined for handling missing data are provided in Section 10.1.3.3.

#### 10.1.3.1.3. Statistical elements

#### 10.1.3.1.3.1. Descriptive statistics

The following descriptive statistics will be provided depending on the nature of considered data:

- Discrete data: number of observed values, number and percentage of patients per class.
- Continuous data: number of observed values, mean and standard deviation, median, first and third quartiles, minimum and maximum.

#### 10.1.3.1.3.2. Estimations and statistical tests

The type I error of the statistical tests will be set at 5% (two-sided situation), which is consistent with the objective of demonstrating the superiority of S201086/GLPG1972 versus placebo (one-sided situation at 2.5%).

The treatment effect will be estimated as well as its accuracy: estimate of the difference, standard error of the estimate and two-sided 95% confidence interval of the estimate.

When formal comparison between treatment groups is performed, the two-sided p-value associated with the treatment effect will also be provided.

#### 10.1.3.2. Study patients: Disposition, baseline characteristics and follow-up

Demographic data and other baseline characteristics such as prognostic factors and baseline value of endpoints will be described by treatment group, to assess their comparability, by treatment group and with the overall in the mRS.

Disposition of patients, including reasons for withdrawal, protocol deviations, extent of exposure and treatment compliance, as well as concomitant treatments will be described in the mRS. Extent of exposure and treatment compliance will also be described in the SS.

The time to patient discontinuation and to premature IMP withdrawal will be described in the mRS, using a Kaplan-Meier analysis in order to assess the drop-out pattern between the treatment groups; as well as withdrawn and completed patients' characteristics in the mRS.

## 10.1.3.3. Efficacy analysis

## 10.1.3.3.1. Primary efficacy endpoint

## **10.1.3.3.1.1.** Primary analysis

## Main analysis strategy:

In order to meet the primary objective of the study, the efficacy of at least one dose of S201086/GLPG1972 as compared to placebo after 52 weeks of treatment in reducing cartilage loss in patients with knee OA will be assessed from the change from baseline to W052 in cartilage thickness as measured in the medial central tibiofemoral compartment on the target knee, in patients of the mRS. A restricted maximum likelihood (REML)-based, mixed-effects model for repeated measures approach (so called Mixed-effects Model for Repeated Measures – MMRM) using all longitudinal observations at each post-baseline visit (W028) (Mallinckrodt & al., 2013) will be used (main analysis). The MMRM as a primary analysis will assume that patients would keep the benefit of the randomized treatment after study discontinuation. A

missing data handling will be used (according to section 10.1.3.1.2) for this analysis. The treatment comparisons associated with the primary analysis will be the contrasts between each dose of S201086/GLPG1972 and placebo at the change from baseline to W52. Analysis will include the fixed, categorical effects of treatment, regions (Asia and Rest of the World), time and treatment-by-time interaction, as well as the continuous, fixed covariates of baseline, time-by-baseline interaction.

The analysis will fit an unstructured covariance matrix, and the assumptions underlying the model will be checked.

The consistency of the results between the Asian-region population and the non-Asian-region population (respectively between Japanese population and non-Japanese population) will be evaluated on primary endpoint, according to the Method 2 defined in Ministry of Health Labor and Welfare Notification (MHLW) Notification "Basic principles on Global Clinical Trials". Treatment effect estimates and confidence intervals will be provided, for each dose, in Asianregion population and non-Asian-region population (respectively between Japanese population and non-Japanese population). In case of a statistically significant overall treatment effect (in favor of S201086/GLPG1972) at a considered dose, the results will be considered consistent if the observed treatment effects in Asian-region and non-Asian-region (respectively between Japanese population and non-Japanese population) patients are favor S201086/GLPG1972.

#### Sensitivity analyses:

To assess the robustness of the analysis results towards the method of handling missing data, a similar procedure will be repeated according to the following variations:

- considering the multiple imputation method for all missing values,
- considering analysis is restricted to patients of the mRS having a non-missing value at W052 for the primary endpoint,
- considering the pattern mixture model, placebo based imputation for each missing data (including patients with an early discontinuation and without any post baseline value for the primary endpoint),
- considering the tipping point method for all missing values, using a single three-way analysis of covariance (ANCOVA) model with treatment and regions as fixed, categorical effects, as well as baseline as continuous fixed covariate. The assumptions underlying the model will be checked.

## 10.1.3.3.1.2. Secondary analyses

For each treatment group, descriptive statistics will be provided for the primary endpoint (in terms of value at each visit and change from baseline to each post-baseline visit), overall and by regions.

## 10.1.3.3.2. Secondary efficacy endpoints

For the proportion of "structural progressors" and proportion of OMERACT-OARSI responders at W052, the difference between each S201086/GLPG1972 dose and placebo will be studied in patients of the mRS, considering a multiple imputation for handling all missing data and using a logistic model, including the fixed, categorical effects of treatment, regions (Asia and Rest of the World), as well as the continuous, fixed covariates of baseline.

The difference between each S201086/GLPG1972 dose and placebo will be studied in patients of the mRS, on continuous secondary efficacy endpoints at W052, with the same strategy as the main analysis of the primary endpoint: multiple imputation for patients without any post-baseline value followed by a MMRM using all the longitudinal observations at each post-baseline visit. Analysis will include the fixed, categorical effects of treatment, regions (Asia Rest of the World), visit and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline, visit-by-baseline interaction.

For the change from baseline to W052 in JSW and the change from baseline to W028 in bone area, the difference between each S201086/GLPG1972 dose and placebo will be studied in patients of the mRS at W052 (respectively W028), considering a multiple imputation method for handling all missing data at W052 (respectively W028), and using an ANCOVA. Analysis will include the fixed, categorical effects of treatment, regions (Asia, US and Rest of the World), as well as the continuous, fixed covariate of baseline.

For analgesic consumption, number and percentage of patients by treatment reported will be provided, overall and by treatment group.

For each treatment group, descriptive statistics will be provided for all secondary endpoints (in terms of value at each visit and change from baseline to each post-baseline visit for continuous endpoint), overall and by regions.

## 10.1.3.4. Safety analysis

#### **10.1.3.4.1.** Adverse events

Number of events, number and percentage of patients reporting at least one event, presented by system organ class and preferred term (depending on the analysis), will be provided for SAEs and EAEs over the study.

EAEs will be described according to the seriousness, the intensity, the relationship, the action taken regarding the IMP, the requirement of added therapy, the outcome and the time to onset.

Of note, the seriousness and the relationship to the IMP of the adverse event correspond to the investigator opinion or, in case of events upgraded by the sponsor for seriousness or for causality in case of SAE, to the sponsor opinion.

#### **10.1.3.4.2.** Clinical laboratory evaluation

The following analyses will be performed, depending on the nature of considered endpoints (*i.e.*, quantitative or qualitative):

- Descriptive statistics on value at baseline, on value at each post-baseline visit under treatment, on last post-baseline value under treatment and, if applicable, on change from baseline to last post-baseline value under treatment.
- Number and percentage of patients with at least one high/low emergent abnormal value under treatment, according to the laboratory reference ranges and to the cut-offs for PCSA values.
- Laboratory parameters classified (number and percentage of patients in each class) according to these reference ranges and cut-offs, and using shift tables from baseline to the worst (high and/or low) values under treatment.

## 10.1.3.4.3. Vital signs, clinical examination and other observations related to safety

## 10.1.3.4.3.1. Vital signs and clinical examination

Blood pressure, pulse rate, body weight and BMI will be described, in terms of value at baseline, value at each post-baseline visit under treatment and last post-baseline value under treatment; as well as in terms of change from baseline to each post baseline visit under treatment and to last post-baseline value under treatment.

Number of emergent relevant decreases/increases, number and percentage of patients with at least one emergent relevant decrease/increase, based on SBP, DBP, pulse rate and weight will be provided.

#### 10.1.3.4.3.2. Electrocardiogram

ECG parameters will be described, in terms of value at baseline, value at each post-baseline visit under treatment and last post-baseline value under treatment; as well as, for quantitative endpoints, in terms of change from baseline to each post baseline visit under treatment and to last post-baseline value under treatment. Moreover values and changes form baseline of corrected QT interval will be described in classes, considering thresholds defined in ICH E14 (i.e.,  $\leq$  450, ]450; 480], ]480; 500] and > 500 ms for values, and  $\leq$  30, ]30; 60] and > 60 ms for changes).

ECG abnormalities will be described.

# 10.1.3.4.3.3. Special situations not associated with an AE

Special situations not associated with an AEs will be described in the mRS.

## 10.1.3.5. Exploratory analysis


# 10.1.4. Interim analysis

Not applicable

# 10.2. Determination of sample size

The determination of the sample size was performed considering the change from baseline to W052 in cartilage thickness in the cMTFC, expressed in mm and measured by qMRI.

The objective is to demonstrate that at least one S201086/GLPG1972 dose is superior to placebo in the mRS, based on a two-sided Dunnett test for multiple comparisons. The Dunnett test is used in order to maintain the experiment wise type I error at 5% (two-sided setting).

Two hundred and thirteen (213) patients per treatment group will provide a minimal power of approximately 70% to conclude for at least one dose that S201086/GLPG1972 is superior to placebo if the true difference is 0.0825 mm for at least one dose, assuming a standard deviation of 0.30 mm (Lohmander et al., 2014).

# 11. DIRECT ACCESS TO SOURCE DATA / DOCUMENTS

The investigator will allow the monitors, the persons responsible for the audit, the representatives of the IRB/IEC, and of the Regulatory Agencies to have direct access to source data / documents.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

#### 12.1. Study monitoring

Clinical site monitoring is conducted to ensure that the rights and well-being of human patients are protected, that the reported trial data are accurate, complete, and verifiable, and that the conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with applicable regulatory requirement(s).

- Monitoring for this study will be performed by the structure mentioned in a separate document (section 1).
- Details of clinical site monitoring are documented in a clinical monitoring plan (CMP) or similar document. The CMP describes in detail who will conduct the monitoring, at what frequency monitoring will be done, at what level of detail monitoring will be performed, and the distribution of monitoring reports.
- Independent audits may be conducted to ensure monitoring practices are performed consistently across all participating sites and that monitors are following the CMP.

# 12.1.1. Before the study

The investigator will allow the monitor to visit the site and facilities where the study will take place in order to ensure compliance with the applicable protocol requirements.

Training sessions may be organized for the investigators and/or instruction manuals may be given to the investigators.

# 12.1.2. During the study

The investigator will allow the monitor to:

- review of the study site's processes and procedures,
- verify appropriate clinical investigator supervision of study site staff and third party vendors,
- inspect the site, the facilities and the material used for the study,
- meet all members of his/her team involved in the study,
- consult the documents relevant to the study,
- have access to the electronic case report forms (*i.e.* access to an analogic phone line or his/her computer) and/or to the e-PRO service provider's database,
- check that the electronic case report forms/e-PRO have been filled out correctly,
- directly access source documents for comparison of data therein with the data in the electronic case report forms and/or to the e-PRO service provider's database,
- verify that the study is carried out in compliance with the protocol and local regulatory requirements.

The study monitoring will be carried out at regular intervals, depending on the recruitment rate and / or the investigation schedule, and arranged between the investigator and monitor.

All information dealt with during these visits will be treated as strictly confidential.

#### 12.2. Computerized medical file

If computerized medical files are used the following requirements apply.

The computerized medical file must:

- Be validated to ensure accuracy, reliability, consistent intended performance, and the ability to discern invalid or altered records
- Have the ability to generate accurate and complete copies of records
- Be ready retrievable and accurate throughout the records retention period
- Make use of secure, computer-generated, time-stamped audit trails
- Be accessible by the study monitor

If the computerized medical files do not fulfil these requirements the computerized medical files including updates or changes need to be printed, numbered, signed, and dated. All printed medical files (and changes therein) should be made available to the monitor during each site visit.

# 12.3. Audit - Inspection

The investigator should be informed that an audit may be carried out during or after the end of the study.

The investigator should be informed that the Regulatory Agencies may also carry out an inspection in the facilities of the sponsor and/or the study centers. The sponsor will inform the investigators concerned immediately upon notification of a pending study centers inspection. Likewise, the investigator will inform the sponsor of any pending inspection.

The investigator must allow the representatives of the Regulatory Agencies and persons responsible for the audit:

- to inspect the site, facilities and material used for the study,
- to meet all members of his/her team involved in the study,
- to have direct access to study data and source documents,
- to consult all of the documents relevant to the study.

If the computerized medical file is considered as not validated, the investigator undertakes to provide all the source-documents and the print-outs of the medical files of the patients and, if the computer system used allows, the record of the changes made during the study.

If the computerized medical file is considered as validated, the investigator undertakes to:

- give access to the representatives of the Regulatory Agencies and persons responsible for the audit to the computerized medical files of all patients,
- provide the print-outs of the changes made during the study, if the tracking of the changes made to the medical files cannot be accessed in the computer.

#### 12.4. Supervisory committees

DSMB recommendations will be forwarded to the IRB/IEC/ Regulatory Agencies only if relevant for the safety of patients.

According to the "Guideline on data monitoring committees" (Guideline CHMP/EWP/5872/03 Corr., 27 July 2005) and "Establishment and Operation of Clinical Trial Data Monitoring Committees" (FDA guidance, March 2006), the decision to set up of a DSMB should take into account the study population as well as the study duration. The present study takes place in patients aged between 40 and 75 years with knee osteoarthritis. As this vulnerable population (include aged patients) will be exposed to study treatment for up to 52-weeks, the set-up of a DSMB is justified in order to detect any potential harm to patients as early as possible.

All along the study, in order to ensure patients' safety, the DSMB will be responsible for a follow up of the patients by a periodical review of patients' data, especially adverse events. The DSMB will be provided with the information on study treatment by the authorized person of the Servier's Clinical Supplies Unit. The DSMB will treat all data as strictly confidential and will not disclose them to anyone else than members of the DSMB.

Details of the role and organization of the DSMB are detailed in a separate DSMB charter.

#### 13. ETHICS

# 13.1. Institutional Review Board(s)/Independent Ethics Committee(s)

The study protocol, the "Patient information and consent form" document, the list of investigators document, the insurance documents, the Investigator's Brochure of administered IMPs will be submitted to (an) IRB(s)/IEC(s) by the investigator(s) or the national coordinator(s) or the sponsor in accordance with local regulations.

The study will not start in a centre before written approval by corresponding IRB/IEC(s) has been obtained, the local regulatory requirements have been complied with, and the signature of the clinical study protocol of each contractual party involved has been obtained.

# 13.2. Study conduct

The study will be performed in accordance with the ethical principles stated in the Declaration of Helsinki 1964 (see Appendix 1) with the GCP and with the applicable regulatory requirements.

#### 13.3. Patient information and informed consent

In any case, the patient (and/or his/her legal representative, when required) must be informed that he/she is entitled to be informed about the outcome of the study by the investigator.

The investigator (or designee) is to collect written consent from each patient before his/her participation in the study. Prior to this, the investigator (or designee) must inform each patient of the objectives, benefits, risks, and requirements imposed by the study, as well as the nature of the IMPs.

The patient will be provided with an informed consent form in clear, simple language. He/she must be allowed ample time to inquire about the details of the study and to decide whether or not he/she wishes to participate.

One original informed consent form must be completed, dated, and signed by the patient and the investigator (or designee). The patient will be given a copy of the signed original informed consent form.

If the patient is unable to read, an impartial witness should be present during the entire informed consent collection process. The patient must give consent orally and, if capable of doing so, complete, sign, and personally date the informed consent form. The witness must then complete, sign and date the form together with the person responsible for collecting the informed consent.

Note that each patient's privacy is protected under the Health Insurance Portability and Accountability Act (HIPAA) privacy and security rules (for US only). The privacy rule requires appropriate safeguards to protect the privacy of personal health information, and sets limits and conditions on the uses and disclosures that may be made of such information without patient authorization. The rule also gives patients the rights over their health information, including rights to examine and obtain a copy of their health records, and to request corrections. The security rule requires appropriate administrative, physical and technical safeguards to ensure the confidentiality, integrity, and security of electronic protected health information.

#### 13.4. Modification of the information and consent form

Any change to the information and consent form constitutes an amendment to this document and must be submitted for approval to the IRB/IEC(s), and if applicable to the Regulatory Agencies.

A copy of the new version of the information and consent form in the language(s) of the country will be given in the amendment to the "Patient Information and consent form".

Such amendments may only be implemented after written approval of the IRB/IEC has been obtained and compliance with the local regulatory requirements, with the exception of an amendment required eliminating an immediate risk to the study patients.

Each patient affected by the amendment or an independent witness must complete, date and sign an original of the new version of the information and consent form together with the person who conducted the informed consent discussion. He/she will receive a copy of the signed original amendment to the information and consent form.

#### 14. DATA HANDLING AND RECORD KEEPING

#### 14.1. Source data

Source data and source documents of the center should be clearly identified in a specific, detailed and signed document before the beginning of the study.

The following documents are considered as source documents:

- Notes in the medical file (including nurse files)
- Therapeutic Unit Tracking Form (TUTF)
- Report/images (e.g. laboratory, ECG, MRI, X-Ray, etc.)
- VAS (pain) and VAS (PGA) recorded by e-PRO or paper (only if ePRO is unavailable)
- WOMAC recorded by e-PRO or paper (only if ePRO is unavailable)
- Requisition form (e.g. PK)

# 14.2. Study data

A 21 CFR Part 11-compliant electronic data capture system is going to be used for this study. An electronic case report form (eCRF) is designed to record the data required by the protocol and collected by the investigator.

The e-CRF will be produced by I.R.I.S. in compliance with its specifications. The investigator or a designated person from his/her team will be trained for the use of the e-CRF by the sponsor.

Data entry at the investigator's site will be performed by the investigator or by the designated person from his/her team after completion of the patient's Medical File.

Upon entry, data will be transmitted via the Internet from the study center to the study database.

The investigator or the designated person from his/her team agrees to complete the e-CRF, at each patient visit, and all other documents provided by the sponsor (e.g. documents relating to the IMP management...).

The eCRF must be completed as soon as possible following each visit.

All corrections of data on the eCRF must be made by the investigator or by the designated person from his/her team using electronic data clarifications according to the provided instructions. All data modification will be recorded using the audit trail feature of Inform software, including date, reason for modification and identification of the person who has made the change.

In order to ensure confidentiality and security of the data, usernames and passwords will be used to restrict system access to authorized personnel only, whether resident within the investigator's sites, the sponsor or third parties.

Data will be verified in accordance with the monitoring strategy defined for the study. After comparing these data to the source documents, the monitor will request correction / clarification from the investigator using electronic data clarifications that should be answered and closed as quickly as possible.

Data can be frozen during the study after their validation. However the investigator has the possibility to modify a data if deemed via a request to the sponsor.

After the last visit of the patient, the investigator or co-investigator must attest the authenticity of the data collected in the eCRF by entering his/her user name and password.

After the data base lock, the investigator, or an authorized member of his/her team, will have to download from the e-CRF an electronic file containing participant data from his/her center for archiving in the study file (see Section 14.4).

#### 14.3. Data management

Data are collected via an eCRF and stored in a secured database.

For data collected on the e-CRF, the Data & Clinical Logistics of I.R.I.S. is responsible for data processing, including data validation according to a specification manual describing the checks to be carried out. As a result of data validation, data may require some changes. An electronic data clarification form is sent to the investigator who is required to respond to the query and make any necessary changes to the data.

The Data & Clinical Logistics Division of I.R.I.S. is responsible for all data transfers.



and PK results will be transferred to the Data & Clinical Logistics Division of I.R.I.S. after clinical database lock.

The Medical Data Department of I.R.I.S. is responsible for data coding including:

- medical / surgical history, AEs and procedures using the Medical Dictionary for Regulatory Activities (MedDRA),
- medications using the World Health Organization, Drug Dictionary (WHO-DRUG).

The coding process is described in a specification manual.

The investigator ascertains he/she will apply due diligence to avoid protocol deviations. Under no circumstances should the investigator contact the sponsor or its representatives monitoring the study, if any, to request approval of a protocol deviation, as no deviations are permitted. If the investigator feels a protocol deviation would improve the conduct of the study this must be considered a protocol amendment, and unless such an amendment is agreed upon by the sponsor and approved by the IRB/IEC it cannot be implemented. All important protocol deviations will be recorded and reported in the clinical study report.

When data validation is achieved, a blind review of the data is performed according to the sponsor standard operating procedure. When the database has been declared to be complete and accurate, it will be locked and the IMP codes will be unblinded and made available for data analysis.

# 14.4. Archiving

The investigator will keep all information relevant to the study for at least 25 years after the end of the study, or more if specified by the local regulation, or for US sites two years after approval of the New Drug Application (NDA) or discontinuation of the Investigational New Drug (IND) (it include all source data, and that these data should be readable during the archiving period).

At the end of the study, the investigator or an authorized member of his/her team, will download an electronic copy of each participant's data from e-CRF and should keep it in a reliable secure and durable location. The file must include appropriate restrictions (password protection) and adequate protection from loss, physical damage or deterioration for the duration of the archiving period. These data include all data and comments reported in the e-CRF, the history of all queries and signatures and the full audit trail reports.

#### 15. INSURANCE

#### 15.1. For non US countries:

I.R.I.S., or any parent company of SERVIER GROUP in charge of the management of clinical trials, is insured under the liability insurance program subscribed by LES LABORATOIRES SERVIER to cover its liability as sponsor of clinical trials on a worldwide basis.

Where an indemnification system and/or a mandatory policy are in place, I.R.I.S. or any parent company of SERVIER GROUP will be insured under a local and specific policy in strict accordance with any applicable law.

All relevant insurance documentation is included in the file submitted to any authorities' approval of which is required.

# 15.2. For US country only:

#### 15.2.1. Indemnification

Under the conditions of a contract concluded between investigator, site and the sponsor Galapagos NV or designee, which shall prevail, the sponsor Galapagos NV shall, except in case of gross negligence or willful misconduct, indemnify and hold harmless the investigator and his/her medical staff from any claim arising from the clinical study activities carried out in compliance with the clinical study protocol (CSP), Galapagos NV's instructions and applicable local regulations.

The investigator must notify the sponsor Galapagos NV immediately upon notice of any claims or lawsuits.

# 15.2.2. Insurance

The sponsor Galapagos NV shall maintain insurance coverage that is sufficient to cover its obligations and that is consistent with human clinical study local regulations. Save in case of gross negligence or willful misconduct of the investigator, and provided that the patient has been treated according to the CSP and Galapagos NV's instructions, any injury caused to a patient which is the direct result of his/her participation to the clinical study shall be covered by Galapagos NV's insurance.

# 16. OWNERSHIP OF THE RESULTS – DATA SHARING POLICY AND PUBLICATION POLICY

Les Laboratoires Servier and Institut de Recherches Servier and Galapagos ("Servier"), and I.R.I.S. affiliate, and Galapagos N.V. ("Galapagos") entered into a Product Development, Option, License and Commercialization Agreement dated as of 28 June 2010 (as amended from time to time, the "Servier-Galapagos Agreement"), which outlines their rights and responsibilities relating to ownership of the results of the Study, data sharing and publications.

As required by the Servier-Galapagos Agreement, each of I.R.I.S. and Galapagos will ensure in their respective territory that the key design elements of this protocol will be posted in a publicly accessible database such as clinicaltrials.gov. In addition, upon study completion and finalization of the study report, the results of this study will be either submitted for publication and/or posted in a publicly accessible database of clinical study results.

Any draft of publication and/or communication relative to the study and/or relative to the obtained results during the study or after the study end shall be submitted to I.R.I.S. and Galapagos. As between I.R.I.S. and Galapagos, each of them shall ensure that the other has the opportunity to review any proposed publication and/or communication in accordance with Article 6 of the Servier-Galapagos Agreement.

The investigator, who submitted the draft, shall take the comments received from either cosponsor into due consideration.

As the study is a multicenter one, the first publication must be performed only with data collected from several centers and analyzed under the responsibility of I.R.I.S for the ROW Territories and Galapagos for US Territory. The investigator commits himself not to publishing or communicating data collected in only one center or part of the centers before the publication of the complete results of the study, unless prior written agreement from the other investigators, I.R.I.S. and Galapagos has been provided.

#### 17. ADMINISTRATIVE CLAUSES

# 17.1. Concerning the sponsor and the investigator

#### 17.1.1. Persons to inform

In accordance with local regulations, the investigator and/or the sponsor will inform the Director of the medical institution, the pharmacist involved in the study and the Director of the analysis laboratory.

With the agreement of the patient, the investigator will inform the patient's general practitioner about his/her patient's participation in a clinical study.

# 17.1.2. Substantial protocol amendment and amended protocol

If the protocol must be altered after it has been signed, the modification or substantial amendment must be discussed and approved by the coordinators and the sponsor.

The substantial protocol amendment must be drafted in accordance with the sponsor standard operating procedure and an amended protocol must be signed by both parties. Both documents must be kept with the initial protocol.

All substantial amendments and corresponding amended protocols must be sent by the investigator(s) or the coordinator(s) or the sponsor, in accordance with local regulations, to the IRB/IEC that examined the initial protocol. They can only be implemented after a favorable opinion of the IRB/IEC has been obtained, local regulatory requirements have been complied with, and the amended protocol has been signed, with the exception of a measure required to eliminate an immediate risk to the study patients.

When the submission is performed by the investigator or the coordinator, the latter must transmit a copy of IRB/IEC's new written opinion to the sponsor, immediately upon receipt.

Furthermore, the substantial amendment and amended protocol are to be submitted to the Regulatory Agencies in accordance with local regulations.

### 17.1.3. Final study report

The study report will be drafted by I.R.I.S. in compliance with I.R.I.S. standard operating procedure and Galapagos requirements.

The sponsors' representatives and the coordinators must mutually agree on the final version. One copy of the final report must be dated and signed by the coordinators and the sponsor's representatives.

# 17.2. Concerning the sponsor

The sponsor undertakes to:

- supply the investigator with adequate and sufficient information concerning the IMP administered during the study to enable him/her to carry out the study,
- supply the investigator with investigator's brochure if the study drug is not marketed,

- obtain any authorization to perform the study and/or import license for the IMP administered that may be required by the local authorities before the beginning of the study,
- provide coordinators annually, or with another frequency defined by the local regulations, with a document describing study progress which is to be sent to the IRB/IEC(s).

# 17.3. Concerning the investigator

# 17.3.1. Confidentiality - Use of information

All documents and information given to the investigator by the sponsor with respect to S201086/GLPG1972 and study CL2-201086-002/GLPG1972-CL-201 are strictly confidential. The investigator expressly agrees that data on his/her professional and clinical experience is collected by the sponsor on paper and computer, and stored for its sole use relating to its activities as the sponsor of clinical trials, in accordance with GCP.

He/she has a right to access, modify, and delete his/her own personal data by applying to the sponsor.

The investigator agrees that he/she and the members of his/her team will use the information only in the framework of this study, for carrying out the protocol. This agreement is binding as long as the confidential information has not been disclosed to the public by the sponsor. The clinical study protocol given to the investigator may be used by him/her or his/her colleagues to obtain the informed consent of study patients. The clinical study protocol as well as any information extracted from it must not be disclosed to other parties without the written authorization of the sponsor.

The investigator must not disclose any information without the prior written consent from the sponsor, except to the representatives of the Regulatory Agencies, and only at their request. In the latter case, the investigator commits himself/herself to informing the sponsor prior to disclosure of information to these authorities.

A patient screening log and a full identification and enrolment list of each patient will be completed and kept in a safe place by the investigator who should agree to provide access on site to the auditor and/or the representatives of the Regulatory Agencies. The information will be treated in compliance with professional secrecy.

The patient screening log must be completed from the moment the investigator checks that a patient could potentially take part in the study (by assessment of patient medical history during a visit or by examination of the medical file).

# 17.3.2. Organization of the center

The Investigator can delegate study tasks under his/her responsibility to others. Tasks can only be delegated to persons that are qualified to perform that specific task. An "Organization of center" or similar document needs to be completed for documentation purposes.

This document should be filled in at the beginning of the study and updated at any change of a person involved in the study in the center.

# 17.3.3. Documentation supplied to the sponsor

The investigator undertakes before the study begins:

- to provide his/her dated and signed English curriculum vitae (CV) or to complete in English the CV form provided by the sponsor or representative and to send it to the sponsor, together with that of his/her co-investigator(s),
- to provide a detailed description of the methods, techniques, and investigational equipment, and the reference values for the parameters measured,
- to provide any other document required by local regulation (e.g. Food & Drug Administration 1572 form),
- to send a copy of the IRB/IEC's opinion with details of its composition and the qualifications of its constituent members.

The CVs of other members of the team involved in the study (if possible in English) will be collected during the course of the study (at least, members involved in the patients' medical follow-up/study-related decision process and persons involved in the measurement of main assessment criteria).

#### 18. REFERENCES

Altman et al. Atlas of individual radiographic features in osteoarthritis, revised, Osteoarthritis and Cartilage (2007) 15, A1 - A56.

Caselli *et al.* Effect Size of the Anti-Aggrecanase-2 Monoclonal Antibody CRB0017 in Rodent Models of Osteoarthritis, ACR/ARHP Annual Meeting, 2015.

Chen P, Zhu S, Wang Y, Mu Q, Wu Y, Xia Q, Zhang X, Sun H, Tao J, Hu H, Lu P, Ouyang H. The amelioration of cartilage degeneration by ADAMTS-5 inhibitor delivered in a hyaluronic acid hydrogel. Biomaterials. 2014 Mar;35(9):2827-36.

Chen S, Huang Y, Zhou Z-J, Hu Z-J, Wang J-Y, Xu W-B, Fang X-Q and Fan S-W. Upregulation of Tumor Necrosis Factor (Alpha) and ADAMTS-5, but Not ADAMTS-4, in Human Intervertebral Cartilage Endplate With Modic Changes. Spine 2014;39(14): E817-E825.

Chiusaroli R, Visentini M, Galimberti C, Casseler C, Mennuni L, Covaceuszach S, Lanza M, Ugolini G, Caselli G, Rovati LC, Visintin MTargeting of ADAMTS5's ancillary domain with the recombinant mAb CRB0017 ameliorates disease progression in a spontaneous murine model of osteoarthritis. Osteoarthritis Cartilage. 2013 Nov;21(11):1807-10.

Chockalingam PS, Sun W, Rivera-Bermudez MA, Zeng W, Dufield DR, Larsson S, Lohmander LS, Flannery CR, Glasson SS, Georgiadis KE, Morris EA. Elevated aggrecanase activity in a rat model of joint injury is attenuated by an aggrecanase specific inhibitor. Osteoarthritis Cartilage. 2011 Mar;19(3):315-23.

Conaghan PG, Hunter DJ, Maillefert JF, Reichmann WM, Losina E. Summary and recommendations of the OARSI FDA osteoarthritis Assessment of Structural Change Working Group. Osteoarthritis Cartilage. 2011 May;19(5):606-10.

Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis 2014;73:1323-1330.

Durigova M, Nagase H, Mort JS, Roughley PJ. MMPs are less efficient than ADAMTS5 in cleaving aggrecan core protein. Matrix Biol. 2011;30(2):145-153.

Eckstein F, Collins JE, Nevitt MC, Lynch JA, Kraus V. Katz JN, Losina E, Wirth W, Guermazi A, Roemer FW, and Hunter DJ for the FNIH OA Biomarkers Consortium. Cartilae Thickness change as an imaging biomarker of knee osteoarthritis progression-data from the FNIH OA biomarkers consortium. Arthritis Rheumatol. 2015 Dec; 67(12):3184-89

Elders MJ. The increasing impact of arthritis on public health. J Rheumatol Suppl 2000;60:6-8.

Fosang AJ and Little CB. Drug insight: aggrecanases as therapeutic targets for osteoarthritis. Nat Clin Pract Rheumatol. 2008 Aug;4(8):420-7. PE0143656.

Germaschewski FM, Matheny CJ, Larkin J, Liu F, Thomas LR, Saunders JS, Sully K, Whittall C, Boyle Y, Peters G, Graham NM. Quantitation OF ARGS aggrecan fragments in synovial fluid, serum and urine from osteoarthritis patients. Osteoarthritis Cartilage 2014;22(5):690-697.

Glasson S, Askew R, Sheppard B, Carito B, Blanchet T *et al.* Deletion of active ADAMTS5 prevents cartilage degradation in a murine model of osteoarthritis. Nature, vol.434(7033), pp.644-648, 2005. PE0143661.

Heinegard D and Saxne T. The role of the cartilage matrix in osteoarthritis. Nat Rev Rheumatol. 2011 Jan;7(1):50-6..

Karsdal MA, Michaelis M, Ladel C, Siebuhr AS, Bihlet AR, Andersen JR, Guehring H, Christiansen C, Bay-Jensen AC, Kraus VB Disease-modifying treatments for osteoarthritis (DMOADs) of the knee and hip: lessons learned from failures and opportunities for the future. Osteoarthritis Cartilage. 2016 Dec;24(12):2013-2021.

Larsson S, Lohmander LS, Struglics A. An ARGS-aggrecan assay for analysis in blood and synovial fluid. Osteoarthritis Cartilage. 2014 Feb;22(2):242-9..

Lohmander LS, Neame PJ, Sandy JD. The structure of aggrecan fragments in human synovial fluid. Evidence that aggrecanase mediates cartilage degradation in inflammatory joint disease, joint injury, and osteoarthritis. Arthritis Rheum. 1993;36(9):1214-1222.

Lohmander LS, Hellot S, Dreher D, Krantz EF, Kruger DS, Guermazi A, Eckstein F. Intraarticular sprifermin (recombinant human fibroblast growth factor 18) in knee osteoarthritis: a randomized, double-blind, placebocontrolled trial. Arthritis Rheumatol. 2014;66(7):1820-1831.

Malfait A, Ritchie J, Gil A, Austin J, Hartke J, Qin W, Tortorella M and Mogil J. "ADAMTS-5 deficient mice do not develop mechanical allodynia associated with osteoarthritis following medial meniscal destabilization. Osteoarthritis Cartilage 2010;18(4):572-580..

Mallinckrodt CH, Lin Q and Molenberghs M. A structured framework for assessing sensitivity to missing data assumptions in longitudinal clinical trials. Pharmaceutical Statistics, 2013;12:1-6

Maschek S, Wirth W, Ladel C, Hellio Le Graverand MP, Eckstein F. Rates and sensitivity of knee cartilage thickness loss in specific central reading radiographic strata from the osteoarthritis initiative. Osteoarthritis Cartilage. 2014 Oct;22(10):1550-3.

Miller RE, Tran PB, Ishihara S, Larkin J, Malfait AM. Therapeutic effects of an anti-ADAMTS-5 antibody on joint damage and mechanical allodynia in a murine model of osteoarthritis. Osteoarthritis Cartilage. 2016 Feb;24(2):299-306.

Sandy JD, Verscharen C. Analysis of aggrecan in human knee cartilage and synovial fluid indicates that aggrecanase (ADAMTS) activity is responsible for the catabolic turnover and loss of whole aggrecan whereas other protease activity is required for C-terminal processing in vivo. Biochem J. 2001;358(Pt 3):615-626.

Sandy JD. A contentious issue finds some clarity: on the independent and complementary roles of aggrecanase activity and MMP activity in human joint aggrecanolysis. Osteoarthritis Cartilage 2006;14(2):95-100.

Struglics A, Hansson M, Lohmander LS. Human aggrecanase generated synovial fluid fragment levels are elevated directly after knee injuries due to proteolysis both in the inter globular and chondroitin sulfate domains. Osteoarthritis Cartilage 2011;19(8):1047-1057.

Verma P and Dalal K. ADAMTS-4 and ADAMTS-5: key enzymes in osteoarthritis. J Cell Biochem. 2011 Dec;112(12):3507-14.

WHO. Background paper 5. Demography, global burden of disease and the preliminary list of priorities. Update on 2004 background paper. 2013.

Zhang E, Yan X, Zhang M, Chang X, Bai Z, He Y, Yuan Z. Aggrecanases in the human synovial fluid at different stages of osteoarthritis. Clin Rheumatol. 2013;32(6):797-803.

Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recomendations for the management of hip and knee osteoarthritis, Part III: change in evidence following systematic cumulative update of research published through January 2009. Osteoarthitis Cartilage 2010;18:476-499.

#### Other regulatory references:

ICH Topic E6 – Guideline for Good Clinical Practice: Consolidated guideline finalised (step 4) in June 1996. Adopted by CPMP, July 96, issued as CPMP/ICH/135/95/step 5, post step errata, July 2002, revision 2 Feb. 2016.

ICH Topic E9 – Statistical Principles for Clinical Trials: Adopted by CPMP, March 1998, issued as CPMP/ICH/363/96/step 5.

ICH Topic E2A – Clinical Safety Data Management: Definitions and Standards for Expedited Reporting, issued as CPMP/ICH/377/95.

ICH E14 – The Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic drugs – Adopted by CHMP, May 2005, issued as CHMP/ICH/2/04.

Detailed guidance on the collection, verification and presentation of adverse event/reaction reports arising from clinical trials on medicinal products for human use ('CT-3'), (2011/C 172/01).

DIRECTIVE 2001/20/EC OF THE EUROPEAN PARLIAMENT AND OF THE COUNCIL of 4 April 2001 on the approximation of the laws, regulations and administrative provisions of the Member States relating to the implementation of good clinical practice in the conduct of clinical trials on medicinal products for human use).

FDA guidance, Guidance for Clinical Trial Sponsors Establishment and Operation of Clinical Trial Data Monitoring Committees March 2006.

Guideline CHMP/EWP/5872/03 Corr., 27 July 2005.

GLPG1972 – investigator's brochure – version n°6/S201086 – investigator's brochure – version n°3.

https://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm

#### 19. APPENDICES

# Appendix 1: World Medical Association Declaration of Helsinki

# WORLD MEDICAL ASSOCIATION DECLARATION OF HELSINKI

# **Ethical Principles for Medical Research Involving Human Subjects**

Adopted by the 18th WMA General Assembly, Helsinki, Finland, June 1964, and amended by the:

29th WMA General Assembly, Tokyo, Japan, October 1975

35th WMA General Assembly, Venice, Italy, October 1983

41st WMA General Assembly, Hong Kong, September 1989

48th WMA General Assembly, Somerset West, Republic of South Africa, October 1996

52nd WMA General Assembly, Edinburgh, Scotland, October 2000

53th WMA General Assembly, Washington DC, USA, 2002 (Note of Clarification added)

55th WMA General Assembly, Tokyo, Japan, 2004 (Note of Clarification added)

59th WMA General Assembly, Seoul, Republic of Korea, October 2008

64th WMA General Assembly, Fortaleza, Brazil, October 2013

### **Preamble**

- 1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving human subjects, including research on identifiable human material and data.
  - The Declaration is intended to be read as a whole and each of its constituent paragraphs should be applied with consideration of all other relevant paragraphs.
- 2. Consistent with the mandate of the WMA, the Declaration is addressed primarily to physicians. The WMA encourages others who are involved in medical research involving human subjects to adopt these principles

### **General Principles**

- 3. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 4. It is the duty of the physician to promote and safeguard the health, well-being and rights of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfillment of this duty.
- 5. Medical progress is based on research that ultimately must include studies involving human subjects.
- 6. The primary purpose of medical research involving human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best proven

- interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 7. Medical research is subject to ethical standards that promote and ensure respect for all human subjects and protect their health and rights.
- 8. While the primary purpose of medical research is to generate new knowledge, this goal can never take precedence over the rights and interests of individual research subjects.
- 9. It is the duty of physicians who are involved in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research subjects. The responsibility for the protection of research subjects must always rest with the physician or other health care professionals and never with the research subjects, even though they have given consent.
- 10. Physicians must consider the ethical, legal and regulatory norms and standards for research involving human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research subjects set forth in this Declaration.
- 11. Medical research should be conducted in a manner that minimizes possible harm to the environment.
- 12. Medical research involving human subjects must be conducted only by individuals with the appropriate ethics and scientific education, training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional.
- 13. Groups that are underrepresented in medical research should be provided appropriate access to participation in research.
- 14. Physicians who combine medical research with medical care should involve their patients in research only to the extent that this is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research study will not adversely affect the health of the patients who serve as research subjects.
- 15. Appropriate compensation and treatment for subjects who are harmed as a result of participating in research must be ensured.

#### Risk, Burdens and Benefits

16. In medical practice and in medical research, most interventions involve risks and burdens.

- Medical research involving human subjects may only be conducted if the importance of the objective outweighs the risks and burdens to the research subjects.
- 17. All medical research involving human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and groups involved in the research in comparison with foreseeable benefits to them and to other individuals or groups affected by the condition under investigation.
  - Measures to minimize the risks must be implemented. The risks must be continuously monitored, assessed and documented by the researcher.
- 18. Physicians may not be involved in a research study involving human subjects unless they are confident that the risks have been adequately assessed and can be satisfactorily managed.

When the risks are found to outweigh the potential benefits or when there is conclusive proof of definitive outcomes, physicians must assess whether to continue, modify or immediately stop the study.

# **Vulnerable Groups and Individuals**

- 19. Some groups and individuals are particularly vulnerable and may have an increased likelihood of being wronged or of incurring additional harm.
  - All vulnerable groups and individuals should receive specifically considered protection.
- 20. Medical research with a vulnerable group is only justified if the research is responsive to the health needs or priorities of this group and the research cannot be carried out in a non-vulnerable group. In addition, this group should stand to benefit from the knowledge, practices or interventions that result from the research.

# **Scientific Requirements and Research Protocols**

- 21. Medical research involving human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 22. The design and performance of each research study involving human subjects must be clearly described and justified in a research protocol.
  - The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, sponsors, institutional affiliations, potential conflicts of interest, incentives for subjects and information regarding provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the research study.

In clinical trials, the protocol must also describe appropriate arrangements for post-trial provisions.

#### **Research Ethics Committees**

23. The research protocol must be submitted for consideration, comment, guidance and approval to the concerned research ethics committee before the study begins. This committee must be transparent in its functioning, must be independent of the researcher, the sponsor and any other undue influence and must be duly qualified. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research subjects set forth in this Declaration.

The committee must have the right to monitor on-going studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No amendment to the protocol may be made without consideration and approval by the committee. After the end of the study, the researchers must submit a final report to the committee containing a summary of the study's findings and conclusions.

# **Privacy and Confidentiality**

24. Every precaution must be taken to protect the privacy of research subjects and the confidentiality of their personal information.

# **Informed Consent**

- 25. Participation by individuals capable of giving informed consent as subjects in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no individual capable of giving informed consent may be enrolled in a research study unless he or she freely agrees.
- 26. In medical research involving human subjects capable of giving informed consent, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the study and the discomfort it may entail, post-study provisions and any other relevant aspects of the study. The potential subject must be informed of the right to refuse to participate in the study or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential subjects as well as to the methods used to deliver the information.

After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.

All medical research subjects should be given the option of being informed about the general outcome and results of the study.

- 27. When seeking informed consent for participation in a research study the physician must be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent must be sought by an appropriately qualified individual who is completely independent of this relationship.
- 28. For a potential research subject who is incapable of giving informed consent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research study that has no likelihood of benefit for them unless it is intended to promote the health of the group represented by the potential subject, the research cannot instead be performed with persons capable of providing informed consent, and the research entails only minimal risk and minimal burden.
- 29. When a potential research subject who is deemed incapable of giving informed consent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.
- 30. Research involving subjects who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research group. In such circumstances the physician must seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the study may proceed without informed consent provided that the specific reasons for involving subjects with a condition that renders them unable to give informed consent have been stated in the research protocol and the study has been approved by a research ethics committee. Consent to remain in the research must be obtained as soon as possible from the subject or a legally authorized representative.
- 31. The physician must fully inform the patient which aspects of their care are related to the research. The refusal of a patient to participate in a study or the patient's decision to withdraw from the study must never adversely affect the patient-physician relationship.
- 32. For medical research using identifiable human material or data, such as research on material or data contained in biobanks or similar repositories, physicians must seek informed consent for its collection, storage and/or reuse. There may be exceptional situations where consent would be impossible or impracticable to obtain for such research. In such situations the research may be done only after consideration and approval of a research ethics committee.

# **Use of Placebo**

33. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best proven intervention(s), except in the following circumstances:

Where no proven intervention exists, the use of placebo, or no intervention, is acceptable; or

Where for compelling and scientifically sound methodological reasons the use of any intervention less effective than the best proven one, the use of placebo, or no intervention is necessary to determine the efficacy or safety of an intervention

and the patients who receive any intervention less effective than the best proven one, placebo, or no intervention will not be subject to additional risks of serious or irreversible harm as a result of not receiving the best proven intervention.

Extreme care must be taken to avoid abuse of this option.

# **Post-Trial Provisions**

34. In advance of a clinical trial, sponsors, researchers and host country governments should make provisions for post-trial access for all patients who still need an intervention identified as beneficial in the trial. This information must also be disclosed to participants during the informed consent process.

# Research Registration and Publication and Dissemination of Results

- 35. Every research study involving human subjects must be registered in a publicly accessible database before recruitment of the first subject.
- Researchers, authors, sponsors, editors and publishers all have ethical obligations with regard to the publication and dissemination of the results of research. Researchers have a duty to make publicly available the results of their research on human subjects and are accountable for the completeness and accuracy of their reports. All parties should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results must be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest must be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

# **Unproven Intervention in Clinical Practice**

In the treatment of an individual patient, where proven interventions do not exist or other known interventions have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgment it offers hope of saving life, re-establishing health or alleviating suffering. This intervention should subsequently be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information must be recorded and, where appropriate, made publicly available.

# **Appendix 2: Western Ontario and McMaster Universities Osteoarthritis Index** (WOMAC)

# WOMAC OSTEOARTHRITIS INDEX VERSION LK3.1

| | INST | RUCTIONS TO | PATIENTS | | |
|---|---|---|---|---|---|
| | | tions are asked in<br>x " in one of the | | g format. Please m | ark |
| EXAMPLES: | | | | | |
| 1. If you put | your " x " ir | the box on the | far left as | shown below, | |
| none | mild | moderate | severe | extreme | |
| then you a | are indicating | that you feel no p | pain. | | |
| 2. If you put | your " 🗶 " in | the box on the | far right as | shown below, | |
| none | mild | moderate | severe | extreme | |
| then you a | are indicating | that you feel extr | eme pain. | | |
| Please no a) that the you fee | further to the | e right you place | your " <b>X</b> ", the | e more pain | |
| b) that the<br>you fee | | e left you place | your " 🗴 ", th | e less pain | |
| c) please | do not place | e your " 🗶 " outsi | ide any of th | ne boxes. | |
| | | on this type of s<br>uring the last 48 | | unt of pain, stiffne | SS |
| | cate the seve | rity of your pain a | and stiffness | nen answering th<br>and the difficulty yo<br>I by the arthritis | u |
| | re which joint | | | n care professiona<br>k before completin | |

Copyright@1996 Nicholas Bellamy All Rights Reserved

WOMA

#### Section A

# PAIN

Think about the pain you felt in your \_\_\_\_\_ (study joint) caused by your arthritis during the <u>last 48 hours</u>.

(Please mark your answers with an " x ".)

| QUESTION: Ho | w much pa | in have you ha | ad | | Study Coordinator<br>Use Only |
|---|---|---|---|---|---|
| 1. when walkin | g on a flat su | rface? | | | 0.0000000000000000000000000000000000000 |
| none | mild | moderate | severe | extreme | PAIN1 |
| 2. when going | up or down s | tairs? | | | |
| none | mild | moderate | severe | extreme | PAIN2 ——— |
| 3. at night while | e in bed? (th | at is - pain that di | sturbs your sl | eep) | |
| none | mild | moderate | severe | extreme | PAIN3 |
| 4. while sitting | or lying down | ? | | | |
| none | mild | moderate | severe | extreme | PAIN4 |
| 5. while standir | ng? | | | | |
| none | mild | moderate | severe | extreme | PAIN5 |

Copyright@1996 Nicholas Bellamy All Rights Reserved

**WOM**<sub>B</sub>

# Section B

| | | | ST | IFFNES | S | |
|---|---|---|---|---|---|---|
| | | | fness (not p<br>e arthritis du | | felt in your<br>ast 48 hours. | (study |
| St | iffness is | a sens | ation of de | creased | ease in mov | ing your joint. |
| (Pl | ease mark yo | our answers | with an " x ".) | | | 0000 |
| 6. | How severe | | tiffness been afte | er you first w | oke up | Study Coordinator<br>Use Only |
| | none | mild | moderate | severe | extreme | STIFF6 |
| 7. | | e has your s<br>g later in th | tiffness been afte<br>e day? | r sitting or lyir | ng down or | |
| | none | mild | moderate | severe | extreme | STIFF7 |

Copyright@1996 Nicholas Bellamy All Rights Reserved

WOMc1-3

#### Section C

# **DIFFICULTY PERFORMING DAILY ACTIVITIES**

Think about the difficulty you had in doing the following daily physical activities caused by the arthritis in your \_\_\_\_\_ (study joint) during the <u>last 48 hours</u>. By this we mean your ability to move around and take care of yourself. (Please mark your answers with an " x ".)

| QUESTION: | How much | difficulty have | you had . | | Study Coordinator<br>Use Only |
|---|---|---|---|---|---|
| 8. when goin | g down the st | airs? | | | 10.700 |
| none | mild | moderate | severe | extreme | PFTN8 |
| 9. when goin | g up the stairs | s? | | | |
| none | mild | moderate | severe | extreme | PFTN9 |
| 10. when getti | ng up from a | sitting position? | | | |
| none | mild | moderate | severe | extreme | PFTN10 |
| 11. while stand | ding? | | | | |
| none | mild | moderate | severe | extreme | PFTN11 |
| 12. when bend | ding to the floo | or? | | | |
| none | mild | moderate | severe | extreme | PFTN12 |
| 13. when walk | ing on a flat s | surface? | | | |
| none | mild | moderate | severe | extreme | PFTN13 |

Copyright@1996 Nicholas Bellamy All Rights Reserved

WOMc2-3

# **DIFFICULTY PERFORMING DAILY ACTIVITIES**

Think about the difficulty you had in doing the following daily physical activities caused by the arthritis in your \_\_\_\_\_ (study joint) during the <u>last 48 hours</u>. By this we mean your ability to move around and take care of yourself. (Please mark your answers with an " x ".)

| QU | JESTION: | How much | difficulty have | you had . | ** | Study Coordinator<br>Use Only |
|---|---|---|---|---|---|---|
| 14. | getting in | or out of a car | , or getting on or | off a bus? | | |
| | none | mild | moderate | severe | extreme | PFTN14 |
| 15. | while goir | ng shopping? | | | | |
| | none | mild | moderate | severe | extreme | PFTN15 |
| 16. | when putt | ing on your so | cks or panty hos | e or stockings | 5? | 11 |
| | none | mild | moderate | severe | extreme | PFTN16 |
| 17. | when gett | ing out of bed | ? | | | |
| | none | mild | moderate | severe | extreme | PFTN17 |
| 18. | when taki | ng off your so | cks or panty hose | e or stockings | ? | |
| | none | mild | moderate | severe | extreme | PFTN18 |
| 19. | while lying | g in bed? | | | | |
| | none | mild | moderate | severe | extreme | PFTN19 |

Copyright@1996 Nicholas Bellamy All Rights Reserved

WOMc3-3

# DIFFICULTY PERFORMING DAILY ACTIVITIES

Think about the difficulty you had in doing the following daily physical activities caused by the arthritis in your \_\_\_\_\_ (study joint) during the <u>last 48 hours</u>. By this we mean your ability to move around and take care of yourself. (Please mark your answers with an " x ".)

| QUESTION: | How much | difficulty have | you had . | | Study Coordinator<br>Use Only |
|---|---|---|---|---|---|
| 20. when getti | ing in or out o | f the bathtub? | | | 11 |
| none | mild | moderate | severe | extreme | PFTN20 |
| 21. while sittin | ıg? | | | | |
| none | mild | moderate | severe | extreme | PFTN21 |
| 22. when getti | ing on or off th | he toilet? | | | |
| none | mild | moderate | severe | extreme | PFTN22 |
| 23. while doin | g heavy hous | sehold chores? | | | |
| none | mild | moderate | severe | extreme | PFTN23 |
| 04 | - E-111 | | | | |
| 24. while doin | 5175 | | | 20 | PFTN24 |
| none | mild | moderate | severe | extreme | P1 11924 |
| _ | _ | _ | _ | _ | |

Copyright@1996 Nicholas Bellamy All Rights Reserved

# **Appendix 3: Knee Pain Visual Analog Scale**

# **KNEE PAIN (Screening visit)**

"How would you rate the pain you have felt in each knee within the last 48 hours?" Please indicate on the line the place that best expresses your pain as you feel it within the last 48 hours. 0 = no pain (on the left) and 100 = extreme pain (on the right) Left Knee: Extreme pain No pain Right knee: No pain Extreme pain **KNEE PAIN (other visits)** "How would you rate the pain you have felt in the study knee within the last 48 hours? If you are unsure which knee is your study knee, please ask your research doctor before answering." Please indicate on the line the place that best expresses your pain as you feel it within the last 48 hours. 0 = no pain (on the left) and 100 = extreme pain (on the right) No pain Extreme pain

# Appendix 4: Patient Global Assessment of disease activity Visual Analog Scale

# PATIENT GLOBAL ASSESSMENT

"Considering all the ways in which your knee osteoarthritis affects you, please rate on this 100 mm scale how well you are doing today"

Please indicate on the line the place that best expresses your feeling as you feel it right now. 0 = very poorly (on the left) and 100 = very well (on the right)



# Appendix 5: Substantial Amendment No 1 to the clinical study protocol

SUBSTANTIAL AMENDMENT N° 1 TO THE CLINICAL Document title

STUDY PROTOCOL

Study title Efficacy and safety of 3 doses of S201086/GLPG1972

administered orally once daily in patients with knee

osteoarthritis. A 52-week international, multi-regional, multicenter, randomized, double-blind, placebo-controlled, dose-

ranging study.

Test drug code S201086/GLPG1972

Osteoarthritis Indication

Phase 2 Development phase

Protocol code CL2-201086-002/GLPG1972-CL-201

EudraCT Number 2017-004581-10

Universal Trial Number

Investigational New

Drug Application

Number

U1111-1205-0321

133039

Country code **INT** 

GALAPAGOS NV (US) Sponsor

Institut de Recherches Internationales Servier (I.R.I.S.) (ex-US)

11<sup>th</sup> July 2018 Date of the document

Version of the document Final version

#### **CONFIDENTIAL**

| > SUBJECT | | |
|---|---|---|
| Inclusion / withdrawal criteria | X | Investigational Medicinal<br>Product (IMP), dosage |
| Number of participants | | Exposure duration to IMP |
| Modification of study design (additional visit / examinations) | | Definition of the end of the trial |
| Primary / secondary endpoints | | New safety information |
| | | Other (management of overdose, X statistics, minor clarifications or changes or corrections compared to previous version) |

#### JUSTIFICATION FOR THE AMENDMENT

The main aim of this substantial amendment is to increase the age of female patients of non-childbearing potential to 50 years old instead of 40 years old (inclusion criterion n°1) (except for female patients surgically sterile)

Information regarding the management of an overdose of S201086/GLPG1972 has been added on the study protocol on section 5.5.1 withdrawal criteria and section 8.9.2.4 special situations

One withdrawal criterion "delta > 60 ms over baseline value (inclusion)" has been added on ECG parameters (section 5.5.1 withdrawal criteria) as beside the absolute values on QTcF the delta is also an important parameter to evaluate for the safety of the patient.

to evaluate also the consistency of the primary analysis' results between Japanese patients and non-Japanese patients (section 10. Statistics). In order to ensure balanced Japanese patients between treatment groups, the stratification factors of the randomization list have been modified consequently.

The choice of the target knee has been clarified in the inclusion criterion n°9.

Minor clarifications or changes or corrections have been made.

#### EFFECTS OF THE AMENDMENT

All sites will be concerned by this amendment after approval by Competent Authorities/Ethics Committees. The participant information and consent form will be also amended.

#### **CHANGES**

Changes and modified text are described below and included in the joined amended protocol.

#### AMENDED TEXT

# Section Cover page concerned by the substantial amendment

Study acronym added: ROCCELLA Study.

# Section Study summary sheet concerned by the substantial amendment

Title of study (acronym added):

ROCCELLA study.

[....]

Methodology:

[...]

The randomization will be stratified by region (Asia and Rest of the World).

#### Diagnosis and main criteria for inclusion:

Main screening criteria are:

Male patients or female patients of nonchildbearing potential, age 40-75 years (both inclusive), body weight > 40 kg,

[...]

#### Criteria for evaluation:

#### Efficacy measurements:

Secondary efficacy endpoints:

 The change from baseline to W052 in WOMAC subscales scores of the target knee for pain, function and stiffness

#### Statistical methods:

#### Analysis sets:

#### - Randomized Set (RS):

All patients to whom a therapeutic unit was randomly assigned using IWRS.

# - Safety Set (SS):

All patients having taken at least one dose of study drug.

#### Methodology:

[...]

The randomization will be stratified by zone (Japan, South Korea/Taiwan and Rest of the World).

#### Diagnosis and main criteria for inclusion:

Main screening criteria are:

Male patients or female patients of nonchildbearing potential, age 40-75 years for male patients and female surgically sterile patients, and 50-75 years for postmenopausal female patients (both inclusive), body weight > 40 kg,

[...]

#### Criteria for evaluation:

Efficacy measurements:

Secondary efficacy endpoints:

 The change from baseline to W052 in WOMAC total score and subscales scores of the target knee for pain, function and stiffness

#### Statistical methods:

Analysis sets:

# Randomized Set (RS):

The Randomised Set (RS) will be constituted of all patients to whom a therapeutic unit was randomly assigned using IWRS. The RS will be used for efficacy analyses. Patients will be analysed according to the randomised treatment. All patients to whom a therapeutic unit was randomly assigned using IWRS.

#### - Safety Set (SS):

The Safety Set (SS) will be constituted of all patients having taken at least one dose of IMP. The SS will be used for safety analyses. Patients will be analysed according to treatment actually received at inclusion. All

patients having taken at least one dose of study drug.

Efficacy analysis:

#### Primary endpoint:

[....]

The MMRM as a primary analysis will assume that patients would keep the benefit of the randomized treatment after study discontinuation. For patients with an early discontinuation from the study (delay between the Early Termination and baseline less than 2 months) and without any post baseline measurement of cartilage thickness, a multiple imputation procedure will be used to impute the missing evaluations.

[...]

The consistency of the results between the Asian population and the non-Asian population will be evaluated on primary endpoint, according to the Method 2 defined in Ministry of Health Labor and Welfare Notification (MHLW) Notification "Basic principles on Global Clinical Trials". Treatment effect estimates and confidence intervals will be provided, for each dose, in Asian population and non-Asian population. In case of a statistically significant overall treatment effect (in favor of S201086/GLPG1972) at a considered dose, the results will be considered consistent if the observed treatment effects in Asian and nonpatients Asian favor are in S201086/GLPG1972.

[...]

#### Secondary endpoints:

Analysis will include the fixed, categorical effects of treatment, regions (Asia, US and Rest of the World), as well as the continuous, fixed covariate of baseline.

Efficacy analysis:

#### Primary endpoint:

[...]

The MMRM as a primary analysis will assume that patients would keep the benefit of the randomized treatment after study discontinuation. A missing data Handling will be used for this analysis. For patients with an early discontinuation from the study (delay between the Early Termination and baseline less than 2 months) and without any post baseline measurement of cartilage thickness, a multiple imputation procedure will be used to impute the missing evaluations.

[...]

The consistency of the results between the Asian population and the non-Asian population (respectively between Japanese population and non-Japanese population) will be evaluated on primary endpoint, according to the Method 2 defined in Ministry of Health Labor and Welfare Notification (MHLW) Notification "Basic principles on Global Clinical Trials". Treatment effect estimates and confidence intervals will be provided, for each dose, in Asian population and non-Asian population (respectively between Japanese population and non-Japanese population). In case of a statistically significant overall treatment effect (in favor S201086/GLPG1972) at a considered dose, the results will be considered consistent if the observed treatment effects in Asian and non-Asian (respectively between population and non-Japanese population) are in favor of S201086/GLPG1972.

[...]

#### Secondary endpoints:

Analysis will include the fixed, categorical effects of treatment, regions (Asia, US and Rest of the World), as well as the continuous, fixed covariate of baseline.

Section List of abbreviations concerned by the substantial amendment
| RR: respiratory rate | RR: RR: respiratory rate |
|---|---|
| Section 2. Background information conce | erned by the substantial amendment |
| Typo on drug name | Replace (3 times) |
| S201086/GLPG | S201086/GLPG1972 |
| S201086 | S201086/GLPG1972 |
| GLPG1972 | S201086/GLPG1972 |
| Section 4.1. Endpoints concerned by the s | substantial amendment |
| Secondary efficacy endpoints: - The change from baseline to W052 in WOMAC subscales scores of the target knee for pain, function, and stiffness | |
| Section 4.2.2. Investigation schedule conc | erned by the substantial amendment |
| Secondary WOMAC Safety measurements Laboratory examinations. | Secondary WOMAC [ePRO or paper (only if ePRO is unvailable)] Safety measurements Laboratory examinations (for screening visit). 9. Including Hepatitis B, C and HIV |
| Section 4.3. Measures to minimize bias co | |
| [] The treatment, S201086/GLPG1972 75 mg/day, 150 mg/day, 300 mg/day or matching placebo, will be assigned at randomized visit (W000) by a balanced (1:1:1:1), non-adaptive randomization, with stratification by region (Asia and Rest of the World). [] Pain VAS, and PGA VAS will be recorded using electronic patient reported outcome (ePRO). [] | [] The treatment, S201086/GLPG1972 75 mg/day, 150 mg/day, 300 mg/day or matching placebo, will be assigned at randomized visit (W000) by a balanced (1:1:1:1), non-adaptive randomization, with stratification by zone (Japan, South Korea/Taiwan and Rest of the World). [] |
| | [] |
| childbearing potential. Note: Female patients will be considered of non-childbearing potential if they are either surgically | 1.a. Male patients or female patients of non-childbearing potential and not breastfeeding. Note: Female patients will be considered of non-childbearing potential if they are either surgically sterile (e.g. tubal ligation, hysterectomy) or |

months of amenorrhea in the absence of other biological or physiological causes).

9.Disease stage based on a fixed flexion weightbearing X-ray of the target knee\* and central read out of:

- a. Predominant medial compartment radiographic disease
- b. KL grade 2 or 3
- And OARSI grade 1 or 2 medial tibiofemoral joint space narrowing (JSN)

\*The target knee (right or left) to be followed-up throughout the study will be chosen as follows:

- If both knees fulfill the clinical screening criteria (as described in 5.1) and radiological inclusion criteria, the knee to be chosen should be the most clinically painful one (Higher VAS score at screening).
- If both knees are equally painful, the most severely affected knee on X-ray (higher KL score); in case of similar KL scores, the higher JSN score will be selected.
- If both knees are equally painful and display the same radiological scores, the choice should be left to the investigator's discretion.

postmenopausal (at least 12 consecutive months of amenorrhea in the absence of other biological or physiological causes AND 50 years of age or older).

- 9.a. Disease stage based on a fixed flexion weightbearing X-ray of the target knee\* and central read out of:
  - a. Predominant medial compartment radiographic disease
  - b. KL grade 2 or 3
  - c. And OARSI grade 1 or 2 medial tibiofemoral joint space narrowing (JSN)

\*The target knee (right or left) to be followed-up throughout the study will be chosen as follows:

- If both knees fulfill the clinical screening criteria (as described in Section 5.1) and radiological inclusion criteria, the knee to be chosen should be the most severely affected knee on X-ray (higher KL score); in case of similar KL scores, the higher JSN score will be selected.
- If both knees display the same radiological scores, the knee to be chosen should be the most clinically painful one (Higher VAS score at screening).
- If both knees display the same radiological scores and are equally painful, the choice should be left to the investigator's discretion.

## Section 5.2. Exclusion criteria concerned by the substantial amendment

- 21. Previous osteotomy on the inferior limbs (whichever the side) 21.a. Previous osteotomy on the inferior limbs (whichever the side) other than intervention
- Surgical operation on the target knee within the 12 months prior to the screening visit or planned during the study period.
- Arthroscopy of the target knee within the 6 months prior to the screening visit or planned during the study period.
- 24. Other pathologies affecting the knee such as: septic arthritis, inflammatory joint disease, gout, major chondrocalcinosis (pseudogout), Paget's disease of the bone, ochronosis, acromegaly, haemochromatosis, Wilson's disease, rheumatic symptoms due to malignancies, primary osteochondromatosis, osteonecrosis, osteochondritis dissecans, hemophilia, etc.
- 31. Chronic use of strong opioids (see list under section 6.6 on symptomatic drugs).
- Known moderate to severe renal impairment;
   i.e., estimated Glomerular Filtration Rate (GFR) < 45 mL/min/1.73 m<sup>2</sup> (Modification of the Diet in Renal Disease [MDRD] formula).
- Clinically significant abnormalities detected on a 12-lead ECG performed at screening visit

- 21.a. Previous osteotomy on the inferior limbs (whichever the side) other than intervention for hallux valgus with full clinical recovery after surgery.
- 22.a. Any surgical operation on the target knee (arthroscopic or non-arthroscopic), other than diagnostic arthroscopy, within the 12 months prior to the screening visit or planned during the study period.
- 23.a. Diagnostic arthroscopy of the target knee within the 6 months prior to the screening visit or planned during the study period.
- 24.a. Other pathologies affecting the knee such as:
  septic arthritis, inflammatory joint disease,
  gout, major chondrocalcinosis (pseudogout),
  Paget's disease of the bone, ochronosis,
  acromegaly, haemochromatosis, Wilson's
  disease, rheumatic symptoms due to
  malignancies, primary osteochondromatosis,
  osteonecrosis, osteochondritis dissecans,
  documented severe intra-articular knee injury
  (e.g. intra-articular fracture), hemophilia, etc.
- 31.a. Chronic use of strong opioids (see and use of other prohibited drugs listed under section 6.6 on symptomatic drugs).

- of either rhythm or conduction (e.g., QT interval corrected for HR according to Fridericia's formula [QTcF] interval > 450 ms for males and > 470 ms for females, bradycardia with HR < 50 bpm, measured and stable PR > 280 ms, or second or third degree Atrio-Ventricular Block, complete left branch block)
- 44. Hypersensitivity to the active substance or to any of the excipients.
- 37.a. Known moderate to severe renal impairment; *i.e.*, estimated Glomerular Filtration Rate (GFR) < 45 mL/min/1.73 m<sup>2</sup> (Modification of the Diet in Renal Disease [MDRD] formula).
- 38.a. Clinically significant abnormalities detected on a 12-lead ECG performed at screening visit of either rhythm or conduction (e.g., QT interval corrected for HR according to Fridericia's formula [QTcF] interval > 450 ms for males and > 470 ms for females, bradycardia with HR < 50 bpm, measured and stable PR > 280 ms, or second or third degree Atrio-Ventricular Block, complete left branch block) (central reading)
- 44.a. Hypersensitivity to the active substance or to any of the excipients (e.g.: lactose).

#### Section 5.5.1. withdrawal criteria concerned by the substantial amendment

[...]

Treatment with S201086/GLPG1972 must be discontinued by the investigator and the patient must be withdrawn from the clinical study (preferably after discussion with the medical monitor, who may consult and must inform the sponsor's study physician) for any of the following conditions:

- Life-threatening adverse event (AE) or a SAE that places the patient at immediate risk
- Confirmed pregnancy
- Any ECG and/or laboratory parameter abnormalities such as:
  - QTcF > 500 ms on at least two separate ECGs
  - Increase in liver function tests:
    - ALT or AST > 8x ULN (discontinue the treatment immediately).
    - ALT or AST > 5x ULN confirmed at retest for more than 2 weeks,
    - ALT or AST > 3x ULN and (total bilirubin > 2x ULN or international normalized ratio [INR] > 1.5),
    - ALT or AST > 3x ULN
      with the appearance of
      fatigue, nausea, vomiting,
      right upper quadrant pain or
      tenderness, fever, rash,
      and/or eosinophilia (> 5%),
    - Presence of evocative clinical symptoms such as jaundice.

If any of the above laboratory abnormalities is detected, retesting is

[...]

Treatment with S201086/GLPG1972 must be discontinued by the investigator and the patient must be withdrawn from the clinical study (preferably after discussion with the medical monitor, who may consult and must inform the sponsor's study physician if applicable) for any of the following conditions:

- Life-threatening adverse event (AE) or a SAE that places the patient at immediate risk.
- Confirmed pregnancy
- Any ECG and/or laboratory parameter abnormalities such as:
  - QTcF > 500 ms or a delta > 60 ms over baseline value (inclusion) on at least two separate ECGs
  - Increase in liver function tests:
    - ALT or AST > 8x ULN (discontinue the treatment immediately),
    - ALT or AST > 5x ULN for eonfirmed at retest for more than 2 weeks (a decision to stop the study drug should be taken after a confirmed retest).
    - ALT or AST > 3x ULN and (total bilirubin > 2x ULN or international normalized ratio [INR] > 1.5),
    - ALT or AST > 3x ULN
      with the appearance of
      fatigue, nausea, vomiting,
      right upper quadrant pain or
      tenderness, fever, rash,
      and/or eosinophilia (> 5%),

prompted (for central laboratory) and resampling of the patient should be performed preferably within 48 h after laboratory results are received by the investigator.

Based on the re-test results, it should be determine together with medical monitor if the discontinuation criteria are confirmed. If confirmed, the patient must be withdrawn from the clinical study.

[...]

[...]

The investigator may also decide to stop the The investigator may also decide to stop the treatment with S201086/GLPG1972 (preferably after consultation with the sponsor's study physician) for any of the following reasons:

- Use of concurrent therapy that was not permitted
- Noncompliance with the IMP treatment
- Noncompliance with the clinical study procedures
- Serious or severe AEs
- Worsening of disease condition, which in the investigator's opinion needs an alternative treatment approach not being covered in the clinical study

[...]

5. Presence of evocative clinical symptoms such as jaundice.

In general, an increase of serum aminotransferase (AT) to > 3xULN should be followed by repeat testing preferably within 48h after laboratory results are received by the investigator of all four of the usual serum measures (ALT, AST, ALP, and TBL) to confirm or not the abnormalities.

If any of the above laboratory abnormalities is detected, retesting is prompted (for central laboratory) and resampling of the patient should be performed preferably within 48 h after laboratory results are received by the investigator.

Based on the re-test results, it should be determine together with medical monitor if the discontinuation criteria are confirmed. If confirmed, the patient must be withdrawn from the clinical study.

treatment with S201086/GLPG1972 (preferably after consultation with the sponsor's study physician if applicable) for any of the following reasons:

- Use of concurrent therapy that was not permitted
- Noncompliance with the IMP treatment including overdose
- Noncompliance with the clinical study procedures
- Serious or severe AEs
- Worsening of disease condition, which in the investigator's opinion needs an alternative treatment approach not being covered in the clinical study

# Section 6.1.1. Products administered concerned by the substantial amendment

[...]

The number of TU boxes which will be dispensed to patient at each visit will be different depends on visit: W004, W008 (1 box), W0012, W020 (2 boxes), W028, W040 (3 boxes).

#### Section 6.1.2. IMP management concerned by the substantial amendment

Treatment units will be supplied from the « Unité d'Appui Clinique », Les Laboratoires Servier Industrie, 905 route de Saran, 45520 Gidy, France.

[...]

[...]

# Section 6.6. Previous and concomitant treatments concerned by the substantial amendment

# Treatment prohibited before and during the Treatment prohibited before and during the

Strong opioids: Oxycodone (with or without aspirin, acetaminophen, ibuprofen)

[...]

# study (non-exhaustive list):

Strong opioids: Oxycodone, hydrocodone (with or without aspirin, acetaminophen, ibuprofen)

- Non-pharmacological standard of care (physiotherapy, electrotherapy, etc...) is allowed if stable in the previous 4 weeks and all along the study
- NSAID/Analgesics are authorized during the study without particular conditions for use

# Section 7.2.1. Medical Imaging concerned by the substantial amendment

Before their the study participation CL2-201086-002/GLPG1972-CL-201, all centers will receive a specific training/qualification coordinated by the CRO in charge of medical imaging management.

[...]

In addition, first patient per site will be scanned twice with repositioning at both baseline (W000 visit) and at W052 visit for quantitative measurement to calculate the within study variability.

[...]

Before their participation CL2-201086-002/GLPG1972-CL-201, all centers will receive a specific training/qualification coordinated by the CRO in charge of medical imaging management (MRI qualification protocol).

[...]

In addition, first ONE of the first 3 patients (preferably 3rd) per site will be scanned twice with repositioning at both baseline (W000 visit) and at W052 visit (or if applicable WD visit in case of the patient discontinues the study) for quantitative measurement to calculate the within study variability.

# Section 7.2.2. WOMAC for measurement of pain, function, and stiffness (Appendix 2) concerned by the substantial amendment

WOMAC is a questionnaire designed to assess health status and health outcomes in patients with osteoarthritis of the knee. The questionnaire contains 24 questions targeting areas of pain (5 questions), stiffness (2 questions) and physical function (17 questions). The questionnaire is selfadministered by the patient and can be completed in less than 5 minutes. It refers to the 48h period prior to assessment and will be completed before the clinical examination, preferably in the waiting room.

The WOMAC will be recorded by paper and data will be entered by the investigator or a delegate person on eCRF.

WOMAC (version LK3.1, copyright holder Nicholas Bellamy) is a questionnaire designed to assess health status and health outcomes in patients with osteoarthritis of the knee. The questionnaire contains 24 questions targeting areas of pain (5 questions), stiffness (2 questions) and physical function (17 questions). The questionnaire is self-administered by the patient and can be completed in less than 5 minutes. It refers to the 48h period prior to assessment and will be completed before the clinical examination, preferably in the waiting room.

The WOMAC will be recorded by:

ePRO. The questionnaire will be explained to the patient by the investigator (or a delegate person) and will be filled in by patients during the visits on an electronic

- device (e-PRO). Data entered by the patient will be sent to a central database via a secured transfer,
- paper, in case of unavailability of ePRO, and the original copy will be sent to ePRO provider for data entry and a copy kept by investigator. and data will be entered by the investigator or a delegate person on eCRF.

# Section 7.2.3. and 7.2.4 VAS for pain intensity and for PGA (Appendix 3 & 4) concerned by the substantial amendment

The questionnaire will be explained to the patient by the investigator (or a delegate person) and will be filled in by patients during the visits on an electronic device (e-PRO). Before starting, the patient will need to complete training first. Data entered by the patient will be sent to a central database via a secured transfer.

# Section 8.1. and 8.2. Specification of safety parameters AND Methods and measurement time concerned by the substantial amendment

- Vital signs
- After 5 min. in supine position assessed with automatic blood pressure monitoring (in case of equipment is supplied by the sponsor, equipment has to be used)
  - Systolic blood pressure (SBP) (mmHg)
  - Diastolic blood pressure (DBP) (mmHg)
  - Pulse Rate (bpm)

Vital signs will be evaluated at ASSE, W000, W004, W008, W012, W020, W028, W040, W052, WEND and if applicable at the premature withdrawal visit (WD). Blood pressure will be measured with Automatic Blood Pressure Monitor and SBP and DBP will preferably be measured on the same arm.

- Vital signs
- After 5 min. in supine position assessed
   Assessment with automatic blood pressure monitoring (in ease of equipment is supplied by the sponsor, equipment has to be used) of:
  - Systolic blood pressure (SBP) (mmHg)
  - Diastolic blood pressure (DBP) (mmHg)
  - o Pulse Rate (bpm)

Vital signs will be evaluated at ASSE, W000, W004, W008, W012, W020, W028, W040, W052, WEND and if applicable at the premature withdrawal visit (WD). Blood pressure will be measured with automatic blood pressure monitor and SBP and DBP will preferably be measured on the same arm (in case of equipment is supplied by the sponsor, equipment has to be used).

# Section 8.8. Classification of an adverse event (serious, severity, causality) concerned by the substantial amendment

[...]

[...]

<u>The Severity</u> of AEs should be graded using the modified Common Terminology Criteria for Adverse Events (CTCAE). If a CTCAE criterion does not exist, the investigator should use the grade or adjectives: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (lifethreatening) or Grade 5 (fatal) to describe the maximum intensity of the AE. For purposes of

The Severity of AEs should be graded using the modified Common Terminology Criteria for Adverse Events (CTCAE) version (v.5). If a CTCAE criterion does not exist, the investigator should use the grade or adjectives: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (life-threatening) or Grade 5 (fatal) to describe the maximum intensity of the AE. For purposes of

grades are defined in the table below.

consistency with the CTCAE, these intensity grades are defined in the table below.

[...]

[...]

For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality. This is upon the investigator's assessment.

For AEs associated with laboratory abnormalities, the event should be graded also on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality. This is upon the investigator's assessment.

consistency with the CTCAE, these intensity

# Section 8.9.2.4.2. Special situations concerned by the substantial amendment

 In case of a special situation, the investigator should report it on a "special situation" page of the e-CRF. Any AE associated with a special situation should also be capture in the eCRF («Adverse Event» page).

Any SAE associated with a special situation must be reported following the SAE procedure.

In case the e-CRF is unavailable when the investigator was informed of a special situation, he/she should, within 24 h of knowledge, complete a paper "Special situation" form, send it by fax (or e-mail) to the person(s) designated in the contact details provided in the investigator's study file or outside working hours, the 24-hour phone line is +33.1.55.72.60.00.

As soon as the e-CRF becomes available, the investigator should enter these data in the «Special situation» page of the e-CRF.

If a special situation concerns a person around the study participant, the investigator should not report this on eCRF but must fill in the paper-based "Special Situations Report form" and

- In case of a special situation not associated with an AE (except pregnancy), the investigator should report it on a "special situation not associated with an adverse event" page of the e-CRF.
- In case of a special situation associated with an any AE associated with a special situation, the investigator should report it on an «Adverse Event» page of also be eapture in the eCRF («Adverse Event» page).

Any SAE associated with a special situation must be reported following the SAE procedure.

In case the e-CRF is unavailable when the investigator was informed of a special situation, he/she should, within 24 h of knowledge, complete a paper "Special situation not associated with an adverse event" or "Adverse event", send it by fax (or e-mail) to the person(s) designated in the contact details provided in the investigator's study file or outside working hours, the 24-hour phone line is +33.1.55.72.60.00.

As soon as the e-CRF becomes available, the investigator should enter these data in the «Special situation not associated with an adverse event» or «Adverse event» page of the e-CRF.

- In case of deliberate or accidental S201086/GLPG1972 overdose, general measures to maintain or support the basic vital functions should be taken, if deemed necessary. No experiments have been performed to determine a specific antidote to S201086/GLPG1972.
- If a special situation concerns a person around the study participant, the investigator should not report this on eCRF but must fill in the paper-based "Special Situations Report form" and send it within 24 h of knowledge by fax (or e-mail) to the

send it within 24 h of knowledge by fax (or e-mail) to:



person(s) designated in the contact details provided in the investigator's study file.



# Section 8.9.2.4.3. Pregnancy concerned by the substantial amendment

If pregnancy concerns a patient or a partner of a patient, the investigator immediately after being informed of this event **must fill in the paper-based "Pregnancy Report form"** and send it within 24 h of knowledge by fax (or e-mail) to:



The outcome of pregnancies must be reported. A follow-up contact should be scheduled at the expected time of delivery.

If pregnancy concerns a patient or a partner of a patient, the investigator immediately after being informed of this event **must fill in the paper-based "Pregnancy Report form"** and send it within 24 h of knowledge by fax (or e-mail) to the person(s) designated in the contact details provided in the investigator's study file.



The outcome of pregnancies must be reported. A follow-up contact should be scheduled at the expected time of delivery.

Summary of special situations including pregnancy: Table

## Section 9.2.4. Sampling and storage

| Storage | Storage |
|---------|---------|
| -80°C | -20°C |

## Section 9.3. Other concerned by the substantial amendment

| 9.3 Other Not applicable. | 9.3 Other—Assessment related to exclusion criteria |
|---|---|
| | Not applicable. |
| | The following assessments will be performed on screening samples: |
| | Biological laboratory examinations with Hepatitis B and C, and HIV. |

## Section 10. Statistics concerned by the substantial amendment

| 10.1.1.1.2. Secondary efficacy endpoints The change from baseline to W052 in WOMAC subscales scores for pain, function and stiffness. | |
|---|---|
| 10.1.1.2 Safety endpoints | 10.1.1.2 Safety endpoints |
| [] | [] - Other safety endpoints: Special situations (defined in section 8.5) not associated with an AE. |

# 10.1.1.3

[...]

#### 10.1.2.1 Analysis sets and subgroups

#### - Randomised Set (RS):

All patients to whom a therapeutic unit was randomly assigned using IWRS.

#### - Safety Set (SS):

All patients having taken at least one dose of IMP.

No formal subgroup analysis is planned for this study.

## 10.1.2.2 Treatment groups

Analyses performed on the RS and on the SS will be based on the treatment group assigned as per randomization (randomized treatment).

[...]

# 10.1.3.1.2. Handling of missing data

For the primary analysis, a mixed-effects model for repeated measures approach will be used. For patients with an early discontinuation to the study (delay between the Early Termination and baseline less than 2 months) and without any post baseline measurement of the primary endpoint, a multiple imputation procedure will be used to impute the missing evaluations, assuming that those patients would be in their randomized arm. This approach allows considering that patients will keep the benefit of the randomized treatment after study discontinuation. Multiple imputation, pattern mixture model placebo based imputation, tipping point method and observed cases will be considered for sensitivity analyses (Mallinckrodt & al., 2013).

More details on the strategy defined for handling missing data are provided in Section 10.1.3.3.
[...]

# 10.1.1.3 [...] - [...]

#### 10.1.2.1 Analysis sets and subgroups

#### - Randomised Set (RS):

The Randomised Set (RS) will be constituted of all patients to whom a therapeutic unit was randomly assigned using IWRS. The RS will be used for efficacy analyses. Patients will be analysed according to the randomised treatment.

#### - Safety Set (SS):

The Safety Set (SS) will be constituted of all patients having taken at least one dose of IMP. The SS will be used for safety analyses. Patients will be analysed according to treatment actually received at inclusion.

No formal subgroup analysis is planned for this study.

#### 10.1.2.2. Treatment groups

Treatment groups considered will be S201086/GLPG1972 75 mg, S201086/GLPG1972 150 mg, S201086/GLPG1972 300 mg and placebo.

Analyses performed on the RS and on the SS will be based on the treatment group assigned as per randomization (randomized treatment).

[...]

# 10.1.3.1.2. Handling of missing data

For the primary analysis, a mixed-effects model for repeated measures approach will be used. In this model, two post-baseline time-points will be considered: W028 and W052. From one patient to another, possible distinct situations of remaining missing data have been identified, justifying different statistical treatments.

For patients with only one missing post-baseline measurement, missing data will not be imputed and handled through MMRM. As a reminder, MMRM analysis use all available data, including subjects with partial data (i.e., with missing data) in order to derive an estimate of the treatment effect without filling in the missing items (Mallinckrodt & al., 2013).

For patients for which no post-baseline measurement will be collected for the primary endpoint (regardless the timing of discontinuation), as they cannot be considered

through the MMRM, a MI procedure will be used to impute the missing evaluations as a prior step. This approach allows considering that patients will keep the benefit of the randomized treatment after study discontinuation.

Sensitivity analyses will be performed in order to assess the robustness of the primary analysis results to the handling of missing data method by considering MI, Pattern Mixture Model (PMM) placebo-based imputation, tipping point method and observed cases (Mallinckrodt & al., 2013) detailed in Section 10.1.3.3.1.

For patients with an early discontinuation to the study (delay between the Early Termination and baseline less than 2 months) and without any post baseline measurement of the primary endpoint, a multiple imputation procedure will be used to impute the missing evaluations, assuming that those patients would be in their randomized arm. This approach allows considering that patients will keep the benefit of the randomized treatment after study discontinuation. Multiple imputation, pattern mixture model placebo based imputation, tipping point method and observed cases will be considered for sensitivity analyses (Mallinckrodt & al., 2013).

More details on the strategy defined for handling missing data are provided in Section 10.1.3.3.

[...]

#### **10.1.3.3.1.1.** Primary analysis

#### Main analysis strategy:

In order to meet the primary objective of the study, the efficacy of at least one dose S201086/GLPG1972 as compared to placebo after 52 weeks of treatment in reducing cartilage loss in patients with knee OA will be assessed from the change from baseline to W052 in cartilage thickness as measured in the medial central tibiofemoral compartment on the target knee, in patients of the RS. A restricted maximum likelihood (REML)-based, mixed-effects model for repeated measures approach (so called Mixedeffects Model for Repeated Measures - MMRM) using all longitudinal observations at each postbaseline visit will be used (main analysis). The MMRM as a primary analysis will assume that patients would keep the benefit of the randomized treatment after study discontinuation. For patients with an early discontinuation to the study (delay between the Early Termination and baseline less than 2 months) and without any post baseline measurement of the primary endpoint, a multiple imputation procedure will be used to impute the missing evaluations, assuming that those patients

#### 10.1.3.3.1.1. Primary analysis

#### Main analysis strategy:

In order to meet the primary objective of the study, the efficacy of at least one dose of S201086/GLPG1972 as compared to placebo after 52 weeks of treatment in reducing cartilage loss in patients with knee OA will be assessed from the change from baseline to W052 in cartilage thickness as measured in the medial central tibiofemoral compartment on the target knee, in patients of the RS. A restricted maximum likelihood (REML)-based, mixed-effects model for repeated measures approach (so called Mixedeffects Model for Repeated Measures – MMRM) using all longitudinal observations at each postbaseline visit (W028) (Mallinckrodt et al, 2013) will be used (main analysis). The MMRM as a primary analysis will assume that patients would keep the benefit of the randomized treatment after study discontinuation. A missing data handling will be used (according to section 10.1.3.1.2.) for this analysis. For patients with an early discontinuation to the study (delay between the Early Termination and baseline less than 2 months) and without any post baseline

would be in their randomized arm. For patients with a discontinuation after 2 months since the last MRI, but before the next planned visit, the MRI will be associated with the next planned visit. Other missing evaluations will be handled by the direct likelihood approach through the MMRM modeling. The treatment comparisons associated with the primary analysis will be the contrasts between each dose of \$201086 and placebo at the change from baseline to W52. Analysis will include the fixed, categorical effects of treatment, regions (Asia and Rest of the World), time and treatment-by-time interaction, as well as the continuous, fixed covariates of baseline, time-by-baseline interaction.

The analysis will fit an unstructured covariance matrix, and the assumptions underlying the model will be checked.

The consistency of the results between the Asianregion population and the non-Asian-region population will be evaluated on primary endpoint, according to the Method 2 defined in Ministry of Health Labor and Welfare Notification (MHLW) Notification "Basic principles on Global Clinical Trials". Treatment effect estimates and confidence intervals will be provided, for each dose, in Asianpopulation region and non-Asian-region population. In case of a statistically significant overall treatment effect (in favor S201086/GLPG1972) at a considered dose, the results will be considered consistent if the observed treatment effects in Asian-region and non-Asian-region patients are in favor of S201086/GLPG1972.

[...]

10.1.3.3.1.2. Secondary analyses



measurement of the primary endpoint, a multiple imputation procedure will be used to impute the missing evaluations, assuming that those patients would be in their randomized arm. For patients with a discontinuation after 2 months since the last MRI, but before the next planned visit, the MRI will be associated with the next planned visit. Other missing evaluations will be handled by the direct likelihood approach through the MMRM modeling. The treatment comparisons associated with the primary analysis will be the contrasts between each dose of S201086/GLPG1972 and placebo at the change from baseline to W052. Analysis will include the fixed, categorical effects of treatment, regions (Asia and Rest of the World), time and treatment-by-time interaction, as well as the continuous, fixed covariates of baseline, timeby-baseline interaction.

The analysis will fit an unstructured covariance matrix, and the assumptions underlying the model will be checked.

The consistency of the results between the Asianregion population and the non-Asian-region population (respectively between Japanese population and non-Japanese population) will be evaluated on primary endpoint, according to the Method 2 defined in Ministry of Health Labor and Welfare Notification (MHLW) Notification "Basic principles on Global Clinical Trials". Treatment effect estimates and confidence intervals will be provided, for each dose, in Asianregion population and non-Asian-region population (respectively between Japanese population and non-Japanese population). In case of a statistically significant overall treatment effect (in favor of S201086/GLPG1972) at a considered dose, the results will be considered consistent if the observed treatment effects in Asian-region and non-Asian-region (respectively between Japanese population and non-Japanese population) patients favor are in S201086/GLPG1972.

[...]

10.1.3.3.1.2. Secondary analyses



For each treatment group, descriptive statistics For each treatment group, descriptive statistics will be provided for the primary endpoint (in terms will be provided for the primary endpoint (in terms of value at each visit and change from baseline to of value at each visit and change from baseline to each post-baseline visit), overall and by regions. each post-baseline visit), overall and by regions. [...] [...] 10.1.3.4.3.3. Special situations not associated with an AE Special situations not associated with an AEs will be described in the RS. 10.1.3.5. 10.1.3.5. [...] [...] Section 14.1. Source data concerned by the substantial amendment [...] [...] The following documents are considered as source The following documents are considered as source documents: documents: Notes in the medical file (including nurse Notes in the medical file (including nurse Therapeutic Unit Tracking Form (TUTF) Therapeutic Unit Tracking Form (TUTF) Report/images (e.g. laboratory, ECG, Report/images (e.g. laboratory, ECG, MRI, X-Ray, etc.) MRI, X-Ray, etc.) VAS (pain) and VAS (PGA) recorded by VAS (pain) and VAS (PGA) recorded by Requisition form (e.g. PK) WOMAC recorded by e-PRO or paper (only if ePRO is unavailable) Requisition form (e.g. PK) Section 14.3. Data management concerned by the substantial amendment [...] [...]

The following CROs: MRI central reading center, X-ray central reading center, ePRO provider, ECG central reading center, central laboratory for laboratory central laboratory for tests, bioanalytical data, CRO

IWRS provide electronic transfer of computerized data to the clinical studies data management department. Data are transferred according to a transfer protocol issued by the I.R.I.S. clinical studies data manager.

[...]

The following CROs: MRI central reading center, central medical imaging (X-ray central reading center and MRI data management), ePRO provider, ECG central reading center, central laboratory for laboratory tests, central laboratory for bioanalytical data,

CRO IWRS provide electronic transfer of computerized data to the clinical studies data management department. Data are transferred according to a transfer protocol issued by the I.R.I.S. clinical studies data manager.

# Section 19. Appendices concerned by the substantial amendment

Appendix 2: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)

Appendix 2: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Updated version

Appendix 4: Patient Global Assessment of disease activity Visual Analog Scale

[...]

[....]

Appendix 4: Patient Global Assessment of disease activity Visual Analog Scale

[...]

Please indicate on the line the place that best expresses your feeling as you feel it right now. 0 = very well (on the left) and 100 = very poorly(on the right)

Please indicate on the line the place that best expresses your feeling as you feel it right now.  $0 = \text{very poorly } \frac{\text{well}}{\text{well}}$  (on the left) and 100 = verywell poorly (on the right)

[...]

# Appendix 6: Local Amendment US No 1 to the clinical study protocol

Document title LOCAL AMENDMENT US N° 1 TO THE CLINICAL STUDY

**PROTOCOL** 

Study title Efficacy and safety of 3 doses of S201086/GLPG1972

administered orally once daily in patients with knee

**osteoarthritis.** A 52-week international, multi-regional, multi-center, randomized, double-blind, placebo-controlled, dose-

ranging study.

Test drug code S201086/GLPG1972

Indication Osteoarthritis

Development phase Phase 2

Protocol code CL2-201086-002/GLPG1972-CL-201

*EudraCT Number* 2017-004581-10

Universal Trial Number U1111-1205-0321

Investigational New

Drug Application

Number

133039

Country code INT

Sponsor GALAPAGOS NV (US)

Institut de Recherches Internationales Servier (I.R.I.S.) (ex-US)

Date of the document 12<sup>th</sup> July 2018

Version of the document Final version

## **CONFIDENTIAL**

#### JUSTIFICATION FOR THE AMENDMENT

The main aim of this local amendment for the US is to change the description of the informed consent form (ICF) procedure in the US. The general protocol describes a collection of two original ICFs, whereas in the US the standard way of collection is signing of one original ICF. The patient will be given a copy of the signed original informed consent form.

#### EFFECTS OF THE AMENDMENT

All sites in the US will be concerned by this amendment after approval by Competent Authorities/Ethics Committees.

#### **CHANGES**

Changes and modified text are described below and included in the joined amended protocol in Section 13.3 and Section 13.4.

#### AMENDED TEXT

#### Section 13.3. Patient information and informed consent

[....]

Two original informed consent forms must be completed, dated, and signed by the patient and the investigator (or designee).

If the patient is unable to read, an impartial witness should be present during the entire informed consent collection process. The patient must give consent orally and, if capable of doing so, complete, sign, and personally date the informed consent form. The witness must then complete, sign and date the form together with the person responsible for collecting the informed consent.

The patient will be given one signed original informed consent form, the second original will be kept by the investigator.

[...]

TwoOne original informed consent forms must be completed, dated, and signed by the patient and the investigator (or designee). The patient will be given a copy of the signed original informed consent form.

If the patient is unable to read, an impartial witness should be present during the entire informed consent collection process. The patient must give consent orally and, if capable of doing so, complete, sign, and personally date the informed consent form. The witness must then complete, sign and date the form together with the person responsible for collecting the informed consent.

The patient will be given one signed original informed consent form, the second original will be kept by the investigator.

## Section 13.4. Modification of the information and consent form

[...]

[...]

Each patient affected by the amendment or an independent witness must complete, date and sign two originals of the new version of the

Each patient affected by the amendment or an independent witness must complete, date and sign two-an originals of the new version of the

information and consent form together with information and consent form together with consent discussion. He/she will receive one signed original amendment to the information and consent form.

the person who conducted the informed the person who conducted the informed consent discussion. He/she will receive onea copy of the signed original amendment to the information and consent form.

# Appendix 7: Substantial Amendment No 2 to the clinical study protocol

SUBSTANTIAL AMENDMENT N° 2 TO THE CLINICAL

Document title STUDY PROTOCOL

Study title Efficacy and safety of 3 doses of S201086/GLPG1972

administered orally once daily in patients with knee osteoarthritis. A 52-week international, multi-regional, multi-center, randomized, double-blind, placebo-controlled, dose-

ranging study.

ROCCELLA Study.

Test drug code S201086/GLPG1972

Indication

Osteoarthritis

Development phase

Phase 2

Protocol code

CL2-201086-002/GLPG1972-CL-201

EudraCT Number

2017-004581-10

Universal Trial Number

U1111-1205-0321

Investigational New

Drug Application

Number

133039

Country code

INT

Sponsor

GALAPAGOS NV (US)

Institut de Recherches Internationales Servier (I.R.I.S.) (ex-US)

Date of the document 12 March 2019

Version of the document Final version

#### **CONFIDENTIAL**

| SUBSTANTIAL PROTOCOL AMENDMENT N° 2 | | |
|---|---|---|
| > SUBJECT | > SUBJECT | |
| Inclusion / withdrawal criteria | X | Investigational Medicinal Product (IMP), dosage |
| Number of participants | | Exposure duration to IMP |
| Modification of study design (additional visit / examinations) | | Definition of the end of the trial |
| Primary / secondary endpoints | | New safety information |
| | | Other (specially concomitant X treatments) |
| > CENTRE(S) AND/OR COUNTRIES CONCERNED: ALL | | |

#### JUSTIFICATION FOR THE AMENDMENT

The main justification of this substantial amendment is to widen the recruitment. For that purpose, the following modifications are proposed:

- clarify and/or modify inclusion criteria n°7, 9 and exclusion criteria n° 24, 25, 27, 28, 29, 31, 32, 33, 38, 40, 44
- update of forbidden/authorised concomitant treatments (section 6.6) as regards database reference

These modifications have no impact on the study quality or patient safety.

Minor corrections/clarifications have been made and the main are:

- Section 4.2.2 (laboratory examinations at ASSE visit): A retest is allowed once in case of an unexpected abnormal result, or if the sample could not be analysed.
- Section 5.5.1 withdrawal criteria: other ECG/Laboratory parameter abnormalities detected and not listed in this section will be left at the investigator's judgment for final decision.
- Section 6.2 IMPs administration: clarification on the TU box to use during visits.
- Section 7.2.1 medical imaging:
  - The MRI at baseline is performed before W000 visit (inclusion) because of the Quality Check.
  - Possibility to repeat X-ray/MRI (more than once) after sponsor approval.

- o The results of the study will be given to sites globally and not individually.
- Section 7.2.3 and 7.2.4 VAS: implementation of the VAS paper version in case of unavailability of electronic device (ePRO) (appendix 8).
- Section 8.2: quantitative urinalysis will be performed locally only in case of clinically significant abnormal urinary dipstick result.
- Section 9.2.4: correction made on volumes of blood collected for



- Section 10. Statistics:
  - o Clarification on definition of the randomised set (RS).
  - o Update of position for blood pressure.
- Section 14.1 & 14.4: update of archiving of the eCRF.

#### EFFECTS OF THE AMENDMENT

All sites will be concerned by this amendment after approval by Competent Authorities / Ethics Committees. The participant information and consent form will not be amended.

# **CHANGES**

Changes and modified text are described below and included in the joined amended protocol.

# AMENDED TEXT

| Section Study Summary Sheet concerned by the substantial amendment | |
|---|---|
| Number of patients: | Number of patients: |
| Planned: 852 patients | Planned: approximately 852 patients |
| Per treatment group (arm): 213 patients | Per treatment group (arm): approximately 213 patients |
| Statistical methods: | Statistical methods: |
| Analysis sets: | Analysis sets: |
| - Randomized Set (RS): The Randomised Set (RS) will be constituted of all patients to whom a therapeutic unit was randomly assigned using IWRS. The RS will be used for efficacy analyses. Patients will be analysed according to the randomised treatment. | Modified Randomized Set (mRS): The modified Randomised Set (mRS) will be constituted of all included patients to whom a therapeutic unit was randomly assigned using IWRS. The mRS will be used for efficacy analyses. Patients will be analysed according to the randomised treatment. |
| Section List of abbreviation concerned by the | substantial amendment |
| Poulouis 10 4 | mRS: modified Randomised Set |
| Randomised Set | ROW: Rest of World |
| Section 2. Background information | |
| [] | [] |
| The safety for use during pregnancy has not been established. No data have been generated in nursing women and no data are available on teratogenicity and excretion in milk. Therefore as precaution, women of child-bearing potential (WOCBP) should be excluded from clinical studies with S201086/GLPG1972. | established. No data have been generated in nursing women and no data are available on teratogenicity and excretion in milk. Therefore as precaution, women of |
| Section 4.2.2 Investigation schedule concerned | by the substantial amendment |
| | VAS (pain) [ePRO or paper (only if ePRO is |
| VAS (pain) (ePRO) VAS (PGA) (ePRO) | unavailable)] VAS (PGA) [ePRO or paper (only if ePRO is unavailable)] |
| [] | [] |
| 9. Including Hepatitis B, C and HIV | 9. Including Hepatitis B, C and HIV. If a sample could not be analysed, or in case of unexpected abnormal lab results resampling of the patient for a re-test is allowed once. |
| [] | [] |
| 11.Pre dose PK samples means that patients have to take their IMP at the site | . 11.Pre dose PK samples means that patients have to take their IMP at the site (after the PK-sample was drawn) |
| [] | [] |

## Section 5.1 Inclusion criteria concerned by the substantial amendment

- Symptom severity defined by a pain  $\geq 40 \text{ mm}$  and | 7a. ≤ 90 mm on a 100 mm VAS at screening and inclusion visits (at screening both knees should be assessed for pain and at least one knee should fulfill pain severity defined on this criterion).
- 9.a. Disease stage based on a fixed flexion weightbearing X-ray of the target knee\* and central read out of:
  - a. Predominant medial compartment radiographic disease
  - b. KL grade 2 or 3
  - And OARSI grade 1 or 2 medial tibiofemoral joint space narrowing (JSN)

\*The target knee (right or left) to be followed-up throughout the study will be chosen as follows:

- Symptom severity defined by a pain  $\geq$  40 mm and ≤ 90 mm on a 100 mm VAS at screening and inclusion visits (at screening both knees should be assessed for pain and at least one knee should fulfill pain severity defined on this criterion). A knee not meeting the pain criteria at screening must not be eligible as target knee at inclusion.
- Disease stage based on a fixed flexion weightbearing X-ray of the target knee\* and central read out of:
  - Predominant medial compartment radiographic disease
  - b. KL grade 2 or 3
  - c. And OARSI grade 1 or 2 medial tibiofemoral joint space narrowing (JSN)

\*The target knee (right or left) to be followed-up throughout the study. will be chosen as follows:

# Section 5.2 Exclusion criteria concerned by the substantial amendment

- 24.a. Other pathologies affecting the knee such as: 24b. Other current or medical history of pathologies septic arthritis, inflammatory joint disease, gout, major chondrocalcinosis (pseudogout), Paget's disease of the bone, ochronosis, acromegaly, haemochromatosis, Wilson's disease, rheumatic symptoms due to malignancies, primary osteochondromatosis, osteonecrosis. osteochondritis dissecans, documented severe intra-articular knee injury (e.g. intra-articular fracture), hemophilia, etc.
- 25. Generalized pain syndrome, for example fibromyalgia.
- 27. knee corticosteroid or hyaluronic acid intraarticular injections in the previous 3 months.
- 28. Use of medications with MMP-inhibitory properties (i.e. Tetracycline or structurally related compounds) during the 3 months prior to the screening visit.
- Bisphosphonates, Denozumab, Teriparatide, 29. Strontium ranelate use (in oral or injectable form) in the previous 12 months.
- 31.a. Chronic use of strong opioids and use of other 31b. Chronic use of strong opioids and use of prohibited drugs listed under section 6.6.

- affecting the target knee such as: septic arthritis, inflammatory joint disease, gout, major chondrocalcinosis (pseudogout), Paget's disease ochronosis, of the bone, acromegaly, haemochromatosis, Wilson's disease, rheumatic symptoms due to malignancies, primary osteochondromatosis. osteonecrosis, osteochondritis dissecans, documented severe intra-articular knee injury (e.g. intra-articular fracture), hemophilia, etc.
  - Note: Patients with common risk factors for knee OA - e.g. obesity, meniscectomy - are not excluded.
- 25a. Generalized pain syndrome, for example fibromyalgia Patients with widespread chronic musculoskeletal pain of unclear etiology (i.e. somatic functional syndromes such fibromyalgia, with or without previously documented diagnosis).
- 27a. Knee-Corticosteroid or hyaluronic acid intraarticular injections in the target knee in the previous 3 months.
- 28a. Chronic use of medications with and for MMPinhibitory properties (i.e. Tetracycline or structurally related compounds) during the 3 months prior to the screening visit.
- 29a. Bisphosphonates, denosumab. teriparatide. strontium ranelate, romosozumab use (in oral or injectable form) in the previous 12 months

during 7 days prior to the screening visit (under section 6.6.)

- Any contraindication to MRI according to local 32a. MRI guidelines, including the inability to undergo a knee MRI exam because of inability to fit in the scanner or knee coil.
- 33. Non-pharmacological standard of (Physiotherapy, electrotherapy, etc...) if not stable in the 4weeks prior to the screening visit.
- 38a. Clinically significant abnormalities detected on a 38b. 12-lead ECG performed at screening visit of either rhythm or conduction (e.g., QT interval corrected for HR according to Fridericia's [OTcF] > 450 ms for males and > 470 ms for females, bradycardia with HR < 50 bpm, measured and stable PR > 280 ms, or second or third degree Atrio-Ventricular Block, complete left branch block) (central reading)
- 40. Positive for hepatitis B surface antigen (HBs), anti-hepatitis C virus (HCV) antibodies or antiimmunodeficiency human virus (HIV) antibodies
- of the excipients (e.g.: lactose).

- Any contraindication to MRI according to local MRI guidelines, including or the inability to undergo a knee MRI exam because of inability to fit in the scanner or knee coil. The presence of a pacemaker or any other implanted electronic devices is considered a contraindication to MRI in this study (accommodations will not be made).
- care 33a. Non-pharmacological standard of care for the target knee (physiotherapy, electrotherapy, etc...) if not stable in the initiated less than 4weeks prior to before screening visit.
  - Following elinically significant abnormalities detected on a 12-lead ECG performed at screening visit of either rhythm or conduction (e.g., QT interval corrected for HR according to Fridericia's [OTcF] > 450 ms for males and > 470 ms for females. bradycardia with HR < 50 bpm, measured and stable PR-interval > 280 ms, or second (except Mobitz type 1) or third degree Atrio-Ventricular Block and complete left branch block) as assessed by (central reading).

Any other abnormalies are left to the investigator's judgment for final decision.

- 40a. Positive for anti-human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBs), or anti-hepatitis C virus (HCV) antibodies with a positive test for HCV viral RNA or completion of antiviral HCV treatment ≤ 12 weeks before screening.
- Hypersensitivity to the active substance or to any 44b. Documented hypersensitivity to the active substance or to any of the excipients (e.g.: lactose).

# Section 5.5.1. withdrawal criteria concerned by the substantial amendment

[...]

with S201086/GLPG1972 Treatment discontinued by the investigator and the patient must be withdrawn from the clinical study (preferably after discussion with the monitor, who may consult and must inform the sponsor's study physician if applicable) for any of the following conditions:

- Life-threatening adverse event (AE) or a SAE that places the patient at immediate risk.
- Confirmed pregnancy
- Any ECG and/or laboratory parameter abnormalities such as:
  - QTcF > 500 ms or a delta > 60 ms over baseline value (inclusion) on at least two separate ECGs

[...]

[...]

Treatment with \$201086/GLPG1972 IMP must be discontinued by the investigator and the patient must be withdrawn from the clinical study (preferably after discussion with the monitor, who may consult and must inform the sponsor's study physician if applicable) for any of the following conditions:

- Life-threatening adverse event (AE) or a SAE that places the patient at immediate risk.
- Confirmed pregnancy
- Any The following ECG and/or laboratory parameter abnormalities such as:
  - QTcF > 500 ms or a delta > 60 ms over baseline value (inclusion) on at least two separate ECGs

[....]

The investigator may also decide to stop the treatment with 201086/GLPG1972 (preferably after consultation with the sponsor's study physician if applicable) for any of the following reasons:

[...]

Patients who drop out before the first administration of the IMP will be replaced. Patients who stop taking IMP for any reason will not be replaced.

ſ...

The investigator may also decide to stop the treatment with 201086/GLPG1972 IMP (preferably after consultation with the sponsor's study physician if applicable) for any of the following reasons:

[...]

Patients who drop out before the first administration of the IMP will be replaced. Patients who stop taking IMP for any reason will not be replaced.

[....]

# Section 6.1.1. Products administered concerned by the substantial amendment

[...]

The number of TU boxes which will be dispensed to patient at each visit will be different depends on visit: W004, W008 (1 box), W0012, W020 (2 boxes), W028, W040 (3 boxes).

...]

[...]

The number of TU boxes which will be dispensed to patient at each visit will be different depends on visit: W000, W004, W008 (1 box), W0012, W020 (2 boxes), W028, W040 (3 boxes).

# Section 6.1.2. IMP management concerned by the substantial amendment

[...]

The practical procedures for destruction of unused IMP will be defined by the sponsor and adapted to the center.

[...]

Therapeutic unit tracking form, or an equivalent document, is the source document to fulfill.

...

[...]

The practical procedures for destruction of unused IMP will be defined by the sponsor and adapted to the center.

[...]

Therapeutic unit tracking form, or an equivalent document, is the source document to fulfill be completed.

Section 6.2 IMPs administration concerned by the substantial amendment

[....]

During visits, the IMP will be taken at the site (during the visit) except for W040 (for PK sampling) where IMP will be taken <u>at home</u> and the exact intake time will be reported.

[...]

[...]

[...]

Section 6.3 IMPs dispensing concerned by the substantial amendment

г 1

[....]

The detachable portion of the label on the IMP box must be stuck by the investigator or a delegated person on an IMP label collection form or on the prescription form where the IMPs are dispensed by a pharmacist. ...]

The detachable portion of the label on the IMP box must be stuck by the investigator or a delegated person on an IMP label collection form or on the prescription/IRS form where the IMPs are dispensed by a pharmacist or designee.

Section 6.6 previous and concomitant treatments concerned by the substantial amendment

See on appendix the previous and the new version of tables on prohibited treatments and authorized treatments.

#### Section 7.2.1 Medical imaging concerned by the substantial amendment

#### qMRI

MRI of the target knee will be performed at W000 (inclusion), W028 and W052 visits, and at the withdrawal visit (WD) if the time window between WD and the previous qMRI (W000 or W028) is  $\geq$  2 months.

[...]

All MRI images will be transmitted to the medical imaging management CRO. If a scheduled MRI fails QC, one repeat MRI is allowed.

[...]

All patients results will be returned to the site following finalization of the clinical study report.

#### Radiography (X-ray)

All X-rays will be transmitted to the medical imaging management CRO. If a scheduled X-ray fails QC, one repeat X-ray is allowed (for each knee at the screening visit and for the target knee at every visit when X-ray is scheduled).

[...]

All patients results will be returned to the site following finalization of the clinical study report.

#### qMRI

MRI of the target knee will be performed at after the participant's eligibility (Lab, ECG, X-Ray) has been confirmed and before W000 (inclusion), W028 and W052 visits, and at the withdrawal visit (WD) if the time window between WD and the previous qMRI (W000 or W028) is  $\geq$  2 months.

[...

All MRI images will be transmitted to the medical imaging management CRO. If a scheduled MRI fails QC, one repeat MRI is allowed (for additional MRI repeat the approval of the sponsor is needed).

[...]

All patients results will be returned to the site following finalization of the clinical study report.

#### Radiography (X-ray)

All X-rays will be transmitted to the medical imaging management CRO. If a scheduled X-ray fails QC, one repeat X-ray is allowed (for each knee at the screening visit and for the target knee at every visit when X-ray is scheduled; for additional X-ray repeat the approval of the sponsor is needed)

[...]

All patients results will be returned to the site following finalization of the clinical study report.

# Section 7.2.2 WOMAC concerned by the substantial amendment

[...]

 paper, in case of unavailability of ePRO, and the original copy will be sent to ePRO provider for data entry and a copy kept by investigator. [ ]

 paper, in case of unavailability of ePRO, and a the original copy will be sent to ePRO provider for data entry and the original kept by investigator.

#### Section 7.2.3 & 7.2.4. VAS (pain and PGA) concerned by the substantial amendment

The VAS will be recorded by ePRO. The questionnaire will be explained to the patient by the investigator (or a delegate person) and will be filled in by patients during the visits on an electronic device (e-PRO). Before starting, the patient will need to complete training first. Data entered by the patient will be sent to a central database via a secured transfer.

The VAS will be recorded by:

- ePRO. The questionnaire will be explained to the patient by the investigator (or a delegate person) and will be filled in by patients during the visits on an electronic device (e-PRO). Before starting, the patient will need to complete training first. Data entered by the patient will be sent to a central database via a secured transfer.
- paper, in case of unavailability of ePRO, and a copy will be sent to ePRO provider for data entry and the original kept by investigator (paper version on Appendix 8).

# Section 8.2 Methods and measurement times concerned by the substantial amendment

[...]

Central reading reports overrule local reading for inclusion/exclusion/withdrawal criteria.

[...]

Urinary dipstick will be performed locally. In case of abnormal urinary dipstick result, the investigator or his/her delegate will perform a quantitative urinalysis that will be done locally.

[...]

For the laboratory tests, it is recommended for patients to be fasted (if possible).

[...]

[...]

For Per Protocol inclusion/exclusion/withdrawal criteria, central reading reports overrule local reading.

[...]

Urinary dipstick will be performed locally. In case of clinically significant abnormal urinary dipstick result, the investigator or his/her delegate will perform a quantitative urinalysis that will be done locally.

[....]

For the laboratory tests, it is recommended for patients to be fasted (if possible) and that patients should avoid very vigorous physical exercise or strenuous physical exertion during the 72 hours immediately prior to each blood-draw.

[...

# Section 8.8 Classification of an adverse event concerned by the substantial amendment

AE form

AE form page of the eCRF

#### Section 8.9.2.2 Follow up of adverse event concerned by the substantial amendment

[...]

If the adverse event has not resolved at the patient's final visit in the study, the patient must be followed up suitably and any information on the outcome of the event will be noted on the «Adverse Event» page previously created for the event (e-CRF). The information will be recorded at a follow-up visit.

[...]

[...]

If the adverse event has not resolved at the patient's final visit in the study (WEND), the patient must—will be followed up suitably and any information on the outcome of the event will be noted on the «Adverse Event» page previously created for the event (e CRF). The information will be recorded at a follow up visit until satisfactory resolution (i.e. value back to baseline value or stabilization). Additional information on a patient's AE after resolution can be added at the investigators' discretion to the AE page of the eCRF and to the source documents, until closing of the eCRF for that patient. Thereafter, the investigator can continue to follow-up the patient if deemed necessary, however no further information will be reported into the eCRF.

[...]

# Section 8.9.2.4.2 Special situations concerned by the substantial amendment

S201086/GLPG1972

S201086/GLPG1972 IMP

#### Section 9.1 Pharmacokinetics concerned by the substantial amendment

- At W004, W012, W052 visits and if applicable at the withdrawal visit (WD), one (1) timepoint will be collected (pre-morning dose PK sample). At these visits, the patient takes the IMP at the site.
- At W004, W012, W052 visits and if applicable at the withdrawal visit (WD), one (1) timepoint will be collected (pre-morning dose PK sample). At these visits, the patient takes the IMP at the site.



Section 10. Statistics concerned by the substantial amendment

#### 10.1.1.2. Safety endpoints

The vital signs and clinical examination parameters are the body weight (kg), BMI (kg/m²), supine SBP (mmHg), supine DBP (mmHg) and supine pulse rate (bpm).

#### 10.1.2.1. Analysis sets and subgroups

#### - Randomised Set (RS):

The Randomised Set (RS) will be constituted of all patients to whom a therapeutic unit was randomly assigned using IWRS. The RS will be used for efficacy analyses. Patients will be analysed according to the randomised treatment

#### 10.1.3.4.3.1. Vital signs and clinical examination

Supine blood pressure, body weight and BMI will be described, in terms of value at baseline, value at each post-baseline visit under treatment and last post-baseline value under treatment; as well as in terms of change

#### 10.1.1.2. Safety endpoints

The vital signs and clinical examination parameters are the body weight (kg), BMI (kg/m²), supine SBP (mmHg), supine DBP (mmHg) and supine pulse rate (bpm).

#### 10.1.2.1. Analysis sets and subgroups

# - Modified Randomised Set (mRS):

The modified Randomised Set (mRS) will be constituted of all included patients to whom a therapeutic unit was randomly assigned using IWRS. The mRS will be used for efficacy analyses. Patients will be analysed according to the randomised treatment

#### 10.1.3.4.3.1. Vital signs and clinical examination

Supine Blood pressure, pulse rate, body weight and BMI will be described, in terms of value at baseline, value at each post-baseline visit under treatment and last post-baseline value under treatment; as well as in terms of change from baseline to each post baseline visit under

from baseline to each post baseline visit under treatment and to last post-baseline value under treatment.

treatment and to last post-baseline value under treatment.

Number of emergent relevant decreases/increases, number and percentage of patients with at least one emergent relevant decrease/increase, based on supine SBP, supine DBP and weight will be provided.

Number of emergent relevant decreases/increases, number and percentage of patients with at least one emergent relevant decrease/increase, based on supine SBP, supine DBP, pulse rate and weight will be provided.

10.1.3.5.

10.1.3.5.

# Section 14.1 Source data concerned by the substantial amendment

VAS (pain) and VAS (PGA) recorded by e-PRO

VAS (pain) and VAS (PGA) recorded by e-PRO or paper (only if ePRO is unavailable)

# Section 14.2 Study data concerned by the substantial amendment

[...]

[...]

Data recorded directly on eCRF and considered as source data (see section 14.) must be collected immediately in the eCRF. The other eCRF forms must be completed as soon as possible following each visit.

Data recorded directly on eCRF and considered as source data (see section 14.1) must be collected immediately in the eCRF. The other eCRF forms must be completed as soon as possible following each visit

[...]

L....

After the data base lock, the investigator will receive a CD-ROM containing patient data of his/her center for the study file.

After the data base lock, the investigator will receive a CD ROM containing patient data of his/her center for the study file.

After the data base lock, the investigator, or an authorized member of his/her team, will have to download from the e-CRF an electronic file containing participant data from his/her centre for archiving in the study file (see Section 14.4).

# Section 14.4 Archiving concerned by the substantial amendment

[...]

[...]

At the end of the study, the investigator will be provided with a copy of each patient's data on a CD-ROM support. These data include all data and comments reported in the e-CRF, the history of all queries and signatures and the full audit trail reports.

At the end of the study, the investigator will be provided with a copy of each patient's data on a CD ROM support. These data include all data and comments reported in the e CRF, the history of all queries and signatures and the full audit trail report or an authorized member of his/her team, will download an electronic of each participant's data e-CRF and should keep it in a reliable secure and durable location. The file must include appropriate restrictions (password protection) and adequate protection from loss, physical damage or deterioration for the duration of the archiving period. These data include all data and comments reported in the e-CRF, the history of all queries and signatures and the full audit trail reports.

## Section 18. references concerned by the substantial amendment

[...]

[...]

| | GLPG1972 – investigator's brochure – version n°6/S201086 – investigator's brochure – version n°3. |
|---|---|
| | https://www.fda.gov/Drugs/DevelopmentApprovalProc<br>ess/DevelopmentResources/DrugInteractionsLabeling/<br>ucm093664.htm |
| Section Appendix concerned by the substantia | ll amendment |
| - | Appendix 8: Paper version of the VAS (pain & PGA) |

# Appendix: section 6.6

## Previous version:

Treatment prohibited before and during the study (non-exhaustive list):

| Type of treatment | | | Time since last administration before screening |
|---|---|---|---|
| Symptomatic drugs | oral | Corticosteroids > 7.5 mg/d | 1 month |
| | | Prednisolone or equivalent | |
| | injection | Intra-articular corticosteroids | 3 months |
| | | Intra-articular hyaluronic acid | |
| | oral | Drugs with potential effect on cartilage | 3 months |
| | | e.g. Tetracycline or structurally related compounds | |
| Drugs with an effect on subchondral bone | oral or injection | Bisphosphonates | 12 months |
| subcholidral bolie | Injection | Denozumab | |
| | | Teriparatide | |
| | | Strontium Ranelate | |
| Strong opioids | | Short-acting, More Potent Morphine sulfate Codeine sulfate Oxycodone, hydrocodone (with or without aspirin, acetaminophen, ibuprofen) Hydromorphone Meperidine hydrochloride Fentanyl citrate transmucosal Oxymorphone | Chronic use |
| | | Long-acting Morphine sulfate sustained release Fentanyl transdermal Levorphanol tartrate Oxycodone HCL controlled release Methadone | |



Treatment authorized during the study with particular conditions for use:

| Type of treatment | | | |
|---|---|---|---|
| Symptomatic drugs | oral | Glucosamine (sulphate or others) Chondroitin sulfate diacerein Avocado/soybean unsaponifiables | Under condition of stable dosing for at least 3 months before screening and during the study |

<sup>\*</sup>https://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm

- ✓ Non-pharmacological standard of care (physiotherapy, electrotherapy, etc...) is allowed if stable in the previous 4 weeks and all along the study
- ✓ NSAID/Analgesics are authorized during the study without particular conditions for use

<sup>\*\*</sup>Due to long half-life, Amiodarone is forbidden before and during the study.

# New version:

Table (6.6) 1 - Treatment prohibited during the study (non-exhaustive list)

| Type of treatment | | |
|---|---|---|
| | | Type of treatment |
| Symptomatic drugs | Oral | Chronic corticosteroids > 7.5 mg/d |
| urugs | | Prednisolone or equivalent |
| | Intra-articular injection in the | Corticosteroids |
| | target knee | Hyaluronic acid |
| Experimental or unapproved treatments | Intra-articular<br>injection in the<br>target knee | e.g. amniotic cytokines, platelet-rich plasma |
| Drugs with a potential effect on cartilage | Oral | e.g. Chronic use of tetracycline or structurally related compounds |
| Drugs with an effect on | Oral or injection | Bisphosphonates |
| subchondral<br>bone | | Denosumab |
| | | Teriparatide |
| | | Strontium ranelate |
| | | Romosozumab |

Table (6.6) 2 - Treatment authorized during the study with particular conditions for use

| Table (6.6) 2 - 1 reatment authorized during the study with particular conditions for use | | |
|---|---|---|
| Type of treatment | | |
| Symptomatic oral drugs | Glucosamine (sulphate or others) Chondroitin sulfate Diacerein | Under condition of stable dosing for at least 3 months prior to W000 (inclusion) visit and stable dosing for at least 3 |
| | Avocado/soybean unsaponifiables | months prior W052 visit |
| Intra-articular injection of drugs (except target knee) | Corticosteroids | Allowed if $\geq 1$ month<br>prior to W000 (inclusion)<br>visit and $\geq 1$ month prior<br>to W052 visit |
| Strong opioids | Short-acting, Morphine sulfate Codeine sulfate Oxycodone Hydrocodone (with or without aspirin, acetaminophen, ibuprofen) Hydromorphone Meperidine hydrochloride Fentanyl citrate transmucosal Oxymorphone Long-acting Buprenorphine Morphine sulfate sustained release Fentanyl transdermal Levorphanol tartrate Oxycodone HCL controlled release Methadone | If not chronic use (definition of chronic: 90 days of continuous opioid use or cumulative 120 days of non-continuous opioid use within 1 year.) |
| Non-pharmacological standard of care in the target knee | Physiotherapy, electrotherapy, etc | Allowed if initiated $\geq \frac{4}{2}$ weeks prior to W000 (inclusion) visit and if initiated $\geq 4$ weeks prior to W052 visit |

Table (6.6) 3 - Treatment authorized during the study

| Type of treatment | |
|-------------------------|--------------------------|
| NSAIDs/other analgesics | As needed in the context |
| | of OA standard of care |

# Appendix 8: Paper version of the VAS (pain & PGA)

| STUDY N° CL2-201080-0027 GLPG1972-CL-201 | PATIENT N° | VISIT |
|---|---|---|
| CENTRE N° [ ] | DATE | HOUR : |
| Version 2.0 – 01FEB2018 | Screening visit | |
| K | NEE PAIN | |
| "How would you rate the pain you hav | ve felt in <u>each</u> knee within the last 48 h | ours?" |
| Please indicate on the line the place th<br>48 hours. | nat best expresses your pain as you fel- | t it within the last |
| 0= no pain (on the left) and 100= extre | eme pain (on the right) | |
| Left Knee: | | |
| No pain | Extre | ne pain |
| Right knee: | | |
| No pain | Extre | ne pain |

CL2-201086-002 / GLPG1972-CL-201

1/3

| STUDY N° CL2-201088-002 / GLPG1972-CL-201 | PATIENT N° | VISIT |
|-------------------------------------------|----------------|----------------|
| CENTRE N° LLLLL | DATE dd mm ywy | HOUR : |
| Version 2.0 - 01FEB2018 | | |

# Other visits

# KNEE PAIN

"How would you rate the pain you have felt in the <u>study knee</u> within the last 48 hours? If you are unsure which knee is your study knee, please ask your research doctor before answering."

Please indicate on the line the place that best expresses your pain as you felt it within the last 48 hours.

0= no pain (on the left) and 100= extreme pain (on the right)



CL2-201086-002 / GLPG1972-CL-201

| STUDY N° CL2-201088-002 / GLPG1972-CL-201 | PATIENT N° | VISIT |
|-------------------------------------------|-----------------|----------------|
| CENTRE N° | DATE dd mm yyyy | HOUR : |
| Version 2.0 - 01FEB2018 | | |

# PATIENT GLOBAL ASSESSMENT

"Considering all the ways in which your knee osteoarthritis affects you, please rate on this 100 mm scale how well you are doing today"

Please indicate on the line the place that best expresses how you feel right now. 0= very poorly (on the left) and 100=very well (on the right)

| very poorly | very well |
|-------------|-----------|

CL2-201086-002 / GLPG1972-CL-201

# Appendix 9: Non-substantial Amendment No 3 to the clinical study protocol

NONSUBSTANTIAL AMENDMENT N° 3 TO THE CLINICAL

Document title STUDY PROTOCOL

Study title Efficacy and safety of 3 doses of S201086/GLPG1972

administered orally once daily in patients with knee osteoarthritis. A 52-week international, multi-regional, multi-center, randomized, double-blind, placebo-controlled, dose-

ranging study.

ROCCELLA Study.

Test drug code S201086/GLPG1972

Indication

Osteoarthritis

Development phase

Phase 2

Protocol code

CL2-201086-002/GLPG1972-CL-201

EudraCT Number

2017-004581-10

Universal Trial Number

U1111-1205-0321

Investigational New

Drug Application

Number

133039

Country code

US

Sponsor

GALAPAGOS NV (US)

Institut de Recherches Internationales Servier (I.R.I.S.) (ex-US)

Date of the document 00 r

09 December 2019

Version of the document Final version

## **CONFIDENTIAL**

## JUSTIFICATION FOR THE AMENDMENT



In addition, the sponsor has decided to subcontract with a contract research organization (CRO). The PK data will be transferred from the bioanalytical lab to the modelling CRO. The sponsor will not have access to the PK data. In order to maintain the blind, the modelling CRO will perform its activity independently of the sponsor and will not share data that may lead to unblinding before database lock.

Minor corrections/clarifications have been made.

## EFFECTS OF THE AMENDMENT

All US sites will be concerned by this amendment.

#### **CHANGES**

Changes and modified text are described below and included in the joined amended protocol.

## AMENDED TEXT



| Section 4.1 Endpoints concerned by the amendment | |
|---|---|
| Exploratory endpoints: | Exploratory endpoints: |
| - | - |
| Section 4.2.2 Investigation schedule concerned by the | e amendment |
| Physical examination including knees: Screening, Inclusion, W004, W008, W012, W020, W028, W052, WD, WEND | Physical examination including knees: Screening, Inclusion, W004, W008, W012, W020, W028, W040, W052, WD, WEND |
| [] | [] |
| 11. Pre dose PK samples means that patients have to take their IMP at the site (after the PK-sample was drawn). | 11. Pre dose PK samples means that patients have to take their IMP at the site (after the PK-sample was drawn). At W052 or WD, no IMP should be taken. |
| [] | [] |
| Section 4.3 measures to minimize bias concerned by the amendment | |
| - Samples for pharmacokinetic analysis will be sent to the central laboratory and transferred to the assay center. The assay center in charge of \$201086/GLPG1972 measurement in biological matrices will be provided with the treatment codes so that only samples from patients being treated with \$201086/GLPG1972 will be assayed (patients under active treatment). The results of the \$201086/GLPG1972 plasma concentration will be transferred from assay center to the I.R.I.S. pharmacokinetic department before the clinical database is locked (recoded patient number). In order to prevent a blind break, administration and sample times will only be recorded on the requisition form (not on the electronic case report form [eCRF]). The central laboratory will capture the data of the requisition form and will calculate the time after dose. Real time after dose will be transferred to the assay center for analyses. PK results from | - Samples for pharmacokinetic analysis will be sent to the central laboratory and transferred to the assay center. The assay center in charge of S201086/GLPG1972 measurement in biological matrices will be provided with the treatment codes so that only samples from patients being treated with S201086/GLPG1972 will be assayed (patients under active treatment). The results of the S201086/GLPG1972 plasma concentration will be transferred from assay center to the I.R.I.S. pharmacokinetic department a CRO independent of the sponsor before the clinical database is locked (recoded patient number). During the modelling activity until the database lock, there will be no communication between the sponsor and the CRO. During the study until the database lock, no PK results will be provided to the sponsor in order to avoid any unblinding, and requisition form data will be transferred from the central laboratory to the I.R.I.S. Data Management department. In order to prevent a blind break, |

assay center and requisition form data from the central laboratory will be transferred to the I.R.I.S. Data Management department only after blind broken. administration and sample times will only be recorded on the requisition form (not on the electronic case report form [eCRF]). The central laboratory will capture the data of the requisition form and will calculate the time after dose. Real time after dose will be transferred to the assay center for analyses. PK results from assay center and requisition form data from the central laboratory will be transferred to the I.R.I.S. Data Management department only after blind broken.

#### Section 9.1 Pharmacokinetics concerned by the amendment

[...]

• At W004, W012, W052 visits and if applicable at the withdrawal visit (WD), one (1) time-point will be collected (pre-dose PK sample). At these visits, the patient takes the IMP at the site.

• At W004, W012, W052 visits and if applicable at the withdrawal visit (WD), one (1) time-point will be collected (pre-dose PK sample). At these visits, the patient takes the IMP at the site (at W052 or WD, no IMP should be taken).

[...]



